

A Phase 2, Randomized, Double-Blind, Placebo- Controlled Study of the Efficacy and Safety of CF102 in the Second-Line Treatment of Advanced Hepatocellular Carcinoma in Subjects with Child-Pugh Class B Cirrhosis

# STATISTICAL ANALYSIS PLAN Version 7.0 29 August 2019

#### CONFIDENTIAL

#### **Submitted to:**

Motti Farbstein Chief Operating Officer

Pnina Fishman, PhD Chief Executive Officer Can-Fite BioPharma, Ltd 10 Bareket St. Kiryat Matalon, Petach Tikva 49170 Israel

Michael H Silverman, MD BioStrategics Consulting, Ltd Marblehead, MA 01945 USA

## Prepared by:

David R. Bristol, PhD
Statistical Consulting Services Inc.
2075 Denise Lane
Winston-Salem, North Carolina 27127 USA

# SIGNATURE PAGE

| Prepared by: | |
|---|---|
| David Bristol, PhD Statistical Consulting Services, Inc. | Date |
| Approved by: | |
| Michael H. Silverman, MD<br>BioStrategics Consulting, Ltd. | Date |
| Motti Farbstein<br>Chief Operating Officer<br>Can-Fite BioPharma, Ltd. | Date |
| Pnina Fishman, PhD Chief Executive Officer Can-Fite BioPharma, Ltd. | Date |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| A <sub>3</sub> AR | Adenosine A3 receptor (A <sub>3</sub> AR) |
| AASLD | American Association for the Study of Liver Diseases |
| AE(s) | Adverse event(s) |
| AFP | α-fetoprotein (alpha-fetoprotein) |
| ALT | Alanine Aminotransferase (also referred to as SGPT, ALAT) |
| ANC | Absolute neutrophil count |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase (also referred to as SGOT, ASAT) |
| BID | Twice a day |
| BMI | Body mass index |
| BUN | Blood Urea Nitrogen |
| CBC | Complete blood count |
| CF102 | Sponsor defined name for the study medication |
| CFB | Change From Baseline |
| cm | Centimeter(s) |
| CP | Child-Pugh |
| CPB | Child-Pugh Class B (cirrhosis) |
| CR | Complete Response |
| CRF | Case Report Form |
| CS | Clinically Significant |
| CT | Computed Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DB | Double Blind |
| DC | Disease Control ( $CR + PR + SD$ ) |
| DCR | Disease Control (CR + PR + SD) Rate; also referred to as DC Rate |
| ECG | Electrocardiogram |
| ECOG | Eastern Collaborative Oncology Group |
| EHS | Extrahepatic Spread |
| EOS | End Of Study (end of dosing) |
| HBV | Hepatitis B Virus |
| HCC | Hepatocellular carcinoma |
| HCV | Hepatitis C Virus |
| HR | Heart rate |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| ID | Identification |
| IMP | Investigational medicinal product |
| INR | International normalized ratio |
| ITT | Intent-to-treat |
| kg | Kilogram(s) |
| KM | Kaplan-Meier |
| LD | Longest diameter |
| LDH | Lactate dehydrogenase |

| Abbreviation | Definition |
|---|---|
| LOCF | Last observation carried forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram(s) |
| mmHg | Millimeter of Mercury |
| MRI | Magnetic resonance imaging |
| NAB | Normal Approximation to the Binomial Distribution |
| NCI | National Cancer Institute |
| NCS | Not clinically significant |
| NYHA | New York Heart Association |
| OL | Open Label |
| OR | Objective response (CR + PR) |
| ORR | Objective response (CR + PR) Rate; also referred to as OR Rate |
| OS | Overall Survival |
| PBMC | Peripheral blood mononuclear cells |
| PD | Progressive disease |
| PE | Physical examination |
| PFS | Progression-Free Survival |
| PK | Pharmacokinetic(s) |
| PO | per os; oral(ly) |
| PR | Partial response |
| PS | Performance status |
| PT | Prothrombin Time (laboratory parameter); |
| | Preferred Term (MedDRA) |
| PTT | Partial Thromboplastin Time |
| PVT | Portal Vein Thrombosis |
| QTc | Corrected QT |
| QTcF | Corrected QT (Fridericia) |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Stable disease (also Standard Deviation in tables) |
| SE | Standard Error |
| SGOT | Serum Glutamic Oxaloacetic Transaminase (also referred to as AST) |
| SGPT | Serum Glutamic Pyruvic Transaminase (also referred to as ALT) |
| SOC | System Organ Class (MedDRA) |
| TEAE | Treatment-emergent adverse event |
| TTP | Time To Progression |
| ULN | Upper limit of normal |
| WBC | White blood cell count |

| Section | on TABLE OF CONTENTS | Page |
|---|---|---|
| 1. I | NTRODUCTION AND BACKGROUND | 7 |
| 2. 1 | TRIAL DESIGN | 7 |
| 2.1 | Study Objectives | |
| 2.1 | STUDY DESIGN | |
| 2.3 | STUDY DRUG DOSAGE AND ADMINISTRATION | |
| 2.4 | Dose Modification | |
| 3. S | SAMPLE SIZE, RANDOMIZATION AND BLINDING | 9 |
| 3.1 | Sample Size | 9 |
| 3.2 | RANDOMIZATION AND BLINDING | |
| 4. S | SELECTION AND WITHDRAWAL | 9 |
| 4.1 | Inclusion Criteria | 9 |
| 4.2 | Exclusion Criteria | |
| 4.3 | DISCONTINUATION FROM DOSING | |
| 4.4 | WITHDRAWAL FROM THE TRIAL | 12 |
| 5. ( | CLINICAL PROCEDURES AND ASSESSMENTS | 12 |
| 7 | Table 1–1: Schedule of Events for Double Blind (DB) Period | 13 |
| | Table 1–2: Schedule of Events for Open Label (OL) Period | |
| 6. S | STUDY ENDPOINTS | 17 |
| 6.1 | Efficacy Assessments | 17 |
| | 6.1.1 Time to Event Endpoints | |
| 6 | 5.1.2 Tumor Response | |
| 6 | 5.1.3 Exploratory Efficacy | |
| 6.2 | SAFETY EVALUATIONS | 18 |
| 7. S | STATISTICAL CONSIDERATIONS AND DATA ANALYSIS | 19 |
| 7.1 | ANALYSIS POPULATIONS | 20 |
| 7.2 | GENERAL ANALYSIS | 20 |
| 7.3 | SUBJECT DISPOSITION | |
| 7.4 | | |
| | 7.4.1 Demographics | |
| | 7.4.2 HCC Disease History And Prior Therapies | |
| 7.5 | 7.4.3 Medical History Medicat History Medication and Treatment Analysis | |
| , | 7.5.1 Compliance and Exposure | |
| | 7.5.2 Concomitant Medications | |
| 7.6 | | |
| 7 | 7.6.1 Overall Survival (OS) | |
| | 7.6.2 Time to Progression (TTP) | |
| | 7.6.3 Progression-Free Survival (PFS) | |
| | 7.6.4 Tumor Response | |
| / | 7.6.5 Biomarkers | 24 |

| | 7.6.6 | Chemistry And Coagulation Parameters | 25 |
|---|---|---|---|
| | 7.6.7 | | |
| | 7.6.8 | Subgroup Analyses | |
| 7. | 7 S | SAFETY ANALYSES | |
| | 7.7.1 | Adverse Events | 27 |
| | 7.7.2 | Laboratory Tests | |
| | | ECOG Performance Status | |
| | | Vital Signs and Weight | |
| | | ECG Parameters | |
| | 7.7.6 | Physical Examinations | 29 |
| 8. | MISS | ING DATA | 30 |
| 9. | DIFF | ERENCES AND CHANGES FROM THE PROTOCOL | 30 |
| 10. | AP | PENDICES | 32 |
| 10 | ).1 <i>A</i> | APPENDIX A – CHILD-PUGH CLASSIFICATION OF SEVERITY OF LIVER | 2 DISEASE 32 |
| 10 | ).2 <i>A</i> | APPENDIX B – DETERMINATION OF OVERALL RESPONSE | 33 |
| 10 | ).3 <i>A</i> | APPENDIX C – CLINICAL LABORATORY TESTS | 37 |
| 10 | ).4 <i>A</i> | APPENDIX D – ECOG PERFORMANCE STATUS | 38 |
| 10 | ).5 A | APPENDIX E – CARDIAC FUNCTION CLASSIFICATION | 39 |

#### 1. INTRODUCTION AND BACKGROUND

This Statistical Analysis Plan (SAP; Version 7.0) is to be used in conjunction with the protocol (Amendment 5, dated 6 November 2018) and the corresponding case report forms (CRFs). Table shells and mock listings corresponding to the contents of this document will be prepared and included with the final version. This document, with table shells and mock listings, will be reviewed prior to unblinding, and revised if necessary. The contents of this document were developed prior to unblinding, except as noted.

CF102 is a selective, high affinity agonist for the human adenosine A<sub>3</sub> receptor (A<sub>3</sub>AR) and is being developed as a non-cytotoxic agent for the treatment for hepatocellular carcinoma (HCC). A<sub>3</sub>ARs are expressed primarily in normal lung, liver, kidney and heart tissues, with very little expression in the brain or in skeletal muscle. A<sub>3</sub>ARs are over-expressed by human HCC cells, but not those from healthy donors. A<sub>3</sub>AR expression is also elevated in PBMC isolated from patients with hepatitis C viral (HCV) infections. Further details are given in the protocol.

#### 2. TRIAL DESIGN

#### 2.1 STUDY OBJECTIVES

The primary objective of this trial is to:

• Evaluate the efficacy of orally administered CF102 25 mg BID as compared to placebo, as determined by Overall Survival (OS), when used as second-line therapy in subjects with advanced hepatocellular carcinoma (HCC) and Child-Pugh Class B (CPB) cirrhosis.

The secondary objectives of this trial are to:

- Evaluate other indicators of efficacy of CF102 25 mg BID as compared to placebo, including time to progression (TTP), progression-free survival (PFS), objective response (OR) rate, and disease control (DC) rate in this population;
- Explore exposure-response relationships using sparse pharmacokinetic (PK) sampling;
- Characterize the safety profile of CF102 25 mg BID in subjects with advanced HCC and CPB cirrhosis;
- Characterize the effects of CF102 25 mg BID on laboratory parameters associated with viral hepatitis, hepatic dysfunction, and cirrhosis; and
- Explore the relationship between the white blood cell (WBC) adenosine A<sub>3</sub> receptor (A<sub>3</sub>AR) expression and clinical response.

The planned analyses of PK results will be presented in a separate document.

#### 2.2 STUDY DESIGN

This is a multicenter, randomized, double-blind, placebo-controlled clinical trial in subjects with advanced HCC and CPB cirrhosis who did not tolerate prior sorafenib therapy or experienced disease progression on prior sorafenib therapy. The trial will evaluate the efficacy and safety of CF102 25 mg BID as compared to placebo.

Tumor imaging will be performed every 8 weeks. Treatment will continue until the subject experiences unacceptable drug-related intolerability. Subjects will return for a follow-up visit 28 days after completion of the last dose of study drug, and every attempt will be made to obtain survival data on all randomized subjects. Subjects who discontinue will be followed indefinitely for survival status. Enrollment will continue until 75 deaths have been recorded. All randomized subjects will continue to be followed for survival status after 75 deaths have been recorded.

Once the requisite number of events has occurred and the blind is broken for analysis of the trial results, any surviving subjects who remain on blinded drug will be offered the opportunity to continue dosing with open-label CF102 25 mg BID indefinitely, following the protocol-specified schedule of events (<u>Table 1-2</u>), referred to below as the Open-Label (OL) period. The period prior to breaking the blind is referred to as the Double-Blind (DB) period. Bottles of study drug dispensed to subjects at the start of each treatment cycle during the OL period will contain a sufficient supply of CF102 for one cycle (28 days) of continuous dosing.

#### 2.3 STUDY DRUG DOSAGE AND ADMINISTRATION

Subjects will be randomly assigned in a 2:1 ratio to treatment with either CF102 25 mg or matching placebo. CF102 or placebo will be self-administered orally twice daily (BID) on an empty stomach (1 hour before or 2 hours after meals) beginning on Day 1 of the trial and thereafter at approximately the same times each day of the 28-day cycle.

During the OL period, CF102 will be administrated in continuous 28-day cycles beginning on Day 1 of Cycle 1 of the OL period.

#### 2.4 DOSE MODIFICATION

Any safety-related modification of study drug dosing (i.e., dose reduction or interruption of scheduled dosing) and the reason for such action must be clearly noted on the Adverse Events page of the CRF, and the Medical Monitor informed.

In the case of any Grade 3 toxicity by CTCAE v4.0 judged by the Principal Investigator to be at least "possibly" drug-related, the dose of study drug will be interrupted for up to 7 days. If toxicity does not resolve to Grade  $\leq 1$  within 7 days, the subject will be discontinued from treatment. If toxicity resolves to Grade  $\leq 1$  within 7 days, dosing will be resumed at the decreased dose of 1 capsule per day.

In the case of any Grade 4 toxicity judged by the Principal Investigator to be at least "possibly" drug-related, the dose of study drug will be withdrawn permanently.

Only 1 dose reduction will be allowed. If a Grade 3 or 4 toxicity judged by the Principal Investigator to be at least "possibly" drug-related occurs upon rechallenge at the reduced dose, study drug dosing will be withdrawn permanently.

#### 3. SAMPLE SIZE, RANDOMIZATION AND BLINDING

#### 3.1 SAMPLE SIZE

Approximately 78 subjects will be enrolled during an accrual period estimated to be approximately 102 weeks (24 months) in duration and randomized to either CF102 or placebo using a 2:1 randomization. The post-accrual treatment period will continue until a total of 75 subjects have died. Assuming a hazard ratio of 0.5, 75 deaths will provide 80% power for the logrank test at level 0.05 (EAST 6, Cytel, 2014).

#### 3.2 RANDOMIZATION AND BLINDING

On Day 1, each subject will be randomly assigned to receive either CF102 25 mg BID or placebo BID, using a 2:1 randomization. The subject ID number identifies the subject and consists of the site number followed by the subject number for that site. The randomization number identifies the treatment.

The trial will be double-blind; the subject, Investigator/staff, and Sponsor will not have access to or knowledge of any subject's treatment assignment. Upon completion of the DB period, the blind will be broken and all analyses will be performed. Any surviving subjects who remain on blinded drug will be offered the opportunity to continue dosing with open-label CF102 25 mg BID indefinitely (OL Period).

#### 4. SELECTION AND WITHDRAWAL

#### 4.1 INCLUSION CRITERIA

#### <u>Inclusion Criteria (DB Period)</u>

Subjects must meet all of the following inclusion criteria to be eligible for the trial:

- 1. Males and females at least 18 years of age.
- 2. Diagnosis of HCC:
  - For subjects without underlying cirrhosis at the time of diagnosis, diagnosis of HCC documented by cytology and/or histology.
  - For subjects with underlying cirrhosis at the time of diagnosis, diagnosis of HCC established according to the American Association for the Study of Liver Diseases Practice Guideline algorithm (Appendix E of the protocol).
- 3. HCC is advanced, i.e., treatment-refractory or metastatic, and no standard therapies are expected to be curative.
- 4. Receipt of prior sorafenib therapy for at least 3 weeks and withdrawal from treatment due either to intolerability or to radiographic evidence of disease progression. If treatment was withdrawn due to intolerability manifested as a Grade 3 or 4 event by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE v4.0), less than 3 weeks of continuous prior administration prior to withdrawal is acceptable (see also Exclusion Criterion #3).
- 5. Prior sorafenib treatment was discontinued for at least 2 weeks prior to the Baseline Visit.

- 6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2 (Appendix D).
- 7. Cirrhosis classified as Child-Pugh Class B (Appendix A).
- 8. The following laboratory values must be documented  $\leq 3$  days prior to the first dose of study drug:
  - Absolute neutrophil count (ANC)  $\geq 1.5 \times 10^9/L$
  - Platelet count  $\geq 75 \times 10^9 / L$
  - Serum creatinine  $\leq 2.0 \text{ mg/dL}$
  - Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)
     ≤ 5 × the upper limit of normal (ULN)
  - Total bilirubin  $\leq 3.0 \text{ mg/dL}$
  - Serum albumin  $\geq 2.8 \text{ g/dL}$
  - Prothrombin time (PT) no greater than 6 seconds longer than control.
- 9. Life expectancy of  $\geq 6$  weeks.
- 10. For women of childbearing potential, negative serum pregnancy test result.
- 11. Provide written informed consent to participate.
- 12. Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other trial-related procedures.

#### Inclusion Criteria (OL Period)

- 1. The subject signed the ICF for the Open Label treatment.
- 2. The subject received double blind treatment with CF102/placebo and is still taking the investigational medication when Amendment 5 is approved.

#### 4.2 EXCLUSION CRITERIA

Subjects meeting any of the following criteria are <u>ineligible</u> for the trial:

- 1. Receipt of no, or of >1, prior systemic drug therapies for HCC.
- 2. Receipt of systemic cancer therapy, immunomodulatory drug therapy, immunosuppressive therapy, or corticosteroids > 20 mg/day prednisone or equivalent within 14 days prior to the Baseline Visit or concurrently during the trial.
- 3. Presence of an acute or chronic toxicity of prior chemotherapy that has not resolved to ≤ Grade 1, as determined by CTCAE v 4.0.
- 4. Locoregional treatment within 4 weeks prior to the Baseline Visit.
- 5. Major surgery or radiation therapy within 4 weeks prior to the Baseline Visit.
- 6. Use of any investigational agent within 4 weeks prior to the Baseline Visit.
- 7. Child-Pugh Class A or C cirrhosis or hepatic encephalopathy.
- 8. Occurrence of esophageal or other gastrointestinal hemorrhage requiring transfusion within 4 weeks prior to the Baseline Visit.
- 9. Uncontrolled or clinically unstable thyroid disease, per judgment of the Principal Investigator.
- 10. Active bacterial, viral, or fungal infection requiring systemic therapy, or operative or radiological intervention.
- 11. Known human immunodeficiency virus- or acquired immunodeficiency syndrome- related illness.

- 12. Liver transplant.
- 13. Active malignancy other than HCC.
- 14. Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4) (Appendix E).
- 15. Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
- 16. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to >450 msec for males or >470 msec for females.
- 17. Pregnant or lactating female.
- 18. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the Investigator's opinion, are effective and adequate for the subject's circumstances while on study drug.
- 19. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward.
- 20. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with trial participation or study drug administration; may interfere with the informed consent process and/or with compliance with the requirements of the trial; or may interfere with the interpretation of trial results and, in the Investigator's opinion, would make the subject inappropriate for entry into this trial.

#### 4.3 DISCONTINUATION FROM DOSING

Discontinuation from dosing means that the EOS visit is to be performed upon termination and indefinite monthly survival follow-up will be performed.

Subjects should be discontinued from dosing for the following reasons:

- Grade 3 toxicity considered by the Investigator to be at least "possibly" drugrelated that does not resolve to Grade ≤ 1 within 7 days following interruption of treatment.
- Need for > 1 dose reduction.
- Grade 4 toxicity considered by the Investigator to be at least "possibly" drug-related.
- Treatment interruption or delay for more than 14 days after the next scheduled dose due to an event unrelated to toxicity (e.g., intercurrent illness, scheduled surgery, etc.).
- Subject withdrawal of consent for trial participation at any time, for any reason, and without prejudice.
- Withdrawal of a subject by the Investigator, at his/her discretion, for any reason that the Investigator believes continuation of study drug therapy would not be in the subject's best interest. The reason for the subject's discontinuation must be recorded on the case report form (CRF).

- An intercurrent illness which, in the Investigator's opinion, would prevent completion of trial-related evaluations.
- Pregnancy.
- Subject noncompliance with trial or follow-up procedures.
- Termination of the trial by the Sponsor.

If a subject is withdrawn from treatment, the Investigator will make every effort to complete all final evaluations and laboratory tests required by the protocol. The reason(s) for discontinuation of dosing must be clearly documented on the CRF. Subjects who discontinue from dosing will be followed indefinitely for survival status.

#### 4.4 WITHDRAWAL FROM THE TRIAL

A subject will be considered to be withdrawn from the trial for the following reasons:

- Withdrawal of consent (in which every effort will be made to follow the subject for survival information);
- Termination of the trial by the Sponsor;
- Patient Death;
- Other.

#### 5. CLINICAL PROCEDURES AND ASSESSMENTS

The schedule of clinical procedures and assessments conducted during the study is presented in the following table. Further details are given in the protocol.

TABLE 1–1: SCHEDULE OF EVENTS FOR DOUBLE BLIND (DB) PERIOD

| | | | Cycle 1 | Subse<br>Cy | quent<br>cles | End of Study/ End of Dosing (EOS) <sup>1</sup> | Follow-Up |
|---|---|---|---|---|---|---|---|
| Trial Procedures | Pre-Study (-28 days) | Day 1<br>Baseline | Days 8 and 15 ± 2 days | Day 1 ± 2 days | Day 15 ± 2 days | Day 1 + 2 days | (28 ± 3 Days<br>Post- EOS) |
| Medical history | X | | | | | | |
| Physical examination | X <sup>a</sup> | $X^{a,c}$ | $X^{b}$ | X <sup>b</sup> | $X^{b}$ | $X^b$ | $X^{a}$ |
| Inclusion/exclusion criteria | X | X | | | | | |
| Informed consent | X | | | | | | |
| Body weight | X | X <sup>c</sup> | | X | | X | X |
| Vital signs <sup>d</sup> | X | X | X | X | X | X | X |
| Clinical laboratory testing <sup>e</sup> | X | X <sup>c</sup> | X | X | X | X | X |
| T3. T4, TSH | X | X | | X | | X | X |
| ECG <sup>f</sup> | X | X | X | X | X | X | X |
| Pregnancy test (serum) <sup>g</sup> | X | X <sup>c</sup> | | X | | X | X |
| ECOG PS <sup>g</sup> | X | X <sup>c</sup> | | X | | X | |
| α-fetoprotein (AFP) | | X | | X | | X | X |
| WBC A3AR sample | | X | | X <sup>h</sup> | | | |
| PK samples | | $X^k$ | $X^k$ | X <sup>k</sup> | | | |
| Hepatitis B/C virus serology | X | | | | | | |
| Hepatitis B/C viral load (if | | X | | $X^{i}$ | | $X^{i}$ | |
| seropositive) | | Λ | | | | | |
| Tumor imaging for RECIST | $X^{J}$ | | | $X^{j}$ | | X | |
| Concomitant medications | X | X | X | X | X | X | X |
| Adverse events | | X | X | X | X | X | X |
| Dispense study drug supplies | | X | | X | | | |
| Review treatment compliance | | X | X | X | X | X | |

Symptom-directed examination.

c If Pre-Study assessment was performed \le 3 days prior to the Baseline Visit, assessments do not need to be repeated prior to

d Temperature, pulse, respiration, blood pressure at: Pre-Study; pre-dose at all visits; at 1, 2, 3, 4h (± 5 min), 6 and 8h (± 10 min) post-dose on Cycle 1 Day 1; and at Follow-up.

<sup>e</sup> See list of parameters in Appendix C.

FECG at Pre-Study; pre-dose at all visits; and at 2, 4, and 8h (± 10 min) post-dose on Cycle 1 Day 1; and at Follow-up.

Performed at Pre-Study, prior to the first dose, at the end of each cycle, and at Follow-up.

Day 1 of odd-numbered cycles, unless waived by the Sponsor (selected sites only).

For subjects with measurable viral load at the Baseline Visit; on Day 1 of odd-numbered cycles only and at EOS.

To subjects with heasthable vital load at the Baseline Visit, on Day 1 of odd-humbered cycles only and at EOS.

CT scan or MRI at Pre-Study, the end of Cycle 2, and at the end of subsequent even-numbered cycles. For trial eligibility purposes, a scan performed ≤ 21 days prior to the Pre- Study Visit may be used (allowed time window is of -7/+1 day with respect to day 28 of each even numbered cycles; if performed at +1 day after day 28, CT/MRI scan must be performed before administration of the morning dose of that day)

k Sparse sampling on Day 1 of Cycles 1 and 2 only. Pre-dose trough samples on Cycle 1 Days 8 and 15 only. See Table 10-1 of

the protocol for PK sampling time points.

End of Study visit timeframe is of 2 days since the last administered dose of IMP/matching Placebo.

<sup>&</sup>lt;sup>a</sup> Complete PE performed at the Pre-Study (and/or the Baseline Visit if performed > 3 days prior to first dose) and End of Study/End of Dosing (EOS) visits.

TABLE 1–2: SCHEDULE OF EVENTS FOR OPEN LABEL (OL) PERIOD

| | OL | Cycle 1 | Subsequen | t OL Cycle | OL End of<br>Study/End of<br>Dosing (EOS) <sup>j</sup> | OL Follow-<br>up (28 ± 3 |
|---|---|---|---|---|---|---|
| Trial Procedures | Day 1<br>Baseline | Days 8 and 15<br>± 2 Days | Day 1<br>± 2 Days | Day 15<br>± 2 Days | Day 1<br>± 2 Days | Days Post<br>EOS) |
| Physical examination | $X^b$ | $X^{b}$ | $X^{b}$ | $X^b$ | $X^{a}$ | $X^{b}$ |
| Eligibility criteria for OL | X | | | | | |
| Informed consent for OL | X | | | | | |
| Body weight | X | | X | | X | X |
| Vital signs <sup>c</sup> | X | X | X | X | X | X |
| Clinical laboratory testing <sup>d</sup> | X | X | X | X | X | X |
| T3, T4, TSH | X | | X | | X | X |
| ECG <sup>e</sup> | X | X | X | X | X | X |
| Pregnancy test (serum) <sup>f</sup> | X | | X | | X | X |
| ECOG PS <sup>f</sup> | X | | X | | X | |
| α-fetoprotein (AFP) | X | | X | | X | X |
| WBC A <sub>3</sub> AR sample | X | | $X^g$ | | | |
| Hepatitis B/C viral load (if seropositive) | X | | $X^h$ | | $X^h$ | |
| Tumor imaging for RECIST | | | $X^{i}$ | | X | |
| Concomitant medications | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X |
| Dispense study drug supplies | X | | X | | | |
| Review treatment compliance | X | X | X | X | X | |

a. Complete PE performed at Open Label (OL) End of Study/OL End of Dosing (EOS) visits.

- b. Symptom-directed physical examination.
- c. Temperature, pulse, respiration, blood pressure performed at the following times: pre-dose at all visits; at 1, 2, 3, 4h ( $\pm$  5 min), 6h and 8h ( $\pm$  10 min) post-dose on OL Cycle 1 Day 1 and at OL Follow-up.
- d. See list of parameters in Appendix C.
- e. ECG at pre-dose at all visits; and at 2, 4, and 6h (± 10 min) post-dose on OL Cycle 1 Days 1 and 8; and at OL Follow-up.
- f. Performed pre-dose on Day 1 of each OL cycle, and at OL Follow-up.
- g. Day 1 of odd-numbered cycles, unless waived by the Sponsor (selected sites only).
- h. For subjects with measurable viral load at the Baseline Visit; on Day 1 of OL odd-numbered cycles only and at OL EOS.
- i. CT scan or MRI at the end of OL even-numbered cycles. If performed at +1 day after day 28, CT/MRI scan must be performed before administration of the morning dose of that day).
- j. End of Study OL visit timeframe is of 2 days since the last administered dose of IMP.

#### 6. STUDY ENDPOINTS

Baseline typically refers to Day 1 of Cycle 1 and Screening refers to the Pre-Study Visit. For some variables, Baseline is Cycle 1 Day 1 unless the assessment was performed at Screening which was  $\leq 3$  days prior to Cycle 1 Day 1, in which case the assessment was not to be repeated (footnotes 'a' and 'c' of <u>Table 1-1</u>). In the protocol and footnotes above, some assessments are given as performed at Day 28 or 29 of a cycle; consistent with the table above and the CRFs, these assessments are described below as being performed at Day 1 of the following cycle.

Tumor assessments performed at the End of Study/ End of Dosing (EOS) Visit, the Follow-up Visit, and Unscheduled Visits will be assigned to the next cycle for calculation of summary statistics.

The subjects who are still on blinded treatment when Amendment 5 is approved will be switched to open-label treatment at their next scheduled visit. The first day of open-label study drug dosing will be considered Day 1 (OL) of the trial. During this visit, the OL Cycle 1 Day 1 for OL procedures will be performed ( $\underline{\text{Table 1-2}}$ ). During the OL period, clinic visits will take place within  $\pm$  2 working days of the scheduled day; during these visits, assessments will be performed prior to administration of the study drug dose for that day.

#### 6.1 EFFICACY ASSESSMENTS

Tumor response will be assessed at the Pre-Study Visit, Day 1 of odd-numbered cycles, and at the follow-up visit using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) from Eisenhauer et al. (2009), presented in Appendix A of the protocol, and further described below in Appendix B. In general, target lesions will be assessed as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD) and non-target lesions will be assessed as Complete Response (CR), Incomplete Response/Stable Disease (SD), or Progressive Disease (PD). Tumor responses from target lesions and from non-target lesions will be used to determine Overall Response as described in Appendix B. If the Overall Response is CR or PR, tumor assessments are to be repeated within 4 weeks. Overall Response will be tabulated by cycle and treatment; the responses for target lesions and non-target lesions will be included in listings, but will not be tabulated. If Overall Response of PD is observed at any time, the patient will not automatically be discontinued. Further imaging or target lesion measurements will not be required and all other trial visits and procedures will continue.

If assessments are made after the Overall Response of PD is recorded, then the Overall Response at all subsequent cycles will be PD and will be included at every cycle for which the Overall Response is recorded through Cycle 11 (see Section 7.2).

#### **6.1.1** TIME TO EVENT ENDPOINTS

The primary efficacy endpoint is Overall Survival (OS), the time from Baseline to death due to any cause, calculated as date of death- date of Cycle 1 Day 1+1. Secondary time-to-event endpoints are:

- TTP: the time from Baseline to the first Overall Response of PD, calculated as date of first PD date of Cycle 1 Day 1+1, and
- PFS: the time from Baseline to the first Overall Response of PD or death due to any cause if the subject dies without experiencing PD, calculated as date of first PD or death date of Cycle 1 Day 1+1.

#### **6.1.2** TUMOR RESPONSE

The secondary endpoints which are based directly on tumor response are:

- ORR (OR Rate): proportion of subjects who have CR or PR,
- DCR (DC Rate): proportion of subjects who have CR, PR, or SD, and
- Best Overall Response during the duration of the study.
   (The best overall response for each subject is the best response recorded from the start of the study treatment until the end of study, in the order of CR, PR, SD, or PD from best to worst.)

#### **6.1.3** EXPLORATORY EFFICACY

Laboratory parameters associated with hepatic dysfunction and cirrhosis (ALT, AST, bilirubin, and albumin levels, prothrombin time (PT), and International Normalized Ratio (INR)) will be assessed every cycle and will be considered exploratory efficacy variables.

The effect of CF102 on  $\alpha$ -fetoprotein (alpha-fetoprotein; AFP) will be assessed. AFP levels will be assessed at Baseline and on Day 1 of each subsequent cycle.

Liver chemistry tests and viral load will be presented as exploratory efficacy variables, as will WBC A<sub>3</sub>AR expression. Viral load for Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) will be assessed at Baseline, at Day 1 of each subsequent odd cycle, at the end of dosing, and at the Follow-up visit for subjects with positive serology at Screening.

#### **6.2 SAFETY EVALUATIONS**

Safety parameters assessed throughout the trial include adverse events, ECOG performance status, vital signs, weight, physical examinations, laboratory parameters including thyroid functions, ECG, and concomitant medications. Any clinically significant change from baseline in a laboratory parameter will be reported as an AE. Liver chemistry tests and viral load will be presented as exploratory efficacy variables.

At each visit, all AEs will be recorded in the appropriate section of the CRF and will be evaluated by the Investigator. The minimum information required for each AE includes the following:

- Type of event
- Duration (start and end dates)
- Severity
- Seriousness
- Relationship to study drug (Unrelated, Possibly Related, Probably Related, or Related)
- Action taken
- Outcome.

In most cases, the CTCAE v4.0 criteria will preferably be used to grade severity; however, if an AE is not listed in the CTCAE, the following grading scale may be used: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3), Life-Threatening (Grade 4), or Fatal (Grade 5).

#### 7. STATISTICAL CONSIDERATIONS AND DATA ANALYSIS

Tables and data listings will be prepared using SAS Version 9.0 or higher. A subject's Baseline value for a specified variable will be the measurement for that variable taken on Day 1 of Cycle 1, unless the pre-study assessment was performed within 3 days prior to baseline. In the latter case, assessments do not need to be repeated prior to initiation of dosing for Physical Examination, Body Weight, Clinical Laboratory testing, Pregnancy Test, and ECOG PS, as noted in the Schedule of Procedures in Section 5 and the Baseline value will be the value at Screening.

For any variable with Change From Baseline (CFB) calculated, CFB will be calculated as CFB = Value at Post-Baseline visit – Value at Baseline.

If the final pre-treatment assessment was performed at Screening, prior to Baseline, then CFB is defined as the difference between the value at the post-Baseline visit and the value at Screening.

Simple descriptive statistics for continuous data are: n (number of non-missing observations), mean, standard deviation, maximum, median, and minimum. Categorical data will be summarized by the number and percentage of subjects in each category. The data will be summarized upon completion of the final subject. All data collected for the OL period will be listed and select variables will be summarized. Listings and summaries for the OL period will be presented separately and a separate SAP will be prepared. The following pertains to the analyses and summaries for the DB period.

#### 7.1 ANALYSIS POPULATIONS

Analyses will be conducted using the populations described below.

The **Safety Population** consists of all subjects who received at least one dose of study medication. Analyses of safety assessments will be performed using the Safety Population.

The **Intent-To-Treat (ITT) Population** is defined as all subjects in the Safety Population with any post-Baseline assessment recorded. Exclusion of subjects from the ITT Population will be determined prior to unblinding. All efficacy analyses will be performed using the ITT Population.

The **Per Protocol (PP) Population** is defined as all subjects in the ITT Population with no major protocol deviations, including major violations of inclusion and exclusion criteria and violation of RECIST requirements regarding the number of target lesions at Screening (<u>Appendix B</u>). Exclusion of subjects from the PP Population will be determined prior to unblinding. Tumor response (Sections <u>6.1.2</u> and <u>7.6.4</u>) will be analyzed for the PP Population.

#### 7.2 GENERAL ANALYSIS

The following standards will be applied for analyses unless otherwise specified. Simple descriptive statistics for continuous data are: n (number of non-missing observations), mean, standard deviation, maximum, median, and minimum. Categorical data will be summarized by the number and percentage of subjects in each category. Summaries of efficacy variables will be presented by visit through end of Cycle 11. Best Overall Response will be summarized once for the entire study. All data will be listed for the Safety Population, sorted by investigator number, subject number and, where appropriate, by visit, including data from visits after Cycle 11. The choice of Cycle 11 as the final time for tabulation will be finalized prior to unblinding. Tumor assessments performed at the EOS Visit, the Follow-up Visit, and Unscheduled Visits will be assigned to the next cycle and will be analyzed with that cycle. Tumor responses recorded on the CRF will be listed. Other data from Unscheduled Visits will not be summarized, except for AEs.

#### 7.3 SUBJECT DISPOSITION

The total number of subjects will be presented with the number and percentage of subjects in each analysis population by treatment and overall. The number and percentage of subjects who completed the study, who discontinued, and primary reason for discontinuation will be summarized by treatment for the Safety Population.

#### 7.4 DEMOGRAPHICS AND MEDICAL HISTORY

#### 7.4.1 DEMOGRAPHICS

Demographic parameters, including age, sex, and origin, will be summarized for the Safety Population by treatment and overall. Age will be computed as (the number of days from Date of Birth to Date of Screening Visit)/365.25. After unblinding, it was decided to include the frequency distribution of Child-Pugh (CP) Score at Screening (7, 8, or 9) in the table of demographics and baseline characteristics. The CP Score for Subject 311-003 was recorded as 6, but this was corrected to 7 after unblinding.

#### 7.4.2 HCC DISEASE HISTORY AND PRIOR THERAPIES

HCC disease history includes

- date of initial HCC diagnosis and staging,
- date of most recent relapse and/or re-staging,
- method used for diagnosis (histology / cytology or American Association for the Study of Liver Diseases (AASLD) Practice Guideline algorithm),
- history of viral hepatitis, including date of diagnosis,
- hepatitis B and hepatitis C virus serology (positive or negative), with the last date of testing, and
- known complication(s) of cirrhosis and/or portal hypertension.

History of viral hepatitis is recorded as "Yes, Hepatitis B"; "Yes, Hepatitis C"; "No"; or "Not known", with the date of diagnosis recorded for the first two responses, both of which are possible. The summary statistics will include the counts and percentages for each of the four possible responses by treatment for the Safety Population.

Known complication(s) of cirrhosis and/or portal hypertension are reported on the CRF as "Ascites", "Esophageal varices with bleeding", or "Other (specify)". If none of these responses are selected, then the response should be reported as "None".

Prior therapies include

- modality,
- start and stop dates of treatments,
- numbers of cycles, and
- best response to each treatment.

The number of subjects reporting the use of a modality at least once will be summarized by treatment for the Safety Population. Other variables pertaining to HCC disease history and prior therapies will be listed for the Safety Population.

A table of the number of target hepatic lesions and the number of target non-hepatic lesions (Appendix B) at Screening for the Safety Population will be presented.

A table of the incidence of Extrahepatic Spread (EHS), Portal Vein Thrombosis (PVT) at Baseline, including either EHS or PVT ("Yes" or "No"), will be provided.

#### 7.4.3 MEDICAL HISTORY

Medical history, excluding past HCC, cirrhosis, and viral hepatitis-related history, will be summarized using frequencies and percentages of subjects with a finding or procedure for each body system (or "None") by treatment for the Safety Population by treatment and overall. "Other" will be listed but will not be included in the summaries.

#### 7.5 MEDICATION AND TREATMENT ANALYSIS

#### 7.5.1 COMPLIANCE AND EXPOSURE

Compliance will be calculated as the number of total capsules dispensed (over the duration of the study) minus the total number of capsules returned, and then that quantity is divided by twice the duration of treatment in days. The duration of treatment is date of final dose minus date of Baseline + 1. If the date of final dose is missing or if the subject is still receiving treatment, the date of final dose will be imputed as described in Section 8. Descriptive statistics for compliance and the duration of treatment will be provided for the Safety Population by treatment. The summary statistics pooled across treatments will also be computed for duration of treatment, to be used in efficacy evaluations as described in Sections 7.6.1-7.6.3.

#### 7.5.2 CONCOMITANT MEDICATIONS

Concomitant and prior medications taken within 30 days prior to Screening Visit will be summarized by ATC Level 3.

#### 7.6 EFFICACY

Efficacy will be assessed using the response based upon overall survival, time to progression, RECIST, and hepatitis viral load. Liver chemistry tests and viral load will be presented as exploratory efficacy variables, as will AFP and WBC A<sub>3</sub>AR expression. Summaries of efficacy variables by visit will be presented using visits through end of Cycle 11. Analyses of time to event (OS, TTP, and PFS) and Best Overall Response will not be restricted to visits through Cycle 11. All efficacy data will be listed. Binary response variables will not be analyzed using SAS PROC FREQ, which uses equal variances for the differences, as opposed to the unequal variances given below.

## 7.6.1 OVERALL SURVIVAL (OS)

Overall survival (OS) is the time from Baseline to death due to any cause. OS will be summarized in months, which will be obtained by dividing OS in days by 30 days/month. Subjects who are alive at last contact will be considered censored at the date of last contact. Summary statistics (25<sup>th</sup> percentile, median, and 75<sup>th</sup> percentile) will be determined using the Kaplan-Meier (KM) estimate of the survival function. These summary statistics will be listed to one decimal place, rounded down such as the SAS FLOOR function. The KM curve for OS will be presented. The value of the KM curve for OS at the median duration of therapy (Section 7.5.1) will be presented. The between-treatment comparison will be performed using the logrank test as the primary analysis. Between-treatment comparisons with respect to OS will be also performed using the proportional hazards model with AFP at Baseline and A<sub>3</sub>AR level at Baseline as covariates individually as secondary analyses, including the hazard ratio and the 95% confidence interval for the hazard ratios for both treatment and the covariate. Additional details are given in Section 9.

## 7.6.2 TIME TO PROGRESSION (TTP)

Time to Progression (TTP) is the time from Baseline to the first Overall Response of Progressive Disease (PD), computed as in Section 6.1.1. TTP will be summarized in months, which will be obtained by dividing TTP in days by 30 days/month. Subjects who do not have an Overall Response of PD by the time of last contact will be considered censored at the date of last contact; subjects who died without experiencing PD will be censored at the day of death. Summary statistics (25<sup>th</sup> percentile, median, and 75<sup>th</sup> percentile) will be determined using the KM estimate of the survival function for TTP. These summary statistics will be listed to one decimal place, rounded down such as the SAS FLOOR function. The KM curve for TTP will be presented. The value of the KM curve for TTP at the median duration of therapy (Section 7.5.1) will be presented. The between-treatment comparison will be performed using the logrank test. Additional details are given in Section 9.

# 7.6.3 PROGRESSION-FREE SURVIVAL (PFS)

Progression-free Survival (PFS) is the time from Baseline to the first Overall Response of Progressive Disease (PD) or death due to any cause if the subject dies without experiencing PD, computed as in Section 6.1.1. PFS will be summarized in months, which will be obtained by dividing PFS in days by 30 days/month. Subjects who are alive without experiencing an Overall Response of PD at the time of last contact will be considered censored at the date of last contact. Summary statistics (25<sup>th</sup> percentile, median, and 75<sup>th</sup> percentile) will be determined using the KM estimate of the survival function for PFS. These summary statistics will be listed to one decimal place, rounded down such as the SAS FLOOR function. The KM curve for PFS will be presented. The value of the KM curve for PFS at the median duration of therapy (Section 7.5.1) will be presented. The between-treatment comparison will be performed using the logrank test. Additional details are given in Section 9.

#### 7.6.4 TUMOR RESPONSE

The Objective Response Rate (ORR) is the percentage of subjects who achieved either CR or PR. ORR will be summarized using counts and percentages for the ITT Population by treatment and cycle. The between-treatment comparison will be performed using the normal approximation to the binomial distribution (NAB) with unequal variances, as follows.

For each cycle, let  $p_{CF}$  and  $p_0$  denote the proportions of subjects who experienced CR or PR based on  $n_{CF}$  and  $n_0$  subjects for CF102 and Placebo, respectively, and let

 $Z=(p_{CF}-p_0)/(p_{CF}(1-p_{CF})/n_{CF}+p_0(1-p_0)/n_0)^{1/2}$ .

Then the corresponding p-value is p=2\*(1-PROBNORM(ABS(Z))).

The Disease Control Rate (DCR) is the percentage of subjects who achieved either CR, PR, or SD. DCR will be summarized using counts and percentages for the ITT Population by treatment and cycle. The between-treatment comparison will be performed using the (NAB), similar to that for ORR.

For each subject, the Best Overall Response during the duration of the study will be determined and will be summarized using counts and percentages for the ITT Population by treatment. The between-treatment comparison will be performed using the NAB, for both the percentage of subjects who achieved either CR or PR (similar to ORR) and the percentage of subjects who achieved either CR, PR, or SD (similar to DCR).

#### 7.6.5 BIOMARKERS

The biomarker α-fetoprotein (AFP) will be assessed at Baseline, at Day 1 of each cycle, and at the follow-up visit. Summary statistics for AFP levels and CFB in AFP levels will be provided for the ITT Population by treatment and visit. Between-treatment comparisons will be performed by visit using Analysis of Covariance (ANCOVA) with CFB as the dependent variable and Baseline as the covariate. Summary statistics for AFP and CFB in AFP will be provided for each level of Overall Response for the ITT Population by treatment. Distribution of Overall Response will be presented for subjects with AFP levels <20, 20-200, or >200 ng/mL and for subjects with AFP levels above or at most the pooled median by treatment and cycle; the percentages will be calculated using number of subjects within each category defined by AFP levels as the denominator for each treatment.

WBC A<sub>3</sub>AR expression will be assessed at Baseline and at Day 1 of each odd-numbered cycle. Summary statistics for WBC A<sub>3</sub>AR expression and CFB in WBC A<sub>3</sub>AR expression will be provided for the ITT Population by treatment and visit. Summary statistics for CFB in WBC A<sub>3</sub>AR expression will be provided for each level of Overall Response for the ITT Population by treatment. To assess the relationship between Overall Response and changes in WBC A<sub>3</sub>AR at each visit, the distribution of Overall Response will be presented for subjects with WBC A<sub>3</sub>AR less than the pooled median and for subjects with WBC A<sub>3</sub>AR at least the pooled median at each post-baseline visit.

#### 7.6.6 CHEMISTRY AND COAGULATION PARAMETERS

The following laboratory parameters will be examined as exploratory efficacy variables:

- alanine aminotransferase (ALT)
- albumin
- aspartate aminotransferase (AST)
- bilirubin (direct and total)
- International Normalized Ratio (INR)
- prothrombin time (PT).

The above variables and CFB for each variable will be summarized by treatment and visit for the ITT Population. Between-treatment comparisons will be performed by visit using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate. These variables will be listed for the Safety Population with the other laboratory parameters.

#### 7.6.7 HEPATITIS VIRAL LOAD

Viral load for Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) for subjects with positive serology at Screening will be summarized using summary statistics for log-transformed values using the base 10 logarithm, which will be presented by treatment and visit for the ITT Population. Between-treatment comparisons will be performed by visit using ANCOVA with CFB for log-transformed values as the dependent variable and Baseline as the covariate. These variables (viral load (IU/mL) and log-transformed viral load) will be listed for the Safety Population. Any viral load recorded for subjects who do not have positive serology at Screening will not be included in tables but will be included in listings only.

#### 7.6.8 SUBGROUP ANALYSES

After unblinding, it was decided to perform various subgroup analyses of OS. The subgroup analyses will be performed by the following assessments at Screening or Baseline:

CP Score at Screening (7, 8, 7+8, or 9), Sex, ECOG PS at Screening (0 or 1+2).

AFP (≤400 ng/mL or >400 ng/mL) at Baseline,

Prior Locoregional therapy (HCC Prior Therapies of Radiation or

Chemoembolization =Yes, Otherwise =No),

EHS (Yes or No), PVT (Yes or No), and Either EHS or PVT (Yes or No),

History of HBV (Known history of HBV=Yes or No),

History of HCV (Known history of HCV=Yes or No),

Diagnostic Procedure (Cytology/histology or AASLD), and

Country (based on the first digit of the site number, given as Bulgaria=1, Serbia=2, Israel=3, Romania=5, or United States=7).

The subgroup analyses will be performed as univariate analyses within each level of the corresponding subgrouping variable. For each subgrouping variable, the between-treatment comparisons will be performed using the logrank test (Section 7.6.1). Each analysis will include the hazard ratio with the corresponding 95% confidence interval from proportional hazards model with no additional covariates and the p-value (Chi-Square), as described in Section 9. The subgroup analyses do not include a plot of each KM curve, except for the analyses by CP Score at Screening (CP=7, CP=8, or CP=7 or 8), and do not include the value of the KM curve at the median duration of therapy, provided in the analyses for the ITT Population.

History of viral hepatitis is recorded as "Yes, Hepatitis B"; "Yes, Hepatitis C"; "No"; or "Not known", with the date of diagnosis recorded for the first two responses, both of which are possible. If both of these responses are recorded, then the response for both History of HBV and History of HCV will be considered "Yes". Subjects with responses of "Not known" will be excluded from the subgroup analyses using history of viral hepatitis.

Subgroup analyses for other time-to-event variables or tumor response variables may be presented as further exploratory analyses after review.

#### 7.7 SAFETY ANALYSES

Safety data consist of adverse events (AEs), laboratory tests including thyroid functions, vital signs and weight, and physical examinations. Summaries of safety data will be conducted on all subjects in the Safety Population. Missing safety data will not be imputed. Summaries of all safety variables by visit will be presented for visits at which there are at least 4 subjects in either treatment group. Summaries of AEs, deaths, SAEs, and Discontinuation due to AE will not be restricted to visits with at least 4 subjects in either treatment group. All safety data will be listed.

#### 7.7.1 ADVERSE EVENTS

The original reported (verbatim) terms used by the Investigator to identify adverse events in the CRFs will be entered into the database and coded by Preferred Term using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary (MedDRA MSSO, Reston, Virginia USA). Adverse events will then be grouped by MedDRA Preferred Term (PT) into frequency tables according to System Organ Classification (SOC).

An adverse event that started during the treatment period (on or after the day of the baseline visit) or that was present at Baseline and increased in severity during the treatment period will be considered a treatment-emergent adverse event (TEAE). Events ending prior to the day of the baseline visit and events present at Baseline that do not increase in severity during treatment will be considered as Baseline adverse events and will not be included in the presentation of TEAEs. If the date of a new AE does not allow for determination of whether the AE is treatment emergent, it will be assumed to be a TEAE.

The number and percentage of subjects experiencing TEAEs will be presented for the Safety Population for each body system and preferred term by treatment, and for each severity and relationship to study medication. When an adverse event occurs more than once, the maximum severity grade and relationship will be counted. For severity, only "Mild" and "Moderate" will be included for all SOCs and PTs; "Severe", "Life-Threatening", or "Fatal" will be included for SOCs and PTs only when such are recorded for severity. Similarly, only "Possibly Related" and "Not Related" will be included for all SOCs and PTs; "Definitely Related" and "Probably Related" will be included for SOCs and PTs when such are recorded for relationship.

Serious adverse events and discontinuations due to an adverse event will be provided in separate listings for the Safety Population. Each serious adverse event (SAE) will be listed for subjects in the Safety Population.

#### 7.7.2 LABORATORY TESTS

Laboratory tests (hematology, clinical chemistry, coagulation, urinalysis, and thyroid functions) will be performed at the timepoints specified in Appendix C, which also contains a complete list of all clinical laboratory tests. Clinical laboratory evaluations and CFB for each laboratory value will be listed and summarized using descriptive statistics by treatment and visit for visits with at least 4 subjects in either treatment group for the Safety Population. If a laboratory test is repeated during a visit, only the first values will be included in the summary; all values will be included in the listings. Clinically significant (CS) out-of-range laboratory values should be recorded as AEs. ALT (Alanine Aminotransferase; SGPT) and AST (Aspartate Aminotransferase; SGOT) are referred to as ALAT (SGPT) and ASAT (SGOT), respectively, in the listing of Blood Chemistry parameters. Urinalysis laboratory values will be listed only and CFB will not be computed. Laboratory assessments that are considered exploratory efficacy variables (Section 7.6.7) will be presented both as efficacy variables and laboratory variables, through Cycle 11 when considered exploratory efficacy variables and for all visits when considered safety variables.

#### 7.7.3 ECOG PERFORMANCE STATUS

ECOG Performance Status (PS) is an assessment using a five-point scale, with 0= Normal activity,..., 5=100 % bedridden; details are given in <u>Appendix D</u>. ECOG PS will be recorded at Pre-study visit, Day 1 of Cycle 1 (Baseline), Day 1 of each subsequent cycle, and at Follow-up. ECOG PS and categories of CFB in ECOG PS (decreased, no change, increased) will be presented for the Safety Population by treatment and cycle for cycles with at least 4 subjects in either treatment group.

#### 7.7.4 VITAL SIGNS AND WEIGHT

Vital signs will be recorded at Days 1 and 15 of each cycle, Day 8 of Cycle 1, Hours 1, 2, 3, 4, 6 and 8 on Cycle 1 Day 1, and at Follow-up. Systolic blood pressure (mmHg), diastolic blood pressure (mmHg), respiratory rate (breaths/min), pulse (beats/min), oral temperature (degrees C), and CFB for each of these vital signs will be listed and summarized using descriptive statistics for the Safety Population by treatment and visit for visits with at least 4 subjects in either treatment group. Height (cm) will be recorded at the Pre-Study Visit only and will be included in listings only. Body weight (kg) will be recorded at Days 1 and 15 of each cycle, Day 8 of Cycle 1, and at Follow-up; BMI (kg/m²) will be computed for each of these visits using the height recorded at the Pre-Study Visit.

#### 7.7.5 ECG PARAMETERS

A resting 12-lead electrocardiogram (ECG) will be performed at the Pre-Study visit, Days 1 and 15 of all cycles, Day 8 of Cycle 1, and at 2, 4, and 6 hours post-dose on Day 1 of Cycle 1, and at Follow-up. ECG interval data (Heart Rate [HR], PR, QRS, QT) and the corresponding CFBs will be listed and summarized using descriptive statistics for the Safety Population by treatment and visit for visits with at least 4 subjects in either group. OTc will be computed using Fridericia's treatment QTcF=QT\*(HR/60)<sup>1/3</sup>. QT will not be summarized and will be included in the listing only. ST Segment (normal or abnormal), Cardiac Rhythm (normal or abnormal), and Overall Impression (normal, abnormal- NCS, or abnormal- CS) will be summarized using counts and percentages for the Safety Population by treatment and visit.

#### 7.7.6 PHYSICAL EXAMINATIONS

A physical examination (PE) will be performed at every visit. A complete PE will be performed at the Pre-Study, Cycle 1 Day 1 (the Baseline Visit if the Pre-Study visit not performed within 3 days prior), and End of Study/End of Dosing (EOS) visits, including a thorough review of all body systems (general appearance, head/neck, ears/nose/throat, skin, chest/lungs, heart, abdomen, genitourinary, extremities, musculoskeletal, lymph nodes, neurological and other, specify) as well as measurement of weight (kg) and height (cm). At all other visits, a symptom-directed PE, including weight (kg), will be performed. If the Pre-Study visit is within 3 days of Cycle 1 Day 1, then no responses should be reported for Cycle 1 Day 1.

At the Pre-Study visit, each body system, including "Other" (specify) if appropriate, will be assessed (Normal, Abnormal, or Not Done). At each visit after the Pre-Study visit, assessments will be recorded for any body systems with clinically significant (CS) changes from the PE conducted at the previous assessment (Normal, Abnormal, or Not Done), with details. The CRF indicates that these assessments should be recorded if the body system with a clinically significant change from the PE conducted at the previous assessment is "Abnormal", with a description of the abnormality; these assessments should be recorded for any CS change from the previous PE, not just "Abnormal", including a CS change from "Abnormal" to "Normal".

Assessments at the Pre-Study visit will be summarized by body system (Normal or Abnormal). Any subject with more than one assessment of "Other" will be counted once. Assessments recorded as "Not Done" will not be included in the table. Any description of an abnormality will be included in the corresponding listing. At each visit after the Pre-Study visit, the number of subjects with at least one CS change from the PE conducted at the previous assessment will be summarized for the Safety Population by treatment and visit for visits with at least 4 subjects in either treatment group. Any body systems with a CS change from the PE conducted at the previous assessment will be included in the corresponding listing with the result and description.

#### 8. MISSING DATA

Missing dates will be imputed only when the date is required to calculate the duration of an event for summary. As such, the only missing date that would need to be imputed is the date of final dose, required for calculation of duration of treatment. In such situations, the month and year would be recorded. For subjects who have completed dosing, the missing date of final dose will be imputed as the 15-th of the month; for subjects who are still receiving treatment, the missing date of final dose will be imputed as the date of the last completed visit.

Missing data from intermediate visits for AFP, WBC A3AR, viral load, and laboratory assessments when considered exploratory efficacy variables will be imputed using Last Observation Carried Forward (LOCF). Missing data for the latter laboratory variables will not be imputed when examined with laboratory assessments as safety variables. Due to the nature of the study, there is no imputation due to discontinuation.

The protocol specifies that certain assessments will not be repeated at Baseline (Cycle 1 Day 1) if assessed at the Pre-Study visit <= 3 days prior to Cycle 1 Day 1, resulting in missing values for Baseline; in such cases, the missing value at Baseline will be imputed by the value from the Pre-Study visit.

#### 9. DIFFERENCES AND CHANGES FROM THE PROTOCOL

The protocol states that disease history includes duration of prior sorafenib therapy, reason(s) for discontinuation of sorafenib, and if applicable, nature of intolerability to sorafenib. The duration is not directly collected, but can be computed from the start and stop dates, as provided for all prior HCC therapies. The reasons(s) for discontinuation, including nature of intolerability, were not collected for prior HCC therapies, including sorafenib.

The protocol states that the listing of "dosing interruptions and dose reductions" will be provided. This listing is not provided, as these data were not specifically recorded, but are available as the "Action Taken" for AEs.

In the protocol, ITT Population is defined as "all subjects in the Safety Population who have any post-Baseline efficacy data, including Liver Chemistry Tests and/or INR on Day 8 of Cycle 1, or death or discontinuation due to disease progression at any time." According to SAP, ITT Population "is defined as all subjects in the Safety Population with any post-Baseline assessment recorded". The difference has no impact, especially since no subjects were excluded from the ITT Population.

Summaries of all safety variables by visit will be presented for visits at which there are at least 4 subjects in either treatment group. AEs, deaths, SAEs, and Discontinuation due to AE are not subject to this constraint. This restriction was not given in the protocol.

Summaries and analyses of efficacy variables by visit will be presented using visits through end of Cycle 11. Analyses of time to event (OS, TTP, and PFS) and Best Overall Response will not be restricted to visits through Cycle 11. This restriction was not given in the protocol.

Analyses of time to event (OS, TTP, and PFS) originally included summary statistics (25th percentile, median, and 75th percentile) from the KM estimate of the survival function and the value of the KM curve at the median duration of therapy. The between-treatment comparisons were performed using the logrank test. After unblinding, it was decided to include the hazard ratio with the corresponding 95% confidence interval from proportional hazards model with no additional covariates and the p-value (Chi-Square). The subgroup analyses of OS (Section 7.6.8) were not presented in the protocol.

After unblinding, it was decided to present incidence of EHS and PVT at Baseline (Section 7.4.2), which are not given in the protocol.

Any changes not presented in this or any subsequent version of the SAP will be described in the clinical study report.

#### 10. APPENDICES

# 10.1 APPENDIX A – CHILD-PUGH CLASSIFICATION OF SEVERITY OF LIVER DISEASE

Child-Pugh classification of severity of liver disease is defined using the degree of ascites, plasma concentrations of bilirubin and albumin, prothrombin time, and the degree of encephalopathy.

Class A (well-compensated disease): total score of 5-6.

Class B (significant functional compromise): total score of 7-9.

Class C (decompensated disease): total score of 10-15.

| <b>D</b> | Points Assigned | | |
|------------------------|-----------------|-----------|-----------|
| Parameter – | 1 | 2 | 3 |
| Ascites | Absent | Slight | Moderate |
| Bilirubin, mg/dL | <2 | 2-3 | >3 |
| Albumin, g/dL | >3.5 | 2.8-3.5 | <2.8 |
| Prothrombin time | | | |
| * Seconds over control | 1-3 | 4-6 | >6 |
| * INR | <1.7 | 1.7-2.3 | >2.3 |
| Encephalopathy | None | Grade 1-2 | Grade 3-4 |

| Parameter | 1 | 2 | 3 |
|--------------------------|-----|-------|-----|
| Total bilirubin (µmol/L) | <34 | 34-50 | >50 |
| Albumin (g/L) | >35 | 28-35 | <28 |

# 10.2 APPENDIX B – DETERMINATION OF OVERALL RESPONSE

Tumor status will be assessed at the Pre-Study Visit, Day 1 of odd-numbered cycles, and at the follow-up visit using Response Evaluation Criteria In Solid Tumors (RECIST), as presented in Appendix A of the protocol. The protocol states that tumor status will be assessed "at baseline and every 8 weeks thereafter (i.e., at the end of even-numbered cycles) by computed tomography (CT) scan or magnetic resonance imaging (MRI)"; however, the "baseline" assessment is performed at the Pre-Study Visit and the assessments of tumor status are recorded on CRF for Day 1 of odd-numbered cycles.

Details regarding the calculation of Overall Response, and related variables, are presented here. The following details are from RECIST v1.1 (Eisenhauer et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). *European J Cancer*. 45(2009): 228-247), the subsequent modification (Santoro et al. Tivantinib for second-line treatment of advanced hepatocellular carcinoma: a randomized, placebo-controlled phase 2 study. *Lancet Oncol*. 2013; 14: 55-63), and the protocol.

At Screening, target lesions are assessed: Up to 5 liver lesions and up to 2 lesions from other organs that can be accurately measured in at least one dimension with longest diameter  $\geq 20$  mm using conventional techniques (CT scan or MRI) or  $\geq 10$  mm with spiral CT scan. The LD for each target lesion should be compared to these minima, and any discrepancies noted for investigation and possible query. Lesions with LD less than these values and lesions from various sites which are "truly non-measurable" (Eisenhauer et al, 2009) are assessed as non-target lesions.

#### Target Lesions

The lesions identified at Screening as "Target Lesions" will be measured and the longest diameter (LD) of each target lesion is recorded, as well as the sum of the longest diameters. The sum of the longest diameters is recorded on CRF but should be recomputed for accuracy; any discrepancy between this calculated value and the recorded sum will be noted for investigation and possible query, except in the case of minor round-off discrepancies. In the latter case, the recorded value will be presented in the listings, but the calculated value will be used for all subsequent calculations. At each visit after Screening, the LDs for target lesions identified at Screening will be assessed; any new lesions will be recorded as such with "Non-Target Lesions" and discussed below.

Listing 16.2.6.1.1 (Tumor Evaluations: Target Lesions) is the listing of assessment (LD) for each target lesion by subject and visit. Listing 16.2.6.1.2 (Summary of Target Lesions) is the listing of "Sum of Longest Diameters (mm), Smallest Sum On Study (mm), Percent Change from Smallest, Screening Sum on study, and Percent Change From Screening" by subject and visit for target lesions. These variables are recorded on CRF, but should be determined from the individual assessments reported in Listing 16.2.6.1.1 as a check on accuracy. Inconsistencies, other than minor round-off, should be investigated. Percent Change from Smallest and Percent Change From Screening will be listed to one decimal place.

Based on results given in Listing 16.2.6.1.2, Response for Target Lesions can be determined as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD) according to the following algorithm (from CRF).

Pick the one response that applies from most recent assessment for Target Lesions:

| Complete Response (CR) | Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. |
|---|---|
| Partial Response (PR) | At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. |
| Progressive Disease (PD) | At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progression. |
| Stable Disease (SD) | Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. |

Note that CR and PR are assessed relative to the baseline sum of diameters, whereas PD is assessed relative to the smallest sum of diameters. Note that "smallest sum on study" at any visit refers to sums prior to, and including, the visit of interest, including the baseline sum of diameters.

Prior to unblinding, it was decided that subjects who can be assigned both PR and PD for target lesions at a cycle will be assigned PR. This will occur at a cycle whenever  $1.2*(Smallest Sum of LDs) \le Sum of LDs$  at Cycle  $\le 0.7*(Sum of LDs)$  at Screening). For Subject 530-006 at Cycle 13, the Investigator recorded the response as PD and chose not to change the recorded response; both responses are provided in listings.

#### Non-Target Lesions

Listing 16.2.6.2 (Tumor Evaluations: Non-Target Lesions) is listing of status (Present, Absent, New, Progressive) for each non-target lesion by subject and visit. Based on results given in Listing 16.2.6.2, Response for Non-Target Lesions can be determined as Complete Response (CR), Non-CR/ Non-PD, or Progressive Disease (PD) according to the following algorithm (from CRF). The assessment also allows for "not evaluated".

| Pick the one response that | t annlies from most recent | t assessment for Non-Target Lesions: |
|---|---|---|
| I ICK the one response that | abblics if the most iccent | i assessinent ivi iivii-i aizet Lesiviis. |

| C1-4- D (CD). | Di |
|---|---|
| Complete Response (CR): | Disappearance of all non-target lesions and normalization |
| | of tumor marker level. All lymph nodes must be non- |
| | pathological in size (< 10 mm short axis). Note: If tumor |
| | markers are initially above the upper normal limit, they |
| | must normalize for a patient to be considered in complete |
| | clinical response. |
| Non-CR/ Non-PD: | Persistence of one or more non-target lesions(s) or/and |
| | maintenance of tumor marker level above the normal limits. |
| Progressive Disease (PD): | Appearance of one or more new lesions and/or unequivocal |
| | progression of existing non-target lesions. Unequivocal |
| | progression should not normally trump target lesion status. |
| | It must be representative of overall disease status change, |
| | not a single lesion increase. |

Listing 16.2.6.3 (Tumor Response) includes Response for Target Lesions (based on results in Listing 16.2.6.1.2 and the above algorithm), Response for Non-Target Lesions (based on results in Listing 16.2.6.2 and the above algorithm), Overall Response, and Best Response. Overall Response is based on the Response for Target Lesions and the Response for Non-Target Lesions, according to the following algorithms, depending on whether subject has measurable disease or non-target lesions only.

| Overall Response - For Patients with Measurable Disease (i.e., Target Disease) | | | |
|---|---|---|---|
| <b>Target Lesions</b> | Non-Target Lesions | New<br>Lesions | Overall Response |
| CR | CR | No | CR |
| CR | Non-CR/Non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-CR/Non-PD/not evaluated | No | PR |
| SD | Non-CR/Non-PD/not evaluated | No | SD |
| PD | Any | Yes or No | PD |
| Any | PD* | Yes or No | PD |
| Any | Any | Yes | PD |
| *In avacational singulations are property and a property of the state | | | |

<sup>\*</sup>In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression

Note that this differs from the CRF; the corrections are given by the italicized entries. If Response for Non-Target Lesions='CR' or if there are no non-target lesions, then the Overall Response will be equal to the Response for Target Lesions.

| Overall Response -For Patients with Non-Measurable Disease (i.e., Non-Target Disease) | | |
|---|---|---|
| Non-Target Lesion | New Lesions | Overall Response |
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD * |
| Not all evaluated | No | Not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

<sup>\* &#</sup>x27;Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as an endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised.

Using the above tables, the overall response, given in Listing 16.2.6.3 is:

Complete Response (CR),

Partial Response (PR),

Progressive Disease (PD),

Stable Disease (SD),

Non-CR/non-PD, or

Unable to evaluate (NE) (with Comment).

Analyses are based on these variables from Listing 16.2.6.3. Although these variables are recorded on the CRF, the algorithms should be programmed as a check on accuracy. Inconsistencies would be investigated.

Other variables to be analyzed are

ORR (OR Rate) = proportion of subjects who have CR or PR,

DCR (DC Rate) = proportion of subjects who have CR, PR, or SD.

Theses variables, ORR and DCR, are analyzed by visit and are also included in Listing 16.2.6.3.
## 10.3 APPENDIX C – CLINICAL LABORATORY TESTS

Except for the "OTHER" category, the following laboratory tests will be performed at Pre-Study Visit; Days 1 (i.e., the Baseline Visit if not performed  $\leq$  3 days prior), 8, and 15 of Cycle 1; Days 1 and 15 of subsequent cycles; EOS; and Follow-Up.

| HEMATOLOGY TESTS | CHEMISTRY TESTS |
|---|---|
| <ul> <li>hematocrit</li> <li>hemoglobin</li> <li>platelet count</li> <li>red blood cell count and differential (absolute and percentage); neutrophils, lymphocytes, monocytes, eosinophils, basophils, and reticulocyte count</li> <li>URINALYSIS</li> <li>glucose</li> <li>ketones</li> <li>occult blood</li> <li>pH</li> <li>protein</li> <li>specific gravity</li> <li>and, when indicated by dipstick abnormality, microscopic sediment evaluation</li> </ul> | <ul> <li>alanine aminotransferase (ALT)*</li> <li>albumin*</li> <li>alkaline phosphatase</li> <li>aspartate aminotransferase (AST)*</li> <li>bicarbonate</li> <li>bilirubin (direct and total)*</li> <li>blood urea nitrogen (BUN)</li> <li>calcium</li> <li>chloride</li> <li>creatinine</li> <li>glucose</li> <li>lactate dehydrogenase (LDH)</li> <li>phosphorus</li> <li>potassium</li> <li>sodium</li> <li>total protein</li> <li>uric acid</li> </ul> |
| COAGULATION PARAMETERS | OTHER |
| <ul> <li>International Normalized Ratio (INR)*</li> <li>partial thromboplastin time (PTT)</li> <li>prothrombin time (PT)*</li> </ul> | <ul> <li>alpha-fetoprotein (AFP): at baseline and Day 1 of each subsequent cycle*</li> <li>thyroid functions (T3, T4, TSH) at Pre-Study, Baseline, Day 1 of subsequent cycles, EOS, and Follow-up</li> <li>serum pregnancy test: females of childbearing potential</li> <li>hepatitis B and C viral load measurement every odd numbered cycle (where applicable)*</li> </ul> |
| *Exploratory efficacy variables | |

## 10.4 APPENDIX D – ECOG PERFORMANCE STATUS

| Level | ECOG Performance Status |
|-------|-------------------------|
| 0 | Normal activity |
| 1 | Symptoms but ambulatory |
| 2 | In bed < 50% of time |
| 3 | In bed > 50 % of time |
| 4 | 100 % bedridden |

# 10.5 APPENDIX E – CARDIAC FUNCTION CLASSIFICATION

| | Cardiac Functional Classification |
|---|---|
| NYHA<br>Class | Symptoms |
| I | Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. |
| II | Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. |
| III | Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20–100 m). Comfortable only at rest. |
| IV | Severe limitations. Experiences symptoms even while <i>at rest</i> . Mostly bedbound patients. |



A Phase 2, Randomized, Double-Blind, Placebo- Controlled Study of the Efficacy and Safety of CF102 in the Second-Line Treatment of Advanced Hepatocellular Carcinoma in Subjects with Child-Pugh Class B Cirrhosis

Mock Tables and Listings Version 7.0 29 August 2019

**CONFIDENTIAL** 

## **Table of Contents**

| 1. | INTRODUCTION | 5 |
|----|-----------------------|------|
| 2. | REPORTING CONVENTIONS | 5 |
| 3. | OUTPUT TITLES | 6 |
| 3 | 3.1. Table Titles | 6 |
| | 3.2. Listing Titles | |
| 4. | EXAMPLES | 12 |
| | 1.1. Table Examples | |
| | Table 14.1.1 | |
| | Table 14.1.2 | |
| | Table 14.1.3 | |
| | Table 14.1.4.1 | |
| | Table 14.1.4.2 | |
| | Table 14.1.4.3 | |
| | Table 14.1.5 | |
| | Table 14.1.6 | |
| | Table 14.1.7 | |
| | Table 14.2.1 | |
| | Figure 14.2.1 | |
| | Figure 14.2.2 | |
| | Figure 14.2.3 | . 24 |
| | Table 14.2.2.1.1 | . 25 |
| | Table 14.2.2.2.1 | . 26 |
| | Table 14.2.3.1 | . 27 |
| | Table 14.2.3.2 | . 28 |
| | Table 14.2.3.3 | 29 |
| | Table 14.2.4.1 | |
| | Table 14.2.4.2 | |
| | Table 14.2.4.3 | |
| | Table 14.2.4.4 | |
| | Table 14.2.5.1 | |
| | Table 14.2.6 | |
| | Table 14.2.7.1 | |
| | Figure 14.2.7.1 | |
| | Table 14.2.7.2 | |
| | Table 14.2.7.3 | |
| | Table 14.2.7.4 | |
| | Table 14.2.7.5 | |
| | Table 14.2.7.6 | |
| | Table 14.2.7.7 | |
| | Table 14.2.7.8 | |
| | Table 14.2.7.9 | . 45 |

| | Table 14.2.7.10 | 46 |
|----|---------------------|------|
| | Table 14.3.1 | 47 |
| | Table 14.3.2 | . 48 |
| | Table 14.3.3 | 49 |
| | Table 14.3.4.1 | . 50 |
| | Table 14.3.4.2 | . 51 |
| | Table 14.3.5 | . 52 |
| | Table 14.3.6.1 | . 53 |
| | Table 14.3.6.4 | . 54 |
| | Table 14.3.7.1 | . 55 |
| | Table 14.3.7.2 | . 56 |
| | Table 14.3.8 | . 57 |
| | Table 14.3.9.1 | . 58 |
| | Table 14.3.9.2 | . 59 |
| | Table 14.3.10.1 | . 60 |
| | Table 14.3.10.2 | 61 |
| | Table 14.3.11 | 62 |
| 4. | 2. Listing Examples | 63 |
| | Listing 16.2.1.1 | 63 |
| | Listing 16.2.1.2 | 64 |
| | Listing 16.2.2.1 | 65 |
| | Listing 16.2.2.2 | 67 |
| | Listing 16.2.3.1 | 69 |
| | Listing 16.2.3.2 | . 70 |
| | Listing 16.2.3.3.1 | . 71 |
| | Listing 16.2.3.3.2 | . 72 |
| | Listing 16.2.3.4 | . 73 |
| | Listing 16.2.3.5 | . 74 |
| | Listing 16.2.3.6 | . 75 |
| | Listing 16.2.4.1 | 76 |
| | Listing 16.2.4.2 | . 77 |
| | Listing 16.2.5.1 | . 78 |
| | Listing 16.2.5.2 | |
| | Listing 16.2.6.1.1 | |
| | Listing 16.2.6.1.2 | |
| | Listing 16.2.6.2 | |
| | Listing 16.2.6.3.1 | |
| | Listing 16.2.6.3.2 | |
| | Listing 16.2.6.4 | |
| | Listing 16.2.6.5.1 | |
| | Listing 16.2.6.5.2 | |
| | Listing 16.2.7 | |
| | Listing 16.2.8.1 | |
| | Listing 16.2.8.2 | |
| | Listing 16.2.8.3 | 95 |

| Listing 16.2.8.4 | 97 |
|-------------------|-----|
| Listing 16.2.8.5 | |
| Listing 16.2.8.6 | |
| Listing 16.2.9.1 | |
| Listing 16.2.9.2 | |
| Listing 16.2.9.3 | |
| Listing 16.2.10.1 | |
| Listing 16.2.10.2 | 105 |
| Listing 16.2.11.1 | 106 |
| Listing 16.2.11.2 | 107 |
| Listing 16.2.12 | 108 |
| Listing 16.2.13 | |

#### 1. INTRODUCTION

This document is to be used in conjunction with the current Statistical Analysis Plan (SAP), protocol (Amendment 5, dated 6 November 2018), and corresponding CRFs.

The following pertains to the double-blind period only. Shells for the open-label period will be presented with a separate SAP.

Hyper-links are identified in this document as blue underlined text.

#### 2. REPORTING CONVENTIONS

All output will be generated by SAS and exported into a Microsoft Word document in RTF format. All output will be in landscape orientation. Left and right margins will be 1 inch from the side; the top and bottom margins will be 1.12 inches. Font size will be Arial 8 pt.

The header containing the sponsor name (Can-Fite BioPharma, Ltd.) and protocol number (CF102-201HCC) will appear on the top left corner of each page of the output. The page number, in the format of "Page x of y", will appear on the top right corner of the output, where y = last page of corresponding output. Horizontal lines will appear after the title, after the column headers and after the main body of the output.

The header and the titles section will be separated by one line. After the header, there will be a blank line. The titles will be presented as:

Line1: Table or Figure [number]

Line2a: [title]

Line2b: [subtitle, if applicable]

Line3: [xxx] Population

Footnotes will be placed after the main body of the table, under the horizontal line. Footnotes that need to reference a specific phrase will use a numeric convention (Example: 1, 2, 3). The last footnote will identify the listing or statistical appendix cross-reference as follows: Source: Listing 16.2.x. The sources for each table are identified in Section 3.1, Table Titles.

#### Table Format Specification

Maximum and minimum values will be reported with the same number of decimal places as collected. Means and medians will be reported to one additional decimal place. Standard deviations and standard errors will be reported to two decimal places more than the collected data. Percents will be reported with one decimal place. P-values will be rounded to three decimal places (e.g., "0.xxx"). If a p-value <0.001, then the p-value will be reported as "<0.001".

If the frequency is 0 or 1 for a category for calculation of a standard deviation or standard error, then enter '(NE)' for calculation of the standard deviation or standard error and add a footnote (penultimate preceding Source) of 'NE= Not Estimable'.

If the frequency for "Total" <2 for a categorical variable for either treatment group, or frequency is "Total" for any category, i.e. a percent of 100 for that category, for both treatment groups, then enter 'NA' for the p-value with a footnote (penultimate preceding "Source") of 'NA = Not Applicable'.

Data in the tables are formatted as follows:

- Text fields in the body of the tables and listings will be left-justified.
- All numeric values between -1 and 1 are outputted with zero to the left of the decimal point (e.g. 0.12, 0.3).
- Unless otherwise specified, percentage values are output with one digit to the right of the decimal point (e.g., 12.3, 4.5). Percentages that are > 0.0 and < 0.1 (not 0.0) are reported as "< 0.1".</li>
- When no data are available for a table, an empty page with the title will be produced with suitable text. Example: THERE WERE NO SERIOUS ADVERSE EVENTS.

For many variables assessed at Pre-Study Visit, Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1) or if value at Cycle 1 Day 1 is missing. These are variables are identified with a footnote indicating this.

Dates will be presented as recorded. All listings will include the Safety Population and will be sorted by site, subject, and cycle (if appropriate). Treatments are to be formatted as CF102 and Placebo in listings.

#### 3. OUTPUT TITLES

#### 3.1. Table Titles

Table examples related to the following titles are located in the next section. Please footnote all information in the 'Listing Source' column for the corresponding table.

| Number | Title of Table | Analysis<br>Population | Listing Source |
|---|---|---|---|
| Number | DISPOSITION, DEMOGRAPHIC AND TREATMENT DATA | i opulation | Listing Source |
| 14.1.1 | Analysis Populations | Safety | <u>16.2.1.1, 16.2.1.2</u> |
| 14.1.2 | Study Completion and Primary Reason for Withdrawal | Safety | 16.2.1.1 |
| 14.1.3 | Demographic and Baseline Characteristics | Safety | 16.2.3.1 |
| 14.1.4.1 | HCC History and Diagnosis | Safety | <u>16.2.3.2</u> , <u>16.2.3.3.1</u> , |
| | | <b>-</b> | 16.2.3.5 |
| 14.1.4.2 | Number of Target Lesions at Screening | Safety | <del>16.2.6.1</del> .1 |
| 14.1.4.3 | Extrahepatic Spread (EHS) and Portal Vein Thrombosis (PVT) | Safety | 16.2.3.3.2 |
| 14.1.5 | Medical History (Excluding Past HCC, Cirrhosis, and Viral Hepatitis-Related | Safety | 16.2.3.6 |
| | History) | | |
| <u>14.1.6</u> | HCC Prior Therapies | Safety | <u>16.2.3.4</u> |
| <u>14.1.7</u> | Treatment Compliance and Duration of Treatment | Safety | <u>16.2.4.1</u> |
| | <b>EFFICACY</b> | | |
| <u>14.2.1</u> | Time to Event (months) | ITT | <u>16.2.5.1</u> |
| | Figure 14.2.1: Kaplan-Meier curve for OS | ITT | <u>16.2.5.1</u> |
| | Figure 14.2.2: Kaplan-Meier curve for TTP | ITT | 16.2.5.1 |
| | Figure 14.2.3: Kaplan-Meier curve for PFS | ITT | 16.2.5.1 |
| 14.2.2.1.1 | Overall Response Using RECIST Criteria | ITT | <u>16.2.6.3.1</u> |
| 14.2.2.1.2 | Overall Response Using RECIST Criteria | PP<br> | <u>16.2.6.3.1</u> , <u>16.2.1.2</u> |
| 14.2.2.2.1 | Best Overall Response | ITT | <u>16.2.6.3.1</u> |
| 14.2.2.2.2 | Best Overall Response | PP | <u>16.2.6.3.1</u> , <u>16.2.1.2</u> |
| 14.2.3.1 | WBC A3AR expression | ITT | 16.2.6.4 |
| 14.2.3.1 | WBC A3AR expression by Overall Response | ITT | |
| 14.2.3.3 | Overall Response by CFB for WBC A3AR expression | ITT | <u>16.2.6.3.1</u> , <u>16.2.6.4</u><br><u>16.2.6.3.1</u> , <u>16.2.6.4</u> |
| 14.2.4.1 | Alpha-fetoprotein (AFP) | ITT | 16.2.6.4 |
| | Alpha-fetoprotein (AFP) Alpha-fetoprotein (AFP) by Overall Response | ITT | <del></del> |
| 14.2.4.2<br>14.2.4.3 | Overall Response by Categorical Alpha-fetoproterin (AFP) | ITT | <u>16.2.6.3.1</u> , <u>16.2.6.4</u><br>16.2.6.3.1, 16.2.6.4 |
| 14.2.4.4 | Overall Response by CFB for Alpha-fetoproterin (AFP) | ITT | 16.2.6.3.1, 16.2.6.4<br>16.2.6.3.1, 16.2.6.4 |
| 14.2.4.4 | Overall Nesponse by OFD for Alpha-letoproteill (AFF) | 111 | 10.2.0.3.1, 10.2.0.4 |

| Number | Title of Table | Analysis<br>Population | Listing Source |
|---|---|---|---|
| EXPLORATORY EFFICACY | | | |
| 14.2.5.1 | Alanine aminotransferase (ALT) | ITT | 16.2.8.2 |
| 14.2.5.2 | Aspartate aminotransferase (AST) | ITT | 16.2.8.2 |
| 14.2.5.3 | Albumin | ITT | 16.2.8.2 |
| 14.2.5.4 | Bilirubin (direct) | ITT | 16.2.8.2 |
| 14.2.5.5 | Bilirubin (total) | ITT | 16.2.8.2 |
| 14.2.5.6 | International Normalized Ratio (INR) | ITT | 16.2.8.3 |
| 14.2.5.7 | Prothrombin time (PT) | ITT | 16.2.8.3 |
| 14.2.6 | Hepatitis Viral Load | ITT | 16.2.3.3.1, |
| | | | <u>16.2.6.5.1</u> , <u>16.2.6.5.2</u> |
| | SUBGOUP ANALYSES - EFFICACY | | |
| 14.2.7.1 | Overall Survival (OS; months) by Child-Pugh (CP) Score at Screening | ITT | <u>16.2.3.1, 16.2.5.1</u> |
| | Figure 14.2.7.1: Kaplan-Meier curve for OS, CP Score at Screening = 7 | itt | 16.2.3.1, <u>16.2.5.1</u> |
| | Figure 14.2.7.2: Kaplan-Meier curve for OS, CP Score at Screening = 8 | ITT | 16.2.3.1, 16.2.5.1 |
| | Figure 14.2.7.3: Kaplan-Meier curve for OS, CP Score at Screening = 7 or 8 | ITT | 16.2.3.1, 16.2.5.1 |
| 14.2.7.2 | Overall Survival (OS; months) by Sex | ITT | 16.2.3.1, 16.2.5.1 |
| 14.2.7.3 | Overall Survival (OS; months) by ECOG PS at Screening | ITT | 16.2.9.3, 16.2.5.1 |
| 14.2.7.4 | Overall Survival (OS; months) by Alpha-fetoprotein (AFP) at Baseline | ITT | 16.2.6.4, 16.2.5.1 |
| 14.2.7.5 | Overall Survival (OS; months) by Prior Locoregional Therapy | ITT | 16.2.3.4, 16.2.5.1 |
| 14.2.7.6 | Overall Survival (OS; months) by Either EHS or PVT | ITT | <u>16.2.3.3.2, 16.2.5.1</u> |
| 14.2.7.7 | Overall Survival (OS; months) by History of HBV | ITT | <u>16.2.3.3.1</u> , <u>16.2.5.1</u> |
| 14.2.7.8 | Overall Survival (OS; months) by History of HCV | ITT | 16.2.3.3.1, 16.2.5.1 |
| 14.2.7.9 | Overall Survival (OS; months) by Diagnostic Procedure | ITT | 16.2.3.2, 16.2.5.1 |
| 14.2.7.10 | Overall Survival (OS; months) by Country | ITT | 16.2.1.1, 16.2.5.1 |
| | THE PREVIOUS SHOULD BE IN THE SAME ORDER AS IN TEXT | | |
| | SAFETY | | |
| | Adverse Events | | |
| 14.3.1 | Incidence of Treatment-Emergent Adverse Events | Safety | 16.2.7 |
| 14.3.2 | Incidence of Treatment-Emergent Adverse Events by Relationship | Safety | 16.2.7 |
| 14.3.3 | Incidence of Treatment-Emergent Adverse Events by Severity | Safety | 16.2.7 |
| 14.3.4.1 | Listing of Deaths | Safety | <u>16.2.1.1</u> , <u>16.2.5.1</u> , |
| <u> </u> | | | 16.2.7 |
| 14.3.4.2 | Listing of Serious Adverse Events | Safety | 16.2.7 |
| 14.3.5 | Listing of Discontinuations due to Adverse Events | Safety | 16.2.7 |

| Title of Table | Population | Listing Source |
|---|---|---|
| Laboratory Values | | |
| • | C-f-t- | 40.0.0.4 |
| | • | 16.2.8.1 |
| | Safety | <u>16.2.8.2</u> |
| Clinical Laboratory Evaluations: Coagulation | Safety | <u>16.2.8.3</u> |
| Clinical Laboratory Evaluations: Thyroid Function | Safety | <u>16.2.8.5</u> |
| Other Safety | | |
| ECOG Performance Status (PS) | Safety | 16.2.9.3 |
| | • | 16.2.9.3 |
| | • | 16.2.9.1, 16.2.9.2 |
| | , | 16.2.10.1 |
| | • | 16.2.10.2 |
| | • | 16.2.11.1 |
| | , | 16.2.11.2 |
| · | • | 16.2.12 |
| | Laboratory Values Clinical Laboratory Evaluations: Hematology Clinical Laboratory Evaluations: Blood Chemistry Clinical Laboratory Evaluations: Coagulation | Laboratory ValuesClinical Laboratory Evaluations: HematologySafetyClinical Laboratory Evaluations: Blood ChemistrySafetyClinical Laboratory Evaluations: CoagulationSafetyClinical Laboratory Evaluations: Thyroid FunctionSafetyOther SafetyECOG Performance Status (PS)SafetyChange from Baseline in ECOG Performance StatusSafetyVital Signs And WeightSafetyElectrocardiogram (ECG) ParametersSafetyCategorical Electrocardiogram (ECG) ParametersSafetyPhysical Examination at Pre-Study VisitSafetyPhysical ExaminationSafety |

## 3.2. Listing Titles

| Number | Title of Listing |
|---|---|
| 16.2.1.1 | Completed and Discontinued Subjects with Primary Reason for Withdrawal |
| <u>16.2.1.2</u> | Subjects Excluded from Analysis Populations |
| <u>16.2.2.1</u> | Inclusion Criteria |
| <u>16.2.2.2</u> | Exclusion Criteria |
| <u>16.2.3.1</u> | Demographic and Baseline Characteristics |
| <u>16.2.3.2</u> | HCC Diagnosis |
| <u>16.2.3.3</u> .1 | HCC History |
| <u>16.2.3.3.2</u> | Extrahepatic Spread (EHS) and Portal Vein Thrombosis (PVT) |
| <u>16.2.3.4</u> | HCC Prior Therapies |
| <u>16.2.3.5</u> | Cirrhosis / Virus Complications and Treatment |
| <u>16.2.3.6</u> | Medical History (Excluding Past HCC and Cirrhosis-Related History) |
| <u>16.2.4.1</u> | Study Drug Accountability and Treatment Compliance |
| <u>16.2.4.2</u> | Study Drug Accountability by Visit |
| <u>16.2.5.1</u> | Time to Event |
| <u>16.2.5.2</u> | Survival Follow-up Contact Dates |
| <u>16.2.6.1.1</u> | Tumor Evaluations: Target Lesions |
| <u>16.2.6.1.2</u> | Summary of Target Lesions |
| <u>16.2.6.2</u> | Tumor Evaluations: Non-Target Lesions |
| <u>16.2.6.3.1</u> | Tumor Response |
| <u>16.2.6.3.2</u> | Tumor Response (Investigator Assessments) |
| <u>16.2.6.4</u> | Biomarkers (AFP and WBC A3AR) |
| <u>16.2.6.5.1</u> | Hepatitis B Viral Load |
| <u>16.2.6.5.2</u> | Hepatitis C Viral Load |

| Number | Title of Listing |
|------------------|---------------------------------------------------|
| 16.2.7 | Adverse Events |
| <u>16.2.8.1</u> | Clinical Laboratory Evaluations: Hematology |
| <u>16.2.8.2</u> | Clinical Laboratory Evaluations: Blood Chemistry |
| <u>16.2.8.3</u> | Clinical Laboratory Evaluations: Coagulation |
| <u>16.2.8.4</u> | Clinical Laboratory Evaluations: Urinalysis |
| <u>16.2.8.5</u> | Clinical Laboratory Evaluations: Thyroid Function |
| <u>16.2.8.6</u> | Pregnancy Test |
| <u>16.2.9.1</u> | Vital Signs |
| <u>16.2.9.2</u> | Weight, Height, and BMI |
| <u>16.2.9.3</u> | ECOG Performance Status |
| <u>16.2.10.1</u> | Electrocardiogram (ECG) – Continuous Variables |
| <u>16.2.10.2</u> | Electrocardiogram (ECG) – Categorical Variables |
| <u>16.2.11.1</u> | Physical Examination at Pre-Study Visit |
| <u>16.2.11.2</u> | Physical Examination |
| <u>16.2.12</u> | Prior and Concomitant Medications |
| <u>16.2.13</u> | Investigator Comments |

### 4. EXAMPLES

#### Table Examples 4.1.

Table 14.1.1 **Analysis Populations** 

| | CF102 | Placebo | Total |
|-----------------------------------|-----------|-----------|-----------|
| | (N=xx) | (N=xx) | (N=xx) |
| Safety Population | xx | xx | xx |
| Bulgaria | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serbia | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Israel | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Romania | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| United States | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Exclusions from ITT Population | | | |
| No Post-Baseline Tumor Assessment | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ITT Population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bulgaria | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serbia | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Israel | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Romania | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| United States | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Exclusions from PP Population | | | |
| Reason 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PP Population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bulgaria | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serbia | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Israel | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Romania | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| United States | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Percentages are calculated using the number of subjects in the Safety Population for each treatment (or Total) as the denominator. ITT= Intent-to-Treat

PP=Per Protocol

Country is based on the first digit of the site number (1=Bulgaria, 2=Serbia, 3=Israel, 5=Romania, or 7=United States).

Source: Listings <u>16.2.1.1</u>, <u>16.2.1.2</u>

Programming Notes: Any reasons for exclusion from ITT Population (other than "No Post-Baseline Tumor Assessment") and reasons for exclusion from PP Population, and identification of subjects excluded, will be finalized prior to unblinding.

**Table 14.1.2**Study Completion and Primary Reason for Withdrawal Safety Population

| Status, n(%) | CF102<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|
| Primary Reason for Withdrawal from Dosing | | | |
| Grade 3 toxicity considered by the Investigator to be at least "possibly" drug-related that does not resolve to | | | |
| Grade ≤ 1 within 7 days following interruption of treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 toxicity considered by the Investigator to be at least "possibly" drug-related | xx (xx.x) | xx (xx.x) | XX (XX.X)<br>XX (XX.X) |
| Need for > 1 dose reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment interruption or delay for more than 14 days after the next scheduled dose due to an event unrelated | ** (**.*) | ** (**.*) | ** (**.*) |
| to toxicity | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdrawal of consent for trial participation at any time, for any reason, and without prejudice | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal of a subject by the Investigator, at his/her discretion, for any reason that the Investigator believes | ^^ (^^.^) | ^^ (^^.^) | ^^ (^^.^) |
| continuation of study drug therapy would not be in the subject's best interest. | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| An intercurrent illness which, in the Investigator's opinion, would prevent completion of trial-related evaluations | xx (xx.x) | xx (xx.x) | XX (XX.X)<br>XX (XX.X) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject noncompliance with trial or follow-up procedures | xx (xx.x) | xx (xx.x) | XX (XX.X)<br>XX (XX.X) |
| Termination of the trial by the Sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | ** (**.*) | ** (**.*) | ** (**.*) |
| Primary Reason for Withdrawal from Trial | | | |
| Withdrawal of consent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Termination of the trial by the Sponsor | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Death | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Total | xx (xx.x) | xx (xx.x) | XX (XX.X) |

Percentages are calculated using the number of subjects in the Safety Population for each treatment (or Total) as the denominator. Source: Listing 16.2.1.1

Programming Note: Subjects should have response to either Primary Reason for Withdrawal from Dosing or Primary Reason for Withdrawal from Trial, but not BOTH.

Table 14.1.3

Demographic and Baseline Characteristics
Safety Population

| Parameter (1) Statistic CF102 Placebo Total |
|---------------------------------------------|
|---------------------------------------------|

| | | (N=xx) | (N=xx) | (N=xx) |
|---|---|---|---|---|
| Age (years) | n | xx | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Sex, n (%) | Male | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , , | Female | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx | xx |
| Origin, n (%) | White/Caucasian | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Black/African | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Oriental | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | XX | xx | XX |
| Child-Pugh Score, n (%) | 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 , (, | 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 9 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx | xx |

(1) Age is age at Screening.

Percentages are calculated using the number of subjects in the Safety Population for each treatment (or Total) as the denominator. Source: Listing 16.2.3.1

Table 14.1.4.1 **HCC History and Diagnosis** Safety Population

| | | CF102 | Placebo | Total |
|---|---|---|---|---|
| Parameter | | (N=xx) | (N=xx) | (N=xx) |
| History of Viral Hepatitis, n (%) (1) | Yes – Hepatitis B | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | Yes – Hepatitis C | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Not Known | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hepatitis B Serology, n (%) | Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | XX | XX | XX |
| Hepatitis C Serology, n (%) | Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | XX | XX | XX |
| Complications, n (%) (1) | None | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Ascites | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Esophageal varices with bleeding | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Diagnostic Procedure, n (%) (2) | Cytology/histology | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| - , , , , | AASLD | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | XX | XX | XX |

Percentages are calculated using the number of subjects in the Safety Population for each treatment (or Total) as the denominator. (1) Percentages may sum to more than 100% because more than one response is possible.

Programming Note: Check that no subject has "None" for Complications with another response.

<sup>(2)</sup> AASLD=American Association for the Study of Liver Diseases Source: Listings 16.2.3.2, 16.2.3.3.1, 16.2.3.5

Table 14.1.4.2

Number of Target Lesions at Screening
Safety Population

| | Non- Liver | Number of | | | | Number of L | iver Lesions | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Site Code (1) | Non- Liver Lesions | 0 | 1 | 2 | 3 | 4 | 5 | 7 | Tota |
| CF102 (N=xx) | None | | | | XX | XX | XX | XX | | XX |
| , , | 01 | 1 | | | XX | XX | XX | XX | | XX |
| | | 2 | XX | XX | XX | XX | | XX | | XX |
| | 02 | 1 | | XX | XX | XX | | XX | | XX |
| | | 2 | | XX | XX | XX | XX | XX | | XX |
| | 10 | 1 | | | XX | XX | XX | XX | | XX |
| | 99 | 1 | | XX | XX | XX | XX | XX | | XX |
| | | 2<br>3 | XX | XX | XX | XX | XX | XX | | XX |
| | | 3 | | XX | XX | XX | XX | XX | | XX |
| | Total (2) | | XX | XX | XX | XX | XX | XX | | XX |
| Placebo (N=xx) | None | | | XX | | | XX | XX | | XX |
| | 02 | 0 | | XX | XX | XX | XX | XX | XX | XX |
| | | 1 | | XX | XX | XX | XX | XX | | XX |
| | 04 | 1 | | XX | | | XX | XX | | XX |
| | | 2 | | XX | XX | XX | XX | XX | | XX |
| | 99 | 1 | | XX | XX | | | XX | | XX |
| | | 2<br>3 | | XX | XX | XX | XX | XX | | XX |
| | | 3 | XX | XX | XX | XX | | | | XX |
| | Total (2) | | XX | XX | XX | XX | XX | XX | | XX |
| Γotal (N=xx) | None | | | XX | XX | XX | XX | XX | | XX |
| | 01 | 1 | | | XX | XX | XX | XX | | XX |
| | | 2 | XX | XX | XX | XX | | XX | | XX |
| | 02 | 0 | | XX | XX | XX | XX | XX | XX | XX |
| | | 1 | XX | XX | XX | XX | XX | XX | | XX |
| | | 2 | XX | XX | XX | XX | XX | XX | | XX |
| | 04 | 1 | | XX | | | XX | XX | | XX |
| | | 2 | | XX | XX | XX | XX | XX | | XX |
| | 10 | 1 | | | XX | XX | XX | XX | | XX |
| | 99 | 1 | | XX | XX | XX | XX | XX | | XX |
| | | 2<br>3 | XX | XX | XX | XX | XX | XX | | XX |
| | | 3 | XX | XX | XX | XX | XX | XX | | XX |
| | Total (2) | | XX | XX | XX | XX | XX | XX | | XX |

<sup>(1)</sup> Site Codes: 01 = Abdominal Wall, 02 = Adrenal, 03 = Bladder, 04 = Bone, 05 = Breast, 06 = CNS, 07 = Colon, 08 = Liver, 09 = Lung, 10 = Lymph Nodes,

Source: Listing <u>16.2.6.1.1</u>

Programming Notes: Do not skip numbers for liver lesions for 1 through 5. There should be no subjects with 0 liver lesions or more than 5 liver lesions; if these are observed, include them as above, but otherwise only 1 through 5. Include only non-zero counts. For non-liver lesions, exclude rows with no entries. If any subjects have only liver lesions, include "None" row as non-liver site code. The values will be the counts of lesions at "Screening" from Listing 16.2.6.1.1.

<sup>11 =</sup> Pancreas, 12 = Pelvis, 13 = Pleura, 14 = Rectum, 15 = Retroperitoneal Cavity, 16 = Retroperitoneum, 17 = Small Intestine, 18 = Uterus, 99 = Other

<sup>(2)</sup> Number of non-liver lesions may not sum to Total due to subjects with more than one non-liver site.

Table 14.1.4.3

Extrahepatic Spread (EHS) and Portal Vein Thrombosis (PVT)
Safety Population

| | | CF102 | Placebo | Total |
|------------------------------|-------|-----------|-----------|-----------|
| Parameter, n (%) | | (N=xx) | (N=xx) | (N=xx) |
| Extrahepatic Spread (EHS) | Yes | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | XX | xx | xx |
| Portal Vein Thrombosis (PVT) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ` , | No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx | хх |
| Either EHS or PVT | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx | хх |
| Both EHS and PVT | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx | хх |

Percentages are calculated using the number of subjects for each treatment (or Total) as the denominator.

Source: Listing <u>16.2.3.3.2</u>

Programming Note: "Either EHS or PVT"= "Yes" if EHS= "Yes" or PVT= "Yes" and otherwise "Either EHS or PVT"= "No". "Both EHS and PVT"= "Yes" if EHS= "Yes" and PVT"= "Yes" and otherwise "Both EHS and PVT"= "No".

Table 14.1.5

Medical History (Excluding Past HCC, Cirrhosis, and Viral Hepatitis-Related History)
Safety Population

| | CF102 | Placebo | Total |
|---------------------------------|-----------|-----------|-----------|
| Body System, n (%) | (N=xx) | (N=xx) | (N=xx) |
| None | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Allergy/Immunological | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cardiovascular | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dermatological | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ENT | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gastrointestinal/ Hepatobiliary | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hematological/ Lymphatic | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Metabolic/Endocrine | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Musculoskeletal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neoplastic | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neurological/ Psychiatric | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pulmonary | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Renal/Urological | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reproductive | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Counts represent the number of subjects with a finding or procedure recorded for each body system or None.

Percentages are calculated using the number of subjects in the Safety Population for each treatment (or Total) as the denominator. Source: Listing 16.2.3.6

Programming Notes: Present body systems alphabetically after "None". Check that no subject has "None" for Body System with another response.

Table 14.1.6
HCC Prior Therapies
Safety Population

| | CF102 | Placebo | Total |
|----------------------|-----------|-----------|-----------|
| Prior Therapy, n (%) | (N=xx) | (N=xx) | (N=xx) |
| 01 = Surgery | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | XX | XX | XX |
| 02 = Radiation | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | XX | XX | XX |

The entries are the number (and percentage) of subjects reporting the use of a modality at least once. Percentages are calculated using the number of subjects in the Safety Population for each treatment (or Total) as the denominator.

Source: Listing 16.2.3.4

Programming Note: Continue for Modality Codes: 03 = Chemotherapy, 04 = Immunotherapy, 05 = Hormonal therapy, 06 = Targeted Therapy (sorafenib), 07 = Chemoembolization, 08 = Anti-viral therapy, 09 = Other.

Table 14.1.7

Treatment Compliance and Duration of Treatment
Safety Population

| | CF102 | Placebo | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Compliance Rate, % (1) | • | | • |
| n | XX | XX | XX |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx | xx.xx |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Duration of Treatment (days) | | | |
| n , , , , , , | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | XX, XX | XX, XX |

Source: Listing <u>16.2.4.1</u>

<sup>(1)</sup> A subject's compliance rate during the study is 100% \* (total number of capsules dispensed minus the total number of capsules returned) divided by twice the subject's duration of treatment.

Table 14.2.1 Time to Event (months) ITT Population

| Dorometer | Ctatiotic | CF102 | Placebo |
|---|---|---|---|
| Parameter | Statistic | (N=xx) | (N=xx) |
| Overall Survival (OS) | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Value of KM at Median Duration (%) | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | XX (XX.X) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | Covariate= Baseline AFP | | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| | Covariate= Baseline WBC A3AR | | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| Time To Progression (TTP) | n | XX | XX |
| ······o ··o · ··og··oocio··· (· ··· / | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Value of KM at Median Duration (%) | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | XX (XX.X) |
| | Number (%) censored | XX (XX.X) | XX (XX.X) |
| | P-value (LR) | 0.xxx | λλ (λλ.λ) |
| Progression-free Survival (PFS) | n | XX | xx |
| 1 Togression-nee ourvival (1 1 0) | 25th Percentile | XX.X | XX.X |
| | Median | XX.X<br>XX.X | XX.X<br>XX.X |
| | 75th Percentile | XX.X<br>XX.X | XX.X<br>XX.X |
| | Value of KM at Median Duration (%) | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| D value (LD) -D value using the log | P-value (LR) | 0.xxx | |

P-value (LR) =P-value using the logrank test. KM=Kaplan-Meier

Baseline=Cýcle 1 Day 1

Percentages are calculated using the number of subjects in the ITT Population for each treatment as the denominator. For Median Duration, see <u>Table 14.1.7</u>.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment and the specified covariate in the model

and P-value (PH) is the corresponding p-value (Chi-Square).

Source: Listing <u>16.2.5.1</u>

Figure 14.2.1

Kaplan-Meier curve for OS

ITT Population



Source: Listing <u>16.2.5.1</u>

Figure 14.2.2

Kaplan-Meier curve for TTP ITT Population



Source: Listing <u>16.2.5.1</u>

Programming Note: Include number of patients at any month in the figure.

Figure 14.2.3

Kaplan-Meier curve for PFS
ITT Population



Source: Listing <u>16.2.5.1</u>

Programming Note: Include number of patients at any month in the figure.

Table 14.2.2.1.1

Overall Response Using RECIST Criteria
ITT Population

| | | CF102 | Placebo |
|---------------|-----------------|-----------|-----------|
| Visit | Response, n (%) | (N=xx) | (N=xx) |
| Cycle 3 Day 1 | CR | xx (xx.x) | xx (xx.x) |
| | PR | xx (xx.x) | xx (xx.x) |
| | SD | xx (xx.x) | xx (xx.x) |
| | PD | xx (xx.x) | xx (xx.x) |
| | Total | XX | xx |
| | ORR | xx (xx.x) | xx (xx.x) |
| | P-value | 0.xxxx | ` , |
| | DCR | xx (xx.x) | xx (xx.x) |
| | P-value | 0.xxxx | , , |
| Cycle 5 Day 1 | CR | xx (xx.x) | xx (xx.x) |
| | PR | xx (xx.x) | xx (xx.x) |
| | SD | xx (xx.x) | xx (xx.x) |
| | PD | xx (xx.x) | xx (xx.x) |
| | Total | XX | XX |
| | ORR | xx (xx.x) | xx (xx.x) |
| | P-value | 0.xxxx | |
| | DCR | xx (xx.x) | xx (xx.x) |
| | P-value | 0.xxxx | |

Includes only assessments through Cycle 11.

CR=Complete Response, PR =Partial Response, SD =Stable Disease, PD=Progressive Disease

ORR=Objective Response Rate= proportion of subjects who have response of CR or PR

DCR=Disease Control Rate= proportion of subjects who have response of CR, PR, or SD

Percentages are calculated using the number of subjects in the ITT Population for each treatment as the denominator.

P-values determined using the normal approximation to the binomial distribution using observed responses.

ITT= Intent-to-Treat

NA = Not Applicable

Source: <u>Listing 16.2.6.3.1</u>

Programming Notes: Continue for all cycles through Cycle 11.

Use same structure for Table 14.2.2.1.2 (PP Population) with PP instead of ITT in the two appropriate footnotes and the last footnote changed to "Source: Listings 16.2.6.3.1, 16.2.1.2".

Table 14.2.2.2.1

Best Overall Response
ITT Population

| | CF102 | Placebo |
|------------------------------|-----------|-----------|
| Best Overall Response, n (%) | (N=xx) | (N=xx) |
| CR | xx (xx.x) | xx (xx.x) |
| PR | xx (xx.x) | xx (xx.x) |
| SD | xx (xx.x) | xx (xx.x) |
| PD | xx (xx.x) | xx (xx.x) |
| Total | xx | xx |
| ORR | xx (xx.x) | xx (xx.x) |
| P-value | 0.xxxx | |
| DCR | xx (xx.x) | xx (xx.x) |
| P-value | 0.xxxx | |

CR=Complete Response, PR =Partial Response, SD =Stable Disease, PD=Progressive Disease

ORR=Objective Response Rate= proportion of subjects who have response of CR or PR

DCR=Disease Control Rate= proportion of subjects who have response of CR. PR, or SD

Percentages are calculated using the number of subjects in the ITT Population for each treatment as the denominator.

P-values determined using the normal approximation to the binomial distribution using observed responses.

Best Overall Response is determined for the entire duration of the study and is counted once per subject, although it may occur more than once.

ITT= Intent-to-Treat

NA = Not Applicable Source: Listing 16.2.6.3.1

Programming Notes: Best Overall Response is determined for the entire duration of the study. Use same structure for Table 14.2.2.2.2 (PP Population) with PP instead of ITT in the two appropriate footnotes and the last footnote changed to "Source: Listings 16.2.6.3.1, 16.2.1.2".

Table 14.2.3.1 WBC A3AR expression ITT Population

| | | CF102 | Placebo |
|----------------------|-----------|----------------|----------------|
| Visit | Statistic | (N=xx) | (N=xx) |
| Baseline | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| Cycle 3 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| CFB at Cycle 3 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| Cycle 5 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| CFB at Cycle 5 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |

CFB=Change from Baseline
Baseline=Cycle 1 Day 1
Missing data for intermediate visits are imputed using LOCF.

Source: Listing <u>16.2.6.4</u>

Programming Note: Continue for all visits (Day 1 for each odd-numbered cycle through Cycle 11), including CFB.

Table 14.2.3.2 WBC A3AR expression at Baseline by Overall Response ITT Population

| | | | CF102 | Placebo |
|---|---|---|---|---|
| Visit | Overall Response | Statistic | (N=xx) | (N=xx) |
| Cycle 3 Day 1 | CR | n | xx | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | PR | n | xx | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | XXX.X |
| | | Min, Max | xxx, xxx | XXX, XXX |
| | SD | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | PD | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| CFB at Cycle 3 Day 1 | CR | n | XX | xx |
| , | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | PR | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | SD | n | xx | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | PD | n | хх | хх |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |

Baseline=Cycle 1 Day 1
Missing data for intermediate visits are imputed using LOCF.

Source: Listings <u>16.2.6.3.1</u>, <u>16.2.6.4</u>

Programming Note: Continue for all visits (Day 1 for each odd-numbered cycle through Cycle 11), including CFB.

Table 14.2.3.3 Overall Response by CFB for WBC A3AR expression ITT Population

| | CFB for WBC A3AR | | CF102 | Placebo |
|---|---|---|---|---|
| Visit | expression | Overall Response (n, %) | (N=xx) | (N=xx) |
| Cycle 3 Day 1 | < xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | >= xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| Cycle 5 Day 1 | < xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | >= xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |

CFB=Change from Baseline

Baseline=Cycle 1 Day 1

Percentages are calculated using the number of subjects in the ITT Population for each treatment as the denominator. M=pooled median of CFB for WBC A3AR expression at the specified visit

Missing data for intermediate visits are imputed using LOCF.

Source: Listings <u>16.2.6.3.1</u>, <u>16.2.6.4</u>

Programming Notes: Continue for all visits (Day 1 for each odd-numbered cycle through Cycle 11). Specify the value of the median M (xxx.x) at each visit, followed by "(M)".

Table 14.2.4.1 Alpha-fetoproterin (AFP) ITT Population

| | | CF102 | Placebo |
|----------------------|-------------|----------------|----------------|
| Visit | Statistic | (N=xx) | (N=xx) |
| Cycle 1 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| Cycle 2 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| CFB at Cycle 2 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| | P-value (1) | 0.xxxx | |
| Cycle 3 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| CFB at Cycle 3 Day 1 | n | XX | XX |
| | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | XXX.X | XXX.X |
| | Min, Max | XXX, XXX | XXX, XXX |
| | P-value (1) | 0.xxxx | |

<sup>(1)</sup> P-value determined using ANCOVA with Baseline and Treatment in the model. CFB=Change from Baseline

Baseline=Cycle 1 Day 1
Missing data for intermediate visits are imputed using LOCF.

Source: Listing <u>16.2.6.4</u>

Programming Notes: Continue for all visits (Day 1 of each cycle through Cycle 11), including CFB. P-values are included with each CFB. AFP is collected with lab data. Exclude any data for days other than Day 1.

Table 14.2.4.2

Alpha-fetoproterin (AFP) by Overall Response ITT Population

| | | | CF102 | Placebo |
|---|---|---|---|---|
| Visit | Overall Response | Statistic | (N=xx) | (N=xx) |
| Cycle 3 Day 1 | CR | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | xxx, xxx | XXX, XXX |
| | PR | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | xxx, xxx | XXX, XXX |
| | SD | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | xxx, xxx | XXX, XXX |
| | PD | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |

CFB at Cycle 3 Day 1

Cycle 5 Day 1

CFB=Change from Baseline Baseline=Cycle 1 Day 1

Missing data for intermediate visits are imputed using LOCF.

Source: Listings <u>16.2.6.3.1</u>, <u>16.2.6.4</u>

Programming Notes: Continue for all visits (Day 1 for each odd-numbered cycle through Cycle 11), including CFB. AFP is collected with lab data.

Table 14.2.4.3 Overall Response by Categorical Alpha-fetoproterin (AFP) ITT Population

| | | | CF102 | Placebo |
|---|---|---|---|---|
| Visit | AFP (ng/mL) | Overall Response (n, %) | (N=xx) | (N=xx) |
| Cycle 3 Day 1 | <20 | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | 20-200 | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | >200 | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| Cycle 5 Day 1 | <20 | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | 20-200 | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | >200 | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | xx | xx |

Percentages are calculated using the number of subjects in the ITT Population in each category defined by AFP for each treatment as the denominator.

Missing data for intermediate visits are imputed using LOCF.

Source: Listings <u>16.2.6.3.1</u>, <u>16.2.6.4</u>

Programming Notes: Continue for all visits (Day 1 for each odd-numbered cycle). AFP is collected with lab data.

Table 14.2.4.4

Overall Response by CFB for Alpha-fetoproterin (AFP)

ITT Population

| • | | | CF102 | Placebo |
|---|---|---|---|---|
| Visit | CFB for AFP | Overall Response (n, %) | (N=xx) | (N=xx) |
| Cycle 3 Day 1 | <xxx.x (m)<="" td=""><td>CR</td><td>xx (xx.x)</td><td>xx (xx.x)</td></xxx.x> | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | >= xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| Cycle 5 Day 1 | < xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |
| | >= xxx.x (M) | CR | xx (xx.x) | xx (xx.x) |
| | | PR | xx (xx.x) | xx (xx.x) |
| | | SD | xx (xx.x) | xx (xx.x) |
| | | PD | xx (xx.x) | xx (xx.x) |
| | | Total | XX | XX |

CFB=Change from Baseline

Baseline=Cycle 1 Day 1

M=pooled median of CFB for AFP at the specified visit

Percentages are calculated using the number of subjects in the ITT Population in each category defined by

AFP for each treatment as the denominator.

Missing data for intermediate visits are imputed using LOCF.

Source: Listings <u>16.2.6.3.1</u>, <u>16.2.6.4</u>

Programming Notes: Continue for all visits (Day 1 for all odd-numbered cycles through Cycle 11). Specify the value of the median M (xxx.x) at each visit, followed by "(M)". AFP is collected with lab data.
Table 14.2.5.1

Alanine aminotransferase (ALT)

ITT Population

| | | CF102 | Placebo |
|-----------------------|-------------|------------------|------------------|
| Visit | Statistic | (N=xx) | (N=xx) |
| Pre-Study | n | XX | XX |
| - | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | Median | XXX.XX | XXX.XXX |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| Cycle 1 Day 1 | n | XX | XX |
| | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | Median | XXX.XX | XXX.XXX |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| Cycle 1 Day 8 | n | XX | XX |
| | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | Median | xxx.xx | XXX.XXX |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| CFB to Cycle 1 Day 8 | n | XX | XX |
| | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | Median | XXX.XX | XXX.XXX |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | P-value (1) | 0.xxxx | |
| Cycle 1 Day 15 | n | XX | XX |
| | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | Median | XXX.XX | XXX.XXX |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| CFB to Cycle 1 Day 15 | n | XX | XX |
| - | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | Median | xxx.xx | xxx.xxx |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | P-value (1) | 0.xxxx | |

<sup>(1)</sup> P-value determined using ANCOVA with Baseline and Treatment in the model.

Source: Listing 16.2.8.2

Programming Notes: Continue for remaining visits (Days 1 and 15 through Cycle 11), including CFB. P-values are included with each CFB. The following tables will use the above format: Table 14.2.5.2: Aspartate aminotransferase (AST), Table 14.2.5.3: Albumin, Table 14.2.5.4: Bilirubin (direct), Table 14.2.5.5: Bilirubin (total), Table 14.2.5.6: Prothrombin time (PT) with Source Listing 16.2.8.3, and Table 14.2.5.7: International Normalized Ratio (INR) with Source Listing 16.2.8.3

CFB=Change From Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing ) Missing data for intermediate visits are imputed using LOCF.

Table 14.2.6
Hepatitis Viral Load
ITT Population

| | | | CF102 | Placebo |
|---|---|---|---|---|
| Parameter | Visit | Statistic | (N=xx) | (N=xx) |
| log(HBV Load) | Cycle 1 Day 1 | n | xx | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | xxx, xxx | XXX, XXX |
| | Cycle 3 Day 1 | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | CFB to Cycle 3 Day 1 | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | | P-value (1) | 0.xxxx | |
| log(HCV Load) | Cycle 1 Day 1 | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | Cycle 3 Day 1 | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | CFB to Cycle 3 Day 1 | n | XX | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | | P-value (1) | 0.xxxx | |

<sup>(1)</sup> P-value determined using ANCOVA with Baseline and Treatment in the model.

Missing data for intermediate visits are imputed using LOCF.

Source: Listings <u>16.2.3.3.1</u>, <u>16.2.6.5.1</u>, <u>16.2.6.5.2</u>

Programming Notes: Include only subjects with positive serology at Screening; other subjects should not have data recorded. If subjects without positive serology have viral load recorded, include the values in Listings 16.2.6.5.1 and 16.2.6.5.2, but not in the table. Continue for all visits (Day 1 of odd-numbered cycles through Cycle 11), including CFB. P-values are included with each CFB.

Includes only subjects with positive serology at Screening (Listing 16.2.3.3.1)

HBV =Hepatitis B Viral; HCV =Hepatitis C Viral.

log (Value) is the base 10 logarithm of the value.

CFB= Change From Baseline

Baseline=Cycle 1 Day 1

Table 14.2.7.1 Overall Survival (OS; months) by Child-Pugh (CP) Score at Screening ITT Population

| CD Coore | Chablatia | CF102 | Placebo |
|-----------|----------------------------|--------------|-----------|
| CP Score | Statistic | (N=xx) | (N=xx) |
| CP= 7 | n<br>OStto Domonatilo | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | xx.x | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| CP=8 | n | XX | XX |
| CP=7 or 8 | n | XX | xx |
| CF=7 01 0 | 25th Percentile | | |
| | Median | XX.X<br>XX.X | XX.X |
| | 75th Percentile | | XX.X |
| | | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| CP=9 | n | XX | 0 |
| | 25th Percentile | XX.X | |
| | Median | XX.X | |
| | 75th Percentile | XX.X | |
| | Number (%) observed events | xx (xx.x) | |
| | Number (%) censored | xx (xx.x) | |

P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.3.1</u>, <u>16.2.5.1</u>

Programming Notes: Continue for CP=8.

For CP=9, do not include P-value (LR), HR, 95% CI for HR, and P-value (PH) and only enter 0 for 'n' for Placebo.

Figure 14.2.7.1

Kaplan-Meier curve for OS
CP Score at Screening = 7
ITT Population



Source: Listings <u>16.2.3.1</u>, <u>16.2.5.1</u>

Programming Note: Use same structure for Figures 14.2.7.2 (OS, CP=8) and 14.2.7.3 (OS, CP= 7 or 8).

Table 14.2.7.2 Overall Survival (OS; months) by Sex ITT Population

| | | CF102 | Placebo |
|--------|----------------------------|--------------|-----------|
| Sex | Statistic | (N=xx) | (N=xx) |
| Male | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| Female | n ` ' | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | , , |
| | HR `´ | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category

for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.3.1</u>, <u>16.2.5.1</u>

Table 14.2.7.3 Overall Survival (OS; months) by ECOG PS at Baseline ITT Population

| | | CF102 | Placebo |
|---------|----------------------------|--------------|-----------|
| ECOG PS | Statistic | (N=xx) | (N=xx) |
| 0 | n | xx | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| 1 or 2 | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

P-value (LR) =P-value using the logrank test.
Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.9.3</u>, <u>16.2.5.1</u>

Table 14.2.7.4 Overall Survival (OS; months) by Alpha-fetoprotein (AFP) at Baseline ITT Population

| | | CF102 | Placebo |
|-------------|----------------------------|--------------|-----------|
| AFP | Statistic | (N=xx) | (N=xx) |
| <=400 ng/mL | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| >400 ng/mL | n | XX | XX |
| _ | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | , , |
| | HR `´ | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <a href="16.2.6.4">16.2.6.4</a>, <a href="16.2.6.4">16.2.5.1</a>

Table 14.2.7.5 Overall Survival (OS; months) by Prior Locoregional Therapy ITT Population

| | | CF102 | Placebo |
|---|---|---|---|
| Prior Locoregional Therapy | Statistic | (N=xx) | (N=xx) |
| Yes | n | xx | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| No | n `´´ | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | , , |
| | HR `´ | x.xx | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

Locoregional Therapy = HCC Prior Therapies of Radiation or Chemoembolization

P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.3.4</u>, <u>16.2.5.1</u>

Table 14.2.7.6 Overall Survival (OS; months) by EHS, PVT, and Either EHS or PVT ITT Population

| | | | CF102 | Placebo |
|---|---|---|---|---|
| Parameter | Response | Statistic | (N=xx) | (N=xx) |
| EHS | Yes | n | XX | XX |
| | | 25th Percentile | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | 75th Percentile | XX.X | XX.X |
| | | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | | P-value (LR) | 0.xxx | |
| | | HR | X.XX | |
| | | 95% CI for HR | (x.xx, x.xx) | |
| | | P-value (PH) | 0.xxx | |
| | No | n | xx | XX |
| | | 25th Percentile | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | 75th Percentile | XX.X | XX.X |
| | | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | | P-value (LR) | 0.xxx | ` , |
| | | HR `´´ | x.xx | |
| | | 95% CI for HR | (x.xx, x.xx) | |
| | | P-value (PH) | 0.xxx | |
| PVT | Yes | n `´´ | XX | XX |
| | | 25th Percentile | XX.X | XX.X |
| Either EHS or PVT | Yes | n | xx | XX |
| | | 25th Percentile | XX.X | XX.X |

EHS= Extrahepatic Spread; PVT= Portal Vein Thrombosis P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.3.3.2</u>, <u>16.2.5.1</u>

Programming Note: Continue PVT= Yes and Either EHS or PVT= Yes, and add PVT= No and Either EHS or PVT= No.

Table 14.2.7.7 Overall Survival (OS; months) by History of HBV **ITT** Population

| | | CF102 | Placebo |
|----------------|----------------------------|--------------|-----------|
| History of HBV | Statistic | (N=xx) | (N=xx) |
| Yes | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| No | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

HBV =Hepatitis B Virus

P-value (LR) =P-value using the logrank test.

Percentages calculated using the number of subjects in the ITT Population in the specified subgroup category as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings 16.2.3.3.1, 16.2.5.1

Table 14.2.7.8 Overall Survival (OS; months) by History of HCV ITT Population

| | | CF102 | Placebo |
|----------------|----------------------------|--------------|-----------|
| History of HCV | Statistic | (N=xx) | (N=xx) |
| Yes | n | xx | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| No | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR `´ | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

HCV =Hepatitis C Virus

P-value (LR) =P-value using the logrank test.

Percentages calculated using the number of subjects in the ITT Population in the specified subgroup category as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.3.3.1</u>, <u>16.2.5.1</u>

Table 14.2.7.9 Overall Survival (OS; months) by Diagnostic Procedure ITT Population

| | | CF102 | Placebo |
|----------------------|----------------------------|--------------|-----------|
| Diagnostic Procedure | Statistic | (N=xx) | (N=xx) |
| Cytology/histology | n | xx | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| AASLD | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | ` , |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

Diagnostic Procedure= Cytology/histology or American Association for the Study of Liver Diseases (AASLD) P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square). Source: Listings <u>16.2.3.2</u>, <u>16.2.5.1</u>

Table 14.2.7.10

Overall Survival (OS; months) by Country ITT Population

| | | CF102 | Placebo |
|----------|----------------------------|--------------|-----------|
| Country | Statistic | (N=xx) | (N=xx) |
| Bulgaria | n | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |
| Israel | n ` ´ | XX | XX |
| | 25th Percentile | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | 75th Percentile | XX.X | XX.X |
| | Number (%) observed events | xx (xx.x) | xx (xx.x) |
| | Number (%) censored | xx (xx.x) | xx (xx.x) |
| | P-value (LR) | 0.xxx | |
| | HR `´ | X.XX | |
| | 95% CI for HR | (x.xx, x.xx) | |
| | P-value (PH) | 0.xxx | |

P-value (LR) =P-value using the logrank test.

Percentages are calculated using the number of subjects in the ITT Population in the specified subgroup category for each treatment as the denominator.

HR=Hazard Ratio for Treatment from Proportional Hazards Model with Treatment as the only factor in the model and P-value (PH) is the corresponding p-value (Chi-Square).

Source: Listings <u>16.2.1.1</u>, <u>16.2.5.1</u>

Programming Note: Continue for each country (Bulgaria, Israel, Romania, Serbia, or United States) alphabetically.

Table 14.3.1 Incidence of Treatment-Emergent Adverse Events Safety Population

| MedDRA System Organ Class | MedDRA Preferred Term, n (%) | CF102<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| Any | Any | xx (xx.x) | xx (xx.x) |
| Body as a Whole | Any | xx (xx.x) | xx (xx.x) |
| | Fever | xx (xx.x) | xx (xx.x) |

All AEs in this table are treatment emergent. Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

MedDRA version: 21.0 Source: Listing 16.2.7

Programming Note: Continue for all SOCs and Preferred Terms.

Table 14.3.2 Incidence of Treatment-Emergent Adverse Events by Relationship Safety Population

| MedDRA System Organ Class | MedDRA Preferred Term | Relationship, n (%) | CF102<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| | | | , , | , , |
| Any | Any | Definitely Related | xx (xx.x) | xx (xx.x) |
| | | Probably Related | xx (xx.x) | xx (xx.x) |
| | | Possibly Related | xx (xx.x) | xx (xx.x) |
| | | Not Related | xx (xx.x) | xx (xx.x) |
| Body as a Whole | Any | Definitely Related | xx (xx.x) | xx (xx.x) |
| • | - | Probably Related | xx (xx.x) | xx (xx.x) |
| | | Possibly Related | xx (xx.x) | xx (xx.x) |
| | | Not Related | xx (xx.x) | xx (xx.x) |
| | Fever | Definitely Related | xx (xx.x) | xx (xx.x) |
| | | Probably Related | xx (xx.x) | xx (xx.x) |
| | | Possibly Related | xx (xx.x) | xx (xx.x) |
| | | Not Related | xx (xx.x) | xx (xx.x) |

All AEs in this table are treatment emergent.

Relationship is the most related AE for each MedDRA System Organ Class and Preferred Term for each subject.

Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

MedDRA version: 21.0 Source: Listing 16.2.7

Programming Notes: Continue for all SOCs and Preferred Terms. Include "Possibly Related" and "Not Related" for all SOCs and PTs; include "Definitely Related" and "Probably Related" for SOCs and PTs when such are recorded for relationship.

Table 14.3.3
Incidence of Treatment Emergent Adverse Events By Severity
Safety Population

| MedDRA System Organ Class | MedDRA Preferred Term | Severity, n (%) | CF102<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Any | Any | Mild | xxx (xx.x) | xxx (xx.x) |
| | | Moderate | xxx (xx.x) | xxx (xx.x) |
| | | Severe | xxx (xx.x) | xxx (xx.x) |
| Body as a Whole | Any | Mild | xxx (xx.x) | xxx (xx.x) |
| , | • | Moderate | xxx (xx.x) | xxx (xx.x) |
| | | Severe | xxx (xx.x) | xxx (xx.x) |
| | Fever | Mild | xxx (xx.x) | xxx (xx.x) |
| | | Moderate | xxx (xx.x) | xxx (xx.x) |
| | | Severe | xxx (xx.x) | xxx (xx.x) |

All AEs in this table are treatment emergent.

Severity is the most severe AE, i.e. largest severity grade, for each MedDRA System Organ Class and Preferred Term for each subject. Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

MedDRA version: 21.0 Source: Listing 16.2.7

Programming Notes: Continue for all SOCs and Preferred Terms.AE severity is recorded using grade. Display as Mild, Moderate, Severe, Life-Threatening, or Fatal for Grade 1, Grade 2, Grade 3, Grade 4, or Grade 5, respectively. Include Mild or Moderate for all SOCs and PTs and include Severe, Life-Threatening, or Fatal only for those SOCs and PTs when such are recorded for severity (i.e. with severity of Grades 3, 4 or 5, respectively).

Table 14.3.4.1

Listing of Deaths Safety Population

| Site/<br>Subject | Treatment | Last Visit | Date of<br>Final Dose | Date of Death | Primary Cause of Death | Autopsy<br>Performed? | Date of Autopsy |
|---|---|---|---|---|---|---|---|
| xxx/xxxx<br>xxx/xxxx | xxxxxxxx | xx<br>xx | DD/MM/YY<br>DD/MM/YY | DD/MM/YY<br>DD/MM/YY | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxx<br>xxxx | DD/MM/YY<br>DD/MM/YY |

Includes subjects who discontinued from dosing or discontinued from the study for termination reason of death. All deaths are given in <u>Listing 16.2.5.1</u>. Source: Listings <u>16.2.1.1</u>, <u>16.2.5.1</u>, <u>16.2.5.7</u>

Table 14.3.4.2
Listing of Serious Adverse Events
Safety Population

| Site/<br>Subject | Treatment | System Organ Class /<br>Preferred Term/<br>Verbatim Term | Start<br>Date | Stop<br>Date (1) | Relative<br>Start Day | | Severity (2) | Freq. | Relation<br>(4) | Action<br>Taken<br>(5) | Outcome<br>(6) | Serious? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxx | xxxxx | xxxxxx /<br>xxxxxx/<br>xxxxxxx | DD/MM/YY | DD/MM/YY | xx | xx | х | Х | х | х | Х | Х |
| xxx/xxxx | xxxxx | xxxxxx/<br>xxxxxx/<br>xxxxxxx | DD/MM/YY | DD/MM/YY | XX | XX | х | X | Х | X | X | х |

Relative Start / Stop Dates = Days from Baseline to Start / Stop

- (1) O=AE ongoing
- (2) Severity: 1= Mild, 2= Moderate, 3= Severe but not immediately life-threatening, 4= Life-threatening consequences, 5=Death
- (3) Frequency: 1= Single episode 2= Intermittent 3= Continuous
- (4) Relationship: 1= Definitely related 2= Probably related 3= Possibly related 4= Not related
- (5) Action Taken: 0= None 1= Medication TX 2= Non-medication TX 3= Hospitalization 4= Study drug delayed, 5= Study drug discontinued
- (6) Outcome: 1= Resolved 2= Resolved with sequelae 3= Unresolved 4= Death

MedDRA version: 21.0

Source: Listing 16.2.7

Programming Note: Sort by site, subject and start date.

Table 14.3.5

# Listing of Discontinuations Due to Adverse Events Safety Population

| Site/ | | Date of | Date of Withdrawal from Trial | | |
|---|---|---|---|---|---|
| Subject | Treatment | Final Dose | or Dosing | Primary Reason | Specify |
| xxx/xxxx | XXXXXXXX | DD/MM/YY | DD/MM/YY | xxxxxxxxxxxxxxxx | XXX |

Includes only subjects with AE recorded as reason for withdrawal from dosing or trial Source: Listings <a href="16.2.1.1">16.2.1</a>, <a href="16.2.1.1">16.2.7</a>

Table 14.3.6.1

Clinical Laboratory Evaluations: Hematology
Safety Population

| Parameter (Units) | Visit | Statistic | CF102<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| XXXXXXXXX | Pre-Study | n | XX | (N-XX) |
| | Fie-Study | | | |
| (UNITS) | | Mean(SD)<br>Median | xxx.xx (xxx.xxx) | XXX.XX (XXX.XXX) |
| | | | XXX.XX | XXX.XXX |
| | Cycle 4 Day 4 | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Cycle 1 Day 1 | n<br>M (OD) | XXX | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Cycle 1 Day 8 | n | XXX | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | CFB to Cycle 1 Day 8 | n | XXX | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | xxx.xx | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | XXXXX | n | xxx | xxx |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | xxx.xx | xxx.xxx |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | CFB to xxxxx | n | XXX | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |

CFB=Change From Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Includes visits with at least 4 subjects in either treatment group

Source: Listing 16.2.8.1

Programming Notes: Continue for all parameters and all visits (Days 1, 8, and 15 for Cycle 1, and Days 1 and 15 for subsequent cycles), including CFB. Include visits with at least 4 subjects in either treatment group. The following tables will use the above format:

Table 14.3.6.2 Clinical Laboratory Evaluations: Blood Chemistry (Safety Population) with Source: Listing 16.2.8.2 and

Table 14.3.6.3 Clinical Laboratory Evaluations: Coagulation (Safety Population) with Source: Listing 16.2.8.3.

Table 14.3.6.4 Clinical Laboratory Evaluations: Thyroid Function Safety Population

| Darameter (Unite) | \/ioit | Ctatiatia | CF102 | Placebo |
|---|---|---|---|---|
| Parameter (Units) | Visit | Statistic | (N=xx) | (N=xx) |
| Γ3 (Unit) | Pre-Study | n | XX | XX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Cycle 1 | n | XXX | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | XXX.XX (XXX.XXX) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Cycle 2 | n | XXX | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | CFB to Cycle 2 | n | xxx | XXX |
| | • | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | XXXXX | n | XXX | xxx |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | CFB to xxxxx | n ´ | xxx | XXX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |

CFB=Change From Baseline

Baseline=Cycle 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing) Includes visits with at least 4 subjects in either treatment group

Source: Listing <u>16.2.8.5</u>

Programming Note: Continue for T4 (Unit) and TSH (Unit) and all cycles with at least 4 subjects in either treatment group.

Table 14.3.7.1

ECOG Performance Status
Safety Population

| | | CF102 | Placebo |
|---------------|----------------|-----------|-----------|
| Visit | ECOG PS, n (%) | (N=xx) | (N=xx) |
| Pre-Study | 0 | xx (xx.x) | xx (xx.x) |
| - | 1 | xx (xx.x) | xx (xx.x) |
| | 2 | xx (xx.x) | xx (xx.x) |
| | 3 | xx (xx.x) | xx (xx.x) |
| | 4 | xx (xx.x) | xx (xx.x) |
| | Total | xx | XX |
| Cycle 1 Day 1 | 0 | xx (xx.x) | xx (xx.x) |
| | 1 | xx (xx.x) | xx (xx.x) |
| | 2 | xx (xx.x) | xx (xx.x) |
| | 3 | xx (xx.x) | xx (xx.x) |
| | 4 | xx (xx.x) | xx (xx.x) |
| | Total | xx | XX |
| Cycle 2 Day 1 | 0 | xx (xx.x) | xx (xx.x) |
| | 1 | xx (xx.x) | xx (xx.x) |
| | 2 | xx (xx.x) | xx (xx.x) |
| | 3 | xx (xx.x) | xx (xx.x) |
| | 4 | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx |
| Cycle 3 Day 1 | 0 | xx (xx.x) | xx (xx.x) |
| | 1 | xx (xx.x) | xx (xx.x) |
| | 2 | xx (xx.x) | xx (xx.x) |
| | 2<br>3 | xx (xx.x) | xx (xx.x) |
| | 4 | xx (xx.x) | xx (xx.x) |
| | Total | xx | xx |

0=Normal activity, 1=Symptoms but ambulatory, 2= In bed <50% of time, 3=In bed >50% of time, 4=100% bedridden Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing) Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator. Includes visits with at least 4 subjects in either treatment group Source: Listing 16.2.9.3

Programming Notes: Continue for all cycles with at least 4 subjects in either treatment group. Include '4' only for cycles with a non-zero frequency for at least one treatment.

Table 14.3.7.2 Change from Baseline in ECOG Performance Status Safety Population

| | CFB in | CF102 | Placebo |
|---------------|----------------|-----------|-----------|
| Visit | ECOG PS, n (%) | (N=xx) | (N=xx) |
| Cycle 2 Day 1 | Decrease | xx (xx.x) | xx (xx.x) |
| | No Change | xx (xx.x) | xx (xx.x) |
| | Increase | xx (xx.x) | xx (xx.x) |
| | Total | XX | XX |
| Cycle 3 Day 1 | Decrease | xx (xx.x) | xx (xx.x) |
| • | No Change | xx (xx.x) | xx (xx.x) |
| | Increase | xx (xx.x) | xx (xx.x) |
| | Total | XX | XX |

CFB=Change from Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator. Includes visits with at least 4 subjects in either treatment group

Source: Listing 16.2.9.3

Programming Note: Continue for all visits (Day 1 for all cycles) with at least 4 subjects in either treatment group.

Table 14.3.8

Vital Signs And Weight Safety Population

| Parameter (Units) | Visit | Statistic | CF102<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| | | | , | , , |
| Systolic BP (mmHg) | Pre-Study | n (OD) | XX | XX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | XXX.XX | XXX.XXX |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Baseline | n | XX | XX |
| | | Mean(SD) | xxx.xx (xxx.xxx) | xxx.xx (xxx.xxx) |
| | | Median | xxx.xx | xxx.xxx |
| | | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Cycle 1 Day 1 | | | |
| | Hour 1 | n | xx | XX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | xxx, xxx | XXX, XXX |
| | CFB to | , | 7001, 7001 | 7001, 7001 |
| | Cycle 1 Day 1 Hour 1 | n | XX | XX |
| | Cycle : Bay i riour i | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |

BP=Blood Pressure

BMI=Body mass index

CFB= Change From Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Includes visits with at least 4 subjects in either treatment group

Source: Listings 16.2.9.1, 16,2.9.2

Programming Notes: Continue for Diastolic BP (mmHg), Pulse (beats/min), Temperature (deg C), Respiratory Rate (/min), Weight (kg), and BMI (kg/m2) and visits (Days 1 and 15 of each cycle, Day 8 of Cycle 1, and Hours 1, 2, 3, 4, 6 and 8 on Cycle 1 Day 1) with CFB. Weight (kg) is not recorded at Hours 1, 2, 3, 4, 6 and 8 on Cycle 1 Day 1. Include visits with at least 4 subjects in either treatment group.

Table 14.3.9.1 Electrocardiogram (ECG) Parameters Safety Population

| _ | | | CF102 | Placebo |
|---|---|---|---|---|
| Parameter | Visit | Statistic | (N=xx) | (N=xx) |
| Heart Rate (bpm) | Pre-Study | n | XXX | XXX |
| (25) | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | Baseline | n | XXX | XXX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | Cycle 1 Day 1 Hour 2 | n | XXX | XXX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | CFB to Cycle 1 Day 1 Hour 2 | n | XXX | XXX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| QTcF (msec) (1) | Pre-Study | n | xxx | XXX |
| | · | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | XXX.X |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | Baseline | n | xxx | XXX |
| | | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | XXX.X | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | Cycle 1 Day 1 Hour 2 | n | xxx | XXX |
| | • | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |
| | CFB to Cycle 1 Day 1 Hour 2 | n | XXX | xxx |
| | , , | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | | Median | xxx.x | xxx.x |
| | | Min, Max | XXX, XXX | XXX, XXX |

<sup>(1)</sup> QTcF= QT Correction- Fridericia

Programming Notes: Continue for QRS Complex (msec), PR Interval (msec), and QTcF (msec) in that order and all visits (pre-Study, pre-dose at all visits, and at 2, 4, and 6 hours post-dose on Days 1 and 8 of Cycle 1) with CFB. Compute QTcF=QT\*(HR/60)<sup>1/3</sup>. Include visits with at least 4 subjects in either treatment group.

CFB= Change From Baseline

Baseline=Cycle 1 Day 1 Hour 0 (or Pre-Study if value at Cycle 1 Day 1 is missing) Includes visits with at least 4 subjects in either treatment group Source: Listing 16.2.10.1

Table 14.3.9.2

Categorical Electrocardiogram (ECG) Parameters
Safety Population

| | | | CF102 | Placebo |
|---|---|---|---|---|
| Parameter | Visit | Response, n (%) | (N=xx) | (N=xx) |
| Overall Impression | Pre-Study | Normal | XXX (XX.X) | xxx (xx.x) |
| • | · | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | XX | XX |
| | Baseline | Normal | XXX (XX.X) | xxx (xx.x) |
| | | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | XX | XX |
| | Cycle 1 Day 1 Hour 2 | Normal | xxx (xx.x) | xxx (xx.x) |
| | · • | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | XX | XX |
| | Cycle 1 Day 1 Hour 4 | Normal | xxx (xx.x) | xxx (xx.x) |
| | | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | XX | XX |
| | Cycle 1 Day 1 Hour 6 | Normal | XXX (XX.X) | xxx (xx.x) |
| | | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | XX | XX |
| | Cycle 1 Day 8 Pre-Dose | Normal | xxx (xx.x) | xxx (xx.x) |
| | | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | XX | XX |
| | Cycle 1 Day 8 Hour 2 | Normal | xxx (xx.x) | xxx (xx.x) |
| | - | NCS | xxx (xx.x) | xxx (xx.x) |
| | | CS | xxx (xx.x) | xxx (xx.x) |
| | | Total | xx | XX |

NCS= Abnormal-not clinically significant (NCS)

CS= Abnormal-clinically significant (CS)

Baseline=Cycle 1 Day 1 Hour 0 (or Pre-Study if value at Cycle 1 Day 1 is missing)

Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

Includes visits with at least 4 subjects in either treatment group

Source: Listing 16.2.10.2.

Programming Notes: Continue for ST Segment and Cardiac Rhythm (Normal, Abnormal, and Total) and all visits (Pre-Study visit, Days 1 and 15 of all cycles, Day 8 of Cycle 1, and at 2, 4, and 6 hours post-dose on Day 1 of Cycle 1, and at Follow-up). Include visits with at least 4 subjects in either treatment group.

Table 14.3.10.1 Physical Examination at Pre-Study Visit Safety Population

| | | CF102 | Placebo |
|--------------------------|-----------------|------------|------------|
| Body System | Response, n (%) | (N=xx) | (N=xx) |
| General Appearance | Normal | xxx (xx.x) | XXX (XX.X) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx | XXX |
| Head and Neck | Normal | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx | XXX |
| Eyes, Ears, Nose, Throat | Normal | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |
| Skin | Normal | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx | XXX |
| Chest / Lungs / Breast | Normal | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx | XXX |
| Heart | Normal | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | xxx |
| Neurological | Normal | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |
| Other (1) | Normal | xxx (xx.x) | xxx (xx.x) |
| (-, | Abnormal | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |

(1) Subjects with more than one assessment of "Other" are counted once. Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

Abnormalities are provided in the listing.

Source: Listing <u>16.2.11 .1</u>

Programming Notes: Include other body systems. Subjects with more than one assessment of "Other" are counted once. Do not include "Not Assessed".

Table 14.3.10.2 Physical Examination Safety Population

| Visit | Clin. Sig. | CF102 | Placebo |
|----------------|--------------------|------------|------------|
| | Changes (1), n (%) | (N=xx) | (N=xx) |
| Cycle 1 Day 1 | Yes | XXX (XX.X) | XXX (XX.X) |
| | No | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |
| Cycle 1 Day 8 | Yes | xxx (xx.x) | xxx (xx.x) |
| | No | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |
| Cycle 1 Day 15 | Yes | xxx (xx.x) | xxx (xx.x) |
| | No | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |
| Cycle 2 Day 1 | Yes | xxx (xx.x) | XXX (XX.X) |
| | No | xxx (xx.x) | xxx (xx.x) |
| | Total | XXX | XXX |
| Cycle 2 Day 15 | Yes | xxx (xx.x) | xxx (xx.x) |
| | No | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx | XXX |

<sup>(1)</sup> Are there any clinically significant changes from the physical examination conducted at the previous assessment?

Source: Listing <u>16.2.11.2</u>

Programming Note: Continue for all visits (Days 1, 8, and 15 of Cycle 1 and Days 1 and 15 of subsequent cycles) with at least 4 subjects in either treatment group.

Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

Abnormalities associated with clinically significant changes are provided in the listing. Includes visits with at least 4 subjects in either treatment group

Table 14.3.11 **Prior and Concomitant Medications** Safety Population

| | CF102 | Placebo |
|--------------------------|-----------|-----------|
| ATC Level 3 Class, n (%) | (N=xx) | (N=xx) |
| None | xx (xx.x) | xx (xx.x) |
| Class 1 | xx (xx.x) | xx (xx.x) |
| Class 2 | xx (xx.x) | xx (xx.x) |

Includes medications taken within 30 days prior to Screening Visit.

Percentages are calculated using the number of subjects in the Safety Population for each treatment as the denominator.

Sum of percentages may exceed 100% because subjects could take Concomitant Medications within more than one ATC Level 3 Class.

Source: Listing 16.2.12

Programming Note: Continue for all observed Therapeutic Classes Individual medications are not tabulated; only the ATC Level 3 Class. Check that no subject has "None" for Complications with another response.

# 4.2. Listing Examples

Listing 16.2.1.1

Completed and Discontinued Subjects with Primary Reason for Withdrawal

| | | | | | Withdrawn | | Primary Reason for | Primary Reason | |
|---|---|---|---|---|---|---|---|---|---|
| Site/ | | | Date of | Complete | from dosing | Date of Early | Withdrawal from | for Withdrawal | Specify / |
| Subject | Country | Treatment | Final Dose | 6 Months? | or from trial? | Termination | Dosing | from Trial | Comment |
| xxx/xxxx | XXXXXXX | XXXXXX | DD/MM/YY | No | Yes | DD/MM/YY | XXXXXXXX | | |
| xxx/xxxx | XXXXXX | XXXXXX | DD/MM/YY | Yes | Yes | DD/MM/YY | | XXXXXXX | |
| xxx/xxxx | XXXXXX | XXXXXX | DD/MM/YY | Yes | No | | | | |
| xxx/xxxx | XXXXXXX | XXXXXXX | DD/MM/YY | No | Yes | DD/MM/YY | | XXXXXXX | XXXXXXX |

Country is based on the first digit of the site number (1=Bulgaria, 2=Serbia, 3=Israel, 5=Romania, or 7=United States). Further information regarding deaths is given in Table 14.3.4.1.

Programming Notes: For Primary Reason for Withdrawal from Dosing, use:

"Grade 3", "Grade 4", "> 1 dose reduction", "Delay > 14 days", "Withdrawal of consent", "Withdrawal of subject by Investigator", "Intercurrent illness", "Pregnancy", "Noncompliance", or "Termination of the trial by Sponsor".

For Primary Reason for Withdrawal from Trial, use: "Withdrawal of consent", "Termination of the trial by Sponsor", "Death", or "Other". The response to "Specify / Comment" is the text description for

Primary Reason for Withdrawal from Dosing = "Grade 3", "Grade 4", or "Withdrawal of subject by Investigator", or Primary Reason for Withdrawal from Trial = 'Other', or 'Comments' at the end of the "Termination" module.

Subjects should have response to either Primary Reason for Withdrawal from Dosing or Primary Reason for Withdrawal from Trial, but not BOTH. Sort listing by site and subject. Present country as Bulgaria, Serbia, Israel, Romania, or United States.

Listing 16.2.1.2

Subjects Excluded from Analysis Populations

| | | Excluded from | Excluded from | |
|---|---|---|---|---|
| Site/ Subject Tr | reatment | ITT Population? | PP Population? | Reason for Exclusion |
| xxx/xxxx xx | XXXXXX | No | Yes | XXXXXXX |
| xxx/xxxx xx | XXXXXX | Yes | Yes | XXXXXXX |

Includes only subjects excluded from the ITT or PP Population.
All subjects excluded from the ITT Population are also excluded from the PP Population.

ITT= Intent-to-Treat

PP=Per Protocol

Programming Notes: Include only subjects excluded from ITT or PP Population.
All subjects excluded from the ITT Population are also excluded from the PP Population.

Listing 16.2.2.1

Inclusion Criteria

| Site/<br>Subject | Treatment | Consent Date | Date of<br>Screening<br>Visit | IN1 | IN2 | IN3 | IN4 | IN5 | IN6 | IN7 | IN8 | IN9 | IN10 | IN11 | IN12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | DD/MM/YYYY | DD/MM/YY | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |
| xxx/xxxx | XXXXX | DD/MM/YYYY | DD/MM/YY | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |

See last page for list of criteria.

Programming Note: Place the criteria definitions on the last page(s).

# Listing 16.2.2.1

Inclusion Criteria

#### Inclusion Criteria Questions

IN1= Males and females at least 18 years of age.

IN2= Diagnosis of HCC:

- For patients without underlying cirrhosis at the time of diagnosis, diagnosis of HCC documented by cytology and/or histology.
- For patients with underlying cirrhosis at the time of diagnosis, diagnosis of HCC established according to the American Association for the Study of Liver Diseases Practice Guideline algorithm.

IN3= HCC is advanced, ie, treatment-refractory or metastatic, and no standard therapies are expected to be curative.

IN4= Receipt of prior sorafenib therapy for at least 3 weeks and withdrawal from treatment due either to:

- a) Intolerability; If treatment was withdrawn due to intolerability manifested as a Grade 3 or 4 event by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE v4.0), less than 3 weeks of continuous prior administration prior to withdrawal is acceptable (see also Exclusion Criterion #3). Or;
- b) Radiographic evidence of disease progression.

IN5= Prior sorafenib treatment was discontinued for at least 2 weeks prior to the Baseline Visit.

IN6= Eastern Collaborative Oncology Group (ECOG) performance status (PS) of ≤ 2.

IN7= Cirrhosis classified as Child-Pugh Class B.

IN8= The following laboratory values must be documented within 3 days prior to the first dose of study drug:

- Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
- Platelet count ≥ 75 x 10^9/L
- Serum creatinine ≤2.0 mg/dL
- Aspartic aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × upper limit of normal (ULN)
- Total bilirubin ≤ 3.0 mg/dL.
- Serum albumin ≥ 2.8 g/dL.
- Prothrombin time (PT) no greater than 6 seconds longer than control.

IN9= Life expectancy of ≥ 6 weeks.

IN10= For women of childbearing potential, negative serum pregnancy test result.

IN11= Provide written informed consent to participate.

IN12= Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other trial related procedures.

Listing 16.2.2.2

Exclusion Criteria

| Site/<br>Subject | Treatment | EX1 | EX2 | EX3 | EX4 | EX5 | EX6 | EX7 | EX8 | EX9 | EX10 | EX11 | EX12 | EX13 | EX14 | EX15 | EX16 | EX17 | EX18 | EX19 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXXX | N | N | N | N | N | N | N | N | N | N | N | N | N | N | N | N | N | N | N |
| xxx/xxxxx | XXXXX | N | Ν | Ν | Ν | N | N | Ν | Ν | Ν | Ν | N | Ν | Ν | Ν | N | Ν | Ν | N | N |

See last page for list of criteria.

Programming Note: Place the criteria definitions on the last page(s).

# Listing 16.2.2.2

#### **Exclusion Criteria**

## **Exclusion Criteria Questions:**

- EX1= Receipt of no, or of >1, prior systemic drug therapies for HCC.
- EX2= Any systemic cancer therapy, immunomodulatory drug therapy, immunosuppressive therapy, or corticosteroids > 20 mg/day prednisone or equivalent, within 14 days prior to the Baseline Visit or concurrently during the trial.
- EX3= Presence of an acute or chronic toxicity of prior chemotherapy that has not resolved to ≤ Grade 1, as determined by CTCAE v 4.0.
- EX4= Locoregional treatment within 4 weeks prior to the Baseline Visit.
- EX5= Major surgery or radiation therapy within 4 weeks prior to the Baseline Visit.
- EX6= Use of any investigational agent within 4 weeks prior to the Baseline Visit.
- EX7= Child-Pugh Class A or C cirrhosis, or hepatic encephalopathy.
- EX8= Occurrence of esophageal or other gastrointestinal hemorrhage requiring transfusion within 4 weeks prior to the Baseline Visit.
- EX9= Uncontrolled or clinically unstable thyroid disease, per judgment of the Principal Investigator.
- EX10= Active bacterial, viral, or fungal infection requiring systemic therapy or operative or radiological intervention.
- EX11= Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
- EX12= Liver transplant.
- EX13= Active malignancy other than HCC.
- EX14= Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4).
- EX15= Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
- EX16= History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females.
- EX17= Pregnant or lactating female.
- EX18= Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Investigator, are effective and adequate for the subject's circumstances while on study drug.
- EX19= Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward.
- EX20= Any severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the subject inappropriate for entry into this study.

Listing 16.2.3.1

Demographic and Baseline Characteristics

| Site/ Subject | Treatment | Age | Date of Birth | Origin | Sex | CP Score (1) |
|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | XX | DD/MM/YY | XXXXX | XXXXX | Х |
| xxx/xxxx | XXXXX | XX | DD/MM/YY | XXXXX | XXXXX | X |

(1) CP Score= Child- Pugh Score at Screening

Programming Note: Compute Age as (the number of days from Date of Birth to Date of Screening Visit)/365.25
Listing 16.2.3.2

HCC Diagnosis

| | | | | | If Diagnosis Established by |
|---|---|---|---|---|---|
| | | | Most recent relapse | Diagnosis | Cytology/histology, specify |
| Site/ Subject | Treatment | Diagnosis Date | and/or re-staging date | Established by (1) | histopathological diagnosis |
| xxx/xxxx | XXXXX | DD/MM/YY | DD/MM/YY | XXXXXX | XXXXXXXXXXX |
| xxx/xxxx | XXXXX | DD/MM/YY | DD/MM/YY | XXXXXX | |
| xxx/xxxx | XXXXX | DD/MM/YY | DD/MM/YY | XXXXXX | XXXXXXXXXXX |

<sup>(1)</sup> AASLD=American Association for the Study of Liver Diseases

Programming Note: If diagnosis was established by American Association for the Study of Liver Diseases, present as AASLD.

# Listing 16.2.3.3.1

**HCC History** 

| Site/<br>Subject | Treatment | Date of<br>Screening<br>Visit | Known History<br>of Viral<br>Hepatitis? | Date of<br>Diagnosis of<br>Hepatitis B | Date of<br>Diagnosis of<br>Hepatitis C | Hepatitis B<br>Virus<br>Serology | Date of Last<br>Hepatitis B<br>Testing | Hepatitis C<br>Virus<br>Serology | Date of Last<br>Hepatitis C<br>Testing | Complications (1) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | DD/MM/YY | Yes | DD/MM/YY | DD/MM/YY | XXXXXXXXXX | DD/MM/YY | XXXXXXXXXXX | DD/MM/YY | XXXXX |
| xxx/xxxx | XXXXX | DD/MM/YY | No | | | XXXXXXXXXX | DD/MM/YY | XXXXXXXXXX | DD/MM/YY | XXXXX |
| xxx/xxxx | XXXXX | DD/MM/YY | Yes | DD/MM/YY | DD/MM/YY | XXXXXXXXXX | | XXXXXXXXXX | DD/MM/YY | XXXXX |
| xxx/xxxx | XXXXX | DD/MM/YY | Yes | DD/MM/YY | | XXXXXXXXXX | DD/MM/YY | XXXXXXXXXX | DD/MM/YY | XXXXX |
| | | | | | | | | | | XXXXX |
| xxx/xxxx | XXXXX | DD/MM/YY | Yes | DD/MM/YY | DD/MM/YY | XXXXXXXXXX | DD/MM/YY | XXXXXXXXXX | DD/MM/YY | None |
| xxx/xxxx | XXXXX | DD/MM/YY | Yes | | DD/MM/YY | XXXXXXXXXX | DD/MM/YY | xxxxxxxxx | DD/MM/YY | XXXXX |

<sup>(1)</sup> Known complication(s) of cirrhosis and/or portal hypertension

Programming Notes: If date of last testing is missing, then the field should be blank. "Serology" should not be blank. If none of the specified responses, including Other, are selected for Complications, then the response should be reported as "None". If "Other, specify" is reported for complication, then report the specified details as the complication. If more than 1 complication is reported, then multiple lines per subject should be used. Date of Screening Visit must match that given in Listing 16.2.2.1.

Listing 16.2.3.3.2

Extrahepatic Spread (EHS) and Portal Vein Thrombosis (PVT)

| Site/ Subject | Treatment | EHS | PVT | Either EHS or PVT | Both EHS and PVT |
|---------------|-----------|-----|-----|-------------------|------------------|
| xxx/xxxx | XXXXX | XXX | XXX | XXX | XX |
| xxx/xxxx | XXXXX | XXX | XXX | XXX | XX |

EHS = Extrahepatic Spread, PVT = Portal Vein Thrombosis

Programming Notes: Record each response as "Yes", "No", or "Unknown". Include only subjects with one of these responses recorded.

# Listing 16.2.3.4

## **HCC** Prior Therapies

| Site/ Subject | Treatment | Modality<br>Code (1) | Modality Details | Intent (2) | Best response to treatment | If Intent="Other",<br>Specify | Start Date | Stop Date |
|---|---|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | XX | XXXXXXXXXXXXXXX | XX | XX | | DD/MM/YY | DD/MM/YY |
| xxx/xxxx | XXXXX | XX | XXXXXXXXXXXXXXX | XX | XX | XXXXXXXX | DD/MM/YY | DD/MM/YY |

Programming Note: There may be multiple lines per subject.

<sup>(1)</sup> Modality Codes: 01 = Surgery, 02 = Radiation, 03 = Chemotherapy, 04 = Immunotherapy, 05 = Hormonal therapy,

<sup>06 =</sup> Targeted Therapy (sorafenib), 07 = Chemoembolization, 08 = Anti-viral therapy, 09 = Other
(2) Intent Codes: 01 = Curative / Palliative, 02 = Adjuvant, 03 = Neo adjuvant, 04 = Diagnostic, 05 = Therapy of Viral Hepatitis, 06 = Therapy for Complication of Portal Hypertension, 09 = Other (specify)

<sup>06 =</sup> Therapy for Complication of Portal Hypertension, 09 = Other (specify)
(3) Best Response Codes: 01 = CR – Complete Response; 02 = PR – Partial Response; 03 = PD – Progressive Disease; 04 = SD – Stable Disease; 09 = Unknown

Listing 16.2.3.5
Cirrhosis / Virus Complications and Treatment

| | | Modality | | | | |
|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Code (1) | Modality Details | Intent (2) | Start Date | Stop Date |
| xxx/xxxx | XXXXX | XX | XXXXXXXXXXXXXXX | XXXXXX | DD/MM/YY | DD/MM/YY |

XXXXXXXXXXXXXX

XXXXXX

DD/MM/YY

DD/MM/YY

XX

Programming Note: There may be multiple lines per subject.

XXXXX

xxx/xxxx

<sup>(1)</sup> Modality Codes: 01 = Surgery, 02 = Radiation, 03 = Chemotherapy, 04 = Immunotherapy, 05 = Hormonal therapy, 06 = Targeted Therapy (sorafenib), 07 = Chemoembolization, 08 = Anti-viral therapy, 09 = Other

<sup>(2)</sup> Intent Codes: 01 = Curative / Palliative, 02 = Adjuvant, 03 = Neo adjuvant, 04 = Diagnostic, 05 = Therapy of Viral Hepatitis, 06 = Therapy for Complication of Portal Hypertension, 09 = Other (specify)

Listing 16.2.3.6

Medical History (Excluding Past HCC, Cirrhosis, and Viral Hepatitis-Related History)

| Site/ Subject | Treatment | Past findings or<br>surgery? (1) | Body System | Finding or Procedure | Start Date | Stop Date |
|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | Yes | XXXXXXXXX | XXXXXXXXXXX | DD/MM/YY | DD/MM/YY |
| | | | XXXXXXXXX | xxxxxxxxxxx | DD/MM/YY | DD/MM/YY |
| xxx/xxxx | XXXXX | Yes | XXXXXXXX | XXXXXXXXXXX | DD/MM/YY | DD/MM/YY |
| xxx/xxxx | XXXXX | No | | | | |
| xxx/xxxx | XXXXX | Yes | XXXXXXXX | XXXXXXXXXXX | DD/MM/YY | DD/MM/YY |

<sup>(1)</sup> Has the patient had any past medical findings or surgical procedures?

Programming Note: There may be multiple lines per subject.

Listing 16.2.4.1
Study Drug Accountability and Treatment Compliance

| Site/ Subject | Treatment | Total Number of<br>Capsules<br>Dispensed | Total Number of<br>Capsules<br>Returned | Date of<br>Final Dose (1) | Date of<br>Baseline<br>Visit | Treatment<br>Duration<br>(Days) | Compliance (%) |
|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXXX | XXX | XXX | DD/MM/YY | DD/MM/YY | XXX | XX.X |
| xxx/xxxxx | XXXXX | XXX | XXX | DD/MM/YY | DD/MM/YY | XXX | XX.X |

The numbers of capsules dispensed and returned by visit are in the next listing.

Programming Notes: Treatment Duration= date of final dose minus date of Baseline + 1.

Compliance (%) =100\*(total number of capsules dispensed over study - total number of capsules returned over study)/ (2\*treatment duration). Total number of capsules dispensed over study = 65\*sum of the Number of Bottles Dispensed from next listing.

Total number of capsules returned over study = 65\*sum of the Number of Unopened Bottles Returned from above table

+ sum of Number of capsules returned (open bottle) from next listing.

<sup>(1)</sup> Date of Last Recorded Visit for subjects who are ongoing.

Listing 16.2.4.2
Study Drug Accountability by Visit

| Site/ Subject | Treatment | Visit | Date | Treatment<br>Number | Number of<br>Bottles<br>Dispensed | Comments | Number of<br>unopened<br>bottles returned | Number of<br>capsules returned<br>(open bottle) | Comments |
|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXXX | Cycle 1 | xx/xxx/xxxxx | XXXX | XXX | XXXXXX | | | |
| | | Cycle 2 | xx/xxx/xxxxx | XXXX | XXX | XXXXXX | XXX | XXX | XXXXXXX |
| | | Cycle 3 | xx/xxx/xxxxx | XXXX | XXX | XXXXX | XXX | XXX | XXXXXXX |
| xxx/xxxxx | XXXXX | Cycle 1 | xx/xxx/xxxxx | XXXX | XXX | XXXXXX | | | |
| | | Cycle 2 | xx/xxx/xxxxx | XXXX | XXX | XXXXX | XXX | XXX | XXXXXXX |
| | | Cycle 3 | xx/xxx/xxxxx | XXXX | XXX | XXXXXX | XXX | XXX | XXXXXXX |
| | | Cycle 4 | xx/xxx/xxxxx | XXXX | XXX | XXXXXX | XXX | XXX | XXXXXXXX |

Programming Note: Continue for all cycles.

# Listing 16.2.5.1

#### Time to Event

| Site/ | | Date of | Progressive | | Date of | Date of First | Date of Last | OS | TTP | PFS |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | First Dose | Disease? | Death? | Death | Progression | Contact | (months) | (months) | (months) |
| xxx/xxxxx | XXXX | DD/MM/YY | Yes | Yes | DD/MM/YY | DD/MM/YY | DD/MM/YY | XX.X | XX.X | XX.X |
| xxx/xxxxx | XXXX | DD/MM/YY | Yes | No | | DD/MM/YY | DD/MM/YY | XX.X * | XX.X | XX.X |
| xxx/xxxxx | XXXX | DD/MM/YY | No | No | | | DD/MM/YY | XX.X * | XX.X * | XX.X * |
| xxx/xxxxx | XXXX | DD/MM/YY | No | Yes | DD/MM/YY | | DD/MM/YY | XX.X | XX.X * | XX.X |

OS= Overall Survival (Time to Death due to any cause); TTP=Time to Progression; PFS= Progression-Free Survival (Time to Progression or Death) \* indicates censored value.

Programming Notes: If an event did not occur, leave the date of the event blank.

Date of Last Contact is the last date known to be alive in next listing.

Add \* for censored values, defined as follows.

OS is time to death due to any cause and is censored at date of last contact if death is not reported.

TTP is time to progression and is censored at date of last contact (including death) if progression is not reported.

PFS is time to progression or death and is censored at date of last contact if neither progression nor death is reported.

Listing 16.2.5.2 Survival Follow-up Contact Dates

| Site/ Subject | Treatment | Follow-up<br>Date | Is the Subject Alive? | Last date known to be alive | If not alive, date of death |
|---|---|---|---|---|---|
| xxx/xxxxx | XXXX | DD/MM/YY | XX | DD/MM/YY | DD/MM/YY |
| | | DD/MM/YY | XX | DD/MM/YY | DD/MM/YY |
| | | DD/MM/YY | XX | DD/MM/YY | DD/MM/YY |
| xxx/xxxxx | XXXX | DD/MM/YY | XX | DD/MM/YY | DD/MM/YY |
| | | DD/MM/YY | XX | DD/MM/YY | DD/MM/YY |
| | | DD/MM/YY | XX | DD/MM/YY | DD/MM/YY |

Includes all subjects who discontinue from dosing.

Programming Notes: Continue for all follow-up dates.

The CRF Page is to be completed for all subjects who discontinue from dosing.

Listing 16.2.6.1.1
Tumor Evaluations: Target Lesions

| Site/ | | | | Site | | Assessment | Method | Longest |
|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | Cycle | Lesion# | Code (1) | Description | Date | Code (2) | Diameter (LD) |
| xxx/xxxx | XXXXX | Screening | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | _ | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | Cycle 3 | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX | |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | Cycle 5 | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |

<sup>(1)</sup> Site Codes:

Programming Notes: Continue for all odd-numbered cycles.

Sort listing by lesion within cycle. There is one line for each target lesion.

#### Column "None?" has been deleted

It was intended only for cases with assessments made and there were no target lesions detected.

This would require "CR" for Target Lesions with disappearance of all Target Lesions; there were no such cases.

<sup>01 =</sup> Abdominal Wall, 02 = Adrenal, 03 = Bladder, 04 = Bone, 05 = Breast, 06 = CNS, 07 = Colon, 08 = Liver, 09 = Lung,

<sup>10 =</sup> Lymph Nodes, 11 = Pancreas, 12 = Pelvis, 13 = Pleura, 14 = Rectum, 15 = Retroperitoneal Cavity, 16 = Retroperitoneum, 17 = Small Intestine, 18 = Uterus, 99 = Other, specify

<sup>(2)</sup> Method Codes:

B = Bone Scan, C = Conventional CT scan, D = Direct Measure by Physical Exam, E = Endoscopy, L = Laparoscopy,

M = Magnetic Resonance Imaging, S = Spiral CT scan, U = Ultrasound, X = X-Ray, O = Other, specify

Listing 16.2.6.1.2
Summary of Target Lesions

| Site/ Subject | Treatment | Cycle | Sum of Longest Diameters (mm) | Smallest Sum<br>On Study (mm) | Percent<br>Change from<br>Smallest: | Screening<br>Sum on study | Percent Change<br>From Screening |
|---|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | Screening | XX | XX | XXX | XXX | XXX |
| | | Cycle 3 | XX | XX | XXX | XXX | XXX |
| | | Cycle 5 | XX | XX | XXX | XXX | XXX |
| xxx/xxxx | XXXXX | Screening | XX | XX | XXX | XXX | XXX |
| | | Cycle 3 | XX | XX | XXX | XXX | XXX |
| | | Cycle 5 | XX | XX | XXX | XXX | XXX |
| xxx/xxxx | XXXXX | Screening | XX | XX | XXX | XXX | XXX |
| | | Cycle 3 | XX | XX | XXX | XXX | XXX |
| | | Cycle 5 | XX | XX | XXX | XXX | XXX |
| | | Cycle 7 | XX | XX | XXX | XXX | XXX |

<sup>&</sup>quot;Smallest sum on study" at any visit refers to sums prior to, and including, the visit of interest, including the baseline sum of diameters.

Programming Notes: Continue for all odd-numbered cycles. There is one line for each cycle.

Column "None?" has been deleted

It was intended only for cases with assessments made and there were no target lesions detected.

This would require "CR" for Target Lesions with disappearance of all Target Lesions; there were no such cases.

Listing 16.2.6.2

Tumor Evaluations: Non-Target Lesions

| | | | | | Site | | Assessment | Method | |
|---|---|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Cycle | None? | Lesion# | Code (1) | Description | Date | Code (2) | Status |
| xxx/xxxx | XXXXX | Screening | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | Cycle 3 | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | Cycle 5 | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | Cycle 7 | None | | | | DD/MM/YY | | |
| | | Cycle 9 | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | - | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |
| | | | | XX | XX | XXXXXX | DD/MM/YY | XXX | XXX |

'None?' = 'None' if no non-target lesions were recorded

#### (2) Method Codes:

B = Bone Scan, C = Conventional CT scan, D = Direct Measure by Physical Exam, E = Endoscopy, L = Laparoscopy, M = Magnetic Resonance Imaging, S = Spiral CT scan, U = Ultrasound, X = X-Ray, O = Other, specify

Programming Notes: Continue for all odd-numbered cycles. Sort by lesion within cycle. There is one line for each non-target lesion.

<sup>(1)</sup> Site Codes:

<sup>01 =</sup> Abdominal Wall, 02 = Adrenal, 03 = Bladder, 04 = Bone, 05 = Breast, 06 = CNS, 07 = Colon, 08 = Liver, 09 = Lung, 10 = Lymph Nodes,

<sup>11 =</sup> Pancreas, 12 = Pelvis, 13 = Pleura, 14 = Rectum, 15 = Retroperitoneal Cavity, 16 = Retroperitoneum, 17 = Small Intestine, 18 = Uterus, 99 = Other, specify

Listing 16.2.6.3.1

Tumor Response

| Site/ Subject | Treatment | Cycle | Assessment<br>Date | Response:<br>Target<br>Lesions (1) | Response:<br>Non-Target<br>Lesions (2) | Comment | Overall<br>Response (3) | OR (4) | DC (5) | Best<br>Response (6) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXX | Cycle 3 | DD/MM/YY | XXX | xxx | | XXX | xxx | xxx | XXX |
| xxx/xxxxx | xxxx | Cycle 3 | DD/MM/YY | xxx | XXX | | xxx | XXX | XXX | |
| | | Cycle 5 | DD/MM/YY | XXX | xxx | | XXX | xxx | xxx | XXX |
| 530/006 | XXXX | Cycle 3 | DD/MM/YY | xxx | xxx | | xxx | XXX | xxx | |
| | | Cycle 5 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 7 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | XXX |
| | | Cycle 9 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 11 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 13 (7) | DD/MM/YY | PR | XXX | | PR | XXX | XXX | |
| | | Cycle 15 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 29 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |

Programming Notes: Continue for all odd-numbered cycles.

Use "Comment" for "Response: Non-Target Lesions" = "Unable to evaluate (NE)".

Record "Best Response" only at visit(s) at which it occurs.

<sup>(1)</sup> CR= Complete Response, PR= Partial Response, SD= Stable Disease, PD= Progressive Disease

<sup>(2)</sup> CR= Complete Response, PD= Progressive Disease, Non-CR/non-PD= Neither CR nor PD, NE= Not evaluated/ Unable to evaluate

<sup>(3)</sup> CR= Complete Response, PR= Partial Response, SD= Stable Disease, PD= Progressive Disease, Non-CR/non-PD= Neither CR nor PD, NE= Not evaluated/ Unable to evaluate

<sup>(4)</sup> OR= Objective Response= Overall Response of CR or PR (Yes or No)

<sup>(5)</sup> DC= Disease Control = Overall Response of CR, PR, or SD (Yes or No)

<sup>(6)</sup> Best Response = Best overall response recorded from the start of the study treatment until the end of study, in the order of CR, PR, SD, or PD from best to worst

<sup>(7)</sup> Subject 530/006 ay Cycle 13 had Response: Target Lesions that met RECIST criteria for both PR and PD, included above as PR.

Listing 16.2.6.3.2

Tumor Response (Investigator Assessments)

| Site/ Subject | Treatment | Cycle | Assessment<br>Date | Response:<br>Target<br>Lesions (1) | Response:<br>Non-Target<br>Lesions (2) | Comment | Overall<br>Response (3) | OR (4) | DC (5) | Best<br>Response (6 |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXX | Cycle 3 | DD/MM/YY | XXX | xxx | | xxx | XXX | XXX | XXX |
| xxx/xxxxx | xxxx | Cycle 3 | DD/MM/YY | XXX | xxx | | XXX | XXX | xxx | |
| | XXXX | Cycle 5 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | XXX |
| 530/006 | xxxx | Cycle 3 | DD/MM/YY | XXX | XXX | | xxx | XXX | xxx | |
| | | Cycle 5 | DD/MM/YY | XXX | XXX | | XXX | xxx | xxx | |
| | | Cycle 7 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | XXX |
| | | Cycle 9 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 11 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 13 (7) | DD/MM/YY | PR | XXX | | PD | XXX | XXX | |
| | | Cycle 15 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |
| | | Cycle 29 | DD/MM/YY | XXX | XXX | | XXX | XXX | XXX | |

Programming Notes: Continue for all odd-numbered cycles.

Use "Comment" for "Response: Non-Target Lesions" = "Unable to evaluate (NE)".

Record "Best Response" only at visit(s) at which it occurs.

Include Tumor Responses as recorded on CRF, including EOS Visit, the Follow-up Visit, and Unscheduled Visits.

<sup>(1)</sup> CR= Complete Response, PR= Partial Response, SD= Stable Disease, PD= Progressive Disease

<sup>(2)</sup> CR= Complete Response, PD= Progressive Disease, Non-CR/non-PD= Neither CR nor PD, NE= Not evaluated/ Unable to evaluate

<sup>(3)</sup> CR= Complete Response, PR= Partial Response, SD= Stable Disease, PD= Progressive Disease, Non-CR/non-PD= Neither CR nor PD, NE= Not evaluated/ Unable to evaluate

<sup>(4)</sup> OR= Objective Response= Overall Response of CR or PR (Yes or No)

<sup>(5)</sup> DC= Disease Control = Overall Response of CR, PR, or SD (Yes or No)

<sup>(6)</sup> Best Response = Best overall response recorded from the start of the study treatment until the end of study, in the order of CR, PR, SD, or PD from best to worst

<sup>(7)</sup> Subject 530/006 ay Cycle 13 had Response: Target Lesions that met RECIST criteria for both PR and PD, included above as PD.

Listing 16.2.6.4
Biomarkers: AFP and WBC A3AR

| | | | | alpha-fetoproterin | CFB in | WBC A3AR | CFB in WBC A3AR |
|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Cycle | Date | (AFP) (1) | AFP | Expression Level | Expression Level |
| xxx/xxxxx | XXXX | Baseline | DD/MM/YY | XXX | | XXX | |
| | | Cycle 2 | DD/MM/YY | XXX | XXX | | |
| | | Cycle 3 | DD/MM/YY | XXX | XXX | XXX | XXX |
| | | Cycle 4 | DD/MM/YY | XXX | XXX | | |
| | | Cycle 5 | DD/MM/YY | XXX | XXX | XXX | XXX |
| xxx/xxxxx | XXXX | Baseline | DD/MM/YY | XXX | | xxx | |
| | | Cycle 2 | DD/MM/YY | XXX | XXX | | |
| | | Cycle 3 | DD/MM/YY | XXX | XXX | XXX | XXX |
| | | Cycle 4 | DD/MM/YY | XXX | XXX | | |
| | | Cycle 5 | DD/MM/YY | xxx | XXX | xxx | xxx |

CFB=Change from Baseline
(1) H=Abnormal High, L=Abnormal Low
Normal ranges are given at the end of the listing.
Baseline=Cycle 1 Day 1

Programming Note: Continue for all cycles.

Listing 16.2.6.4

# Biomarkers: AFP and WBC A3AR Normal Ranges

| Parameter | Low | High |
|------------------|------------------------|------|
| AFP | | XX |
| Normal range for | WBC A3AR not specified | |

Listing 16.2.6.5.1

### Hepatitis B Viral Load

| | | | | Screening | Sample | Viral Load | | CFB in |
|---|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Visit | Date | Serology | Taken? (1) | (IU/mL) | Log (Viral Load) | Log (Viral Load) |
| xxx/xxxxx | XXXX | Baseline | DD/MM/YY | XXXXXXX | XXX | XXXXXX | XXXX.XX | |
| | | Cycle 3 | DD/MM/YY | | XXX | XXXXXX | XXXX.XX | XXXX.XX |
| | | Cycle 5 | DD/MM/YY | | XXX | XXXXXX | XXXX.XX | XXXX.XX |
| | | Cycle 7 | DD/MM/YY | | XXX | XXXXXX | XXXX.XX | XXXX.XX |

<sup>(1)</sup> Yes, No, or NA

Should include only subjects with positive serology at Screening, per protocol. Others are included if viral load was recorded (Listing 16.2.3.3). CFB=Change from Baseline Baseline=Cycle 1 Day 1

Log (Value) is the base 10 logarithm of the value.

Programming Notes: Continue for all odd-numbered cycles. Include Screening Serology as "Positive" or "Negative".

Listing 16.2.6.5.2

Hepatitis C Viral Load

| | | | | Screening | Sample | Viral Load | | CFB in |
|---|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Visit | Date | Serology | Taken? (1) | (IU/mL) | Log (Viral Load) | Log (Viral Load) |
| xxx/xxxxx | XXXX | Baseline | DD/MM/YY | XXXXXXX | XXX | XXXXXX | XXXX.XX | |
| | | Cycle 3 | DD/MM/YY | | XXX | XXXXXX | XXXX.XX | XXXX.XX |
| | | Cycle 5 | DD/MM/YY | | XXX | XXXXXX | XXXX.XX | XXXX.XX |
| | | Cycle 7 | DD/MM/YY | | XXX | XXXXXX | XXXX.XX | XXXX.XX |
| | | • | | | | | | |

(1) Yes, No, or NA

Should include only subjects with positive serology at Screening, per protocol. Others are included if viral load was recorded (Listing <u>16.2.3.3</u>). CFB=Change from Baseline

Baseline=Cycle 1 Day 1
Log (Value) is the base 10 logarithm of the value.

Programming Notes: Continue for all odd-numbered cycles. Include Screening Serology as "Positive" or "Negative".

**Listing 16.2.7** 

#### Adverse Events

| Site/<br>Subject | Treatment | System Organ Class /<br>Preferred Term/<br>Verbatim Term | Start Date | Stop Date (1) | Duration (2) | Severity<br>Grade (3) | Frequency (4) | Relation (5) | Action<br>Taken (6) | Outcome (7) | Serious? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | xxxxxx / | DD/MM/YY | DD/MM/YY | Х | Х | Х | Х | Х | Х | XX |
| xxx/xxxx | xxxxx | xxxxxx/<br>xxxxxxx<br>xxxxxx / | DD/MM/YY | DD/MM/YY | V | x | v | v | v | v | XX |
| **** | **** | XXXXXX/<br>XXXXXXXX | DD/IVIIVI/ I I | DD/WIW/TT | * | ^ | * | * | X | X | ** |

Sorted by Start Date, then alphabetically by SOC and Preferred Term within subject.

Programming Note: Sort by Start Date, then alphabetically by SOC and Preferred Term within subject for AEs starting on the same date.

<sup>(1)</sup> O=AE ongoing

<sup>(2)</sup> Duration (days)= Stop Date - Start Date + 1; Duration = Date of Last Dose - Start Date + 1 if AE is ongoing

<sup>(3)</sup> Severity Grade: 1=Mild, 2=Moderate, 3=Severe or medically significant but not immediately life-threatening, 4=Life-threatening consequences, or 5=Death related to AE.

<sup>(4)</sup> Frequency: 1= Single episode 2= Intermittent 3= Continuous

<sup>(5)</sup> Relationship: 1= Definitely related 2= Probably related 3= Possibly related 4= Not related

<sup>(6)</sup> Action Taken: 0= None 1= Medication TX 2= Non-medication TX 3= Hospitalization 4= Study drug delayed, 5= Study drug discontinued

<sup>(7)</sup> Outcome: 1= Resolved 2= Resolved with sequelae 3= Unresolved 4= Death

Listing 16.2.8.1 Clinical Laboratory Evaluations: Hematology

| Site/ Subject | Treatment | Visit | Day | Date | Laboratory Parameter (Units) | Value (1) | CFB |
|---|---|---|---|---|---|---|---|
| xx/xxxx | XXXXX | Pre-Study | | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | - | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | Baseline | | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | Cycle 1 | 8 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | Cycle 1 | 15 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 2 | 1 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 2 | 15 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 3 | 1 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | - | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |

(1) H=Abnormal High, L=Abnormal Low Normal ranges are given at the end of the listing.

CFB=Change from Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Programming Note: Continue for all cycles, Days 1 and 15.

Listing 16.2.8.1 Clinical Laboratory Evaluations: Hematology Normal Ranges

| Parameter | Gender | Age (Years) | Low - High |
|-----------------------------|--------|-------------|-------------|
| BASOPHILS (%) | _ | 18 - 65+ | 0 - 2 |
| BASOPHILS ABSOLUTE (GI/L) | _ | 18 - 65+ | 0 - 0.2 |
| EOSINOPHILS (%) | _ | 18 - 65+ | 0 - 7 |
| EOSINOPHILS ABSOLUTE (GI/L) | _ | 18 - 65+ | 0.05 - 0.55 |
| HEMATOCRIT (1) | Male | 18 - 64 | 0.41 - 0.50 |
| | Male | 65+ | 0.36 - 0.49 |
| | Female | 18 - 64 | 0.35 - 0.46 |
| | Female | 65+ | 0.33 - 0.46 |
| HEMOGLOBIN (G/L) | Male | 18 - 64 | 138 - 172 |
| | Male | 65+ | 118 - 168 |
| | Female | 18 - 64 | 120 – 156 |
| | Female | 65+ | 111 - 155 |
| LYMPHOCYTES (%) | _ | 18 - 65+ | 16 - 46 |
| LYMPHOCYTES ABSOLUTE (GI/L) | _ | 18 - 65+ | 0.85 - 4.10 |
| MONOCYTES (%) | _ | 18 - 65+ | 0 - 12 |
| MONOCYTES ABSOLUTE (GI/L) | _ | 18 - 65+ | 0.2 - 1.1 |
| PLATELET COUNT (GI/L) | _ | 18 - 65+ | 130 - 400 |
| RED CELL COUNT (TI/L) | Male | 18 - 64 | 4.4 - 5.8 |
| | Male | 65+ | 3.7 - 5.5 |
| | Female | 18 - 64 | 3.9 - 5.2 |
| | Female | 65+ | 3.6 - 5.1 |
| RETICULOCYTES (%) | _ | 18 - 65+ | 0.5 - 2.3 |
| RETICULOCYTES, ABS (10e9/L) | _ | 18 - 65+ | 25 - 85 |
| TOTAL NEUTROPHILS (%) | _ | 18 - 65+ | 40 - 75 |
| TOTAL NEUTROPHILS AB (GI/L) | _ | 18 - 65+ | 1.8 - 8.0 |
| WHITE CELL COUNT (GI/L) | _ | 18 - 65+ | 3.8 - 10.8 |

Ranges are given for adults (age at least 18 years).

Age (Years) = "18 - 65+" indicates that there is no restriction on normal due to age in adults.

Listing 16.2.8.2 Clinical Laboratory Evaluations: Blood Chemistry

| Site/ Subject | Treatment | Visit | Day | Date | Laboratory Parameter (Units) | Value (1) | CFB |
|---|---|---|---|---|---|---|---|
| (XX/XXXX | XXXXX | Pre-Study | | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | - | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | Baseline | | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | |
| | | Cycle 1 | 8 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 1 | 15 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 2 | 1 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 2 | 15 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | Cycle 3 | 1 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | - | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |

(1) H=Abnormal High, L=Abnormal Low Normal ranges are given at the end of the listing.

CFB=Change from Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Programming Note: Continue for all cycles, Days 1 and 15.

Listing 16.2.8.2 Clinical Laboratory Evaluations: Blood Chemistry Normal Ranges

| Parameter | Gender | Age (Years) | Low - High |
|-------------------------------|--------|-------------|-------------|
| ALAT (SGPT) (U/L) | _ | 18 - 65+ | 0 - 48 |
| ALBUMIN (G/L) | _ | 18 - 65+ | 32 - 50 |
| ALKALINE PHOSPHATASE (U/L) | _ | 20+ | 20 - 125 |
| ASAT (SGOT) (U/L) | _ | 18 - 64 | 0 - 42 |
| | _ | 65+ | 0 - 55 |
| BILIRUBIN, DIRECT (UMOL/L) | _ | 18 - 65+ | 0 - 6 |
| BILIRUBIN, TOTAL (UMOL/L) | _ | 18 - 65+ | 0 - 22 |
| CALCIUM (MMOL/L) | _ | 18 - 65+ | 2.12 - 2.56 |
| CARBON DIOXIDE (CO2) (MMOL/L) | _ | 18 - 65+ | 20 - 32 |
| CHLORIDE (MMOL/L) | _ | 18 - 65+ | 95 - 108 |
| GLUCOSE (MMOL/L) | _ | 18 - 49 | 3.9 - 6.4 |
| | _ | 50+ | 3.9 - 6.9 |
| LACTIC DEHYDROGENASE (U/L) | _ | 18 - 64 | 0 - 250 |
| | _ | 65+ | 0 - 270 |
| PHOSPHORUS INORGANIC (MMOL/L) | _ | 18 - 64 | 0.80 - 1.45 |
| | _ | 65+ | 0.7 - 1.4 |
| POTASSIUM (MMOL/L) | _ | 18 - 65+ | 3.5 - 5.3 |
| PROTEIN, TOTAL SERUM (G/L) | _ | 18 - 64 | 60 - 85 |
| | _ | 65+ | 58 - 81 |
| SODIUM (MMOL/L) | _ | 18 - 65+ | 135 - 146 |
| UREA NITROGEN (MMOL/L) | _ | 18 - 64 | 2.5 - 9 |
| | _ | 65+ | 2.5 - 10.5 |
| URIC ACID (UMOL/L) | Male | 18 - 65+ | 240 - 510 |
| . , | Female | 18 - 65+ | 150 - 450 |

Ranges are given for adults (age at least 18 years).

Age (Years) = "18 - 65+" indicates that there is no restriction on normal due to age in adults.

Listing 16.2.8.2 Clinical Laboratory Evaluations: Blood Chemistry Normal Ranges (CREATININE ENZ)

| Parameter | Gender | Age (Years) | Low - High |
|------------------------------|--------|-------------|--------------|
| CREATININE ENZ, SER (UMOL/L) | Male | 20 - 29 | 70.7 - 114.9 |
| | Male | 30 - 39 | 69.8 - 117.6 |
| | Male | 40 - 49 | 69.0 - 118.5 |
| | Male | 50 - 59 | 67.2 - 129.1 |
| | Male | 60 - 69 | 67.2 - 129.1 |
| | Male | 70+ | 59.2 - 136.1 |
| | Female | 30 - 39 | 51.3 - 93.7 |
| | Female | 40 - 49 | 52.2 - 94.6 |
| | Female | 50 - 59 | 53.0 - 97.2 |
| | Female | 60 - 69 | 53.0 - 104.3 |
| | Female | 70+ | 55.7 - 107.8 |

Ranges are given for adults (age at least 18 years).

Age (Years) = "18 - 65+" indicates that there is no restriction on normal due to age in adults.

Listing 16.2.8.3 Clinical Laboratory Evaluations: Coagulation

| | | | | | PTT | | INR | | PT | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site/<br>Subject | Treatment | Visit | Day | Date | Value (1) | CFB | Value (1) | CFB | Value (1) | CFB |
| xxx/xxxx | XXXXX | Pre-Study | - | MM/DD/YYYY | XXX | | XXX | | XXX | |
| | | Baseline | | MM/DD/YYYY | XXX | | XXX | | XXX | |
| | | Cycle 1 | 8 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | • | 15 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Cycle 2 | 1 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | - | 15 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Cycle 3 | 1 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | - | 15 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |

PTT= Partial Thromboplastin Time; INR= International Normalized Ratio; PT= Prothrombin Time (1) H=Abnormal High, L=Abnormal Low

Normal ranges are given at the end of the listing.

CFB=Change from Baseline

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Programming Note: Continue for all cycles, Days 1 and 15.

Listing 16.2.8.3

# Clinical Laboratory Evaluations: Coagulation Normal Ranges

| Parameter | Gender | Age (Years) | Low - High |
|-----------|--------|-------------|------------|
| PTT | _ | 18 - 65+ | 22 - 34 |
| INR | _ | 18 - 65+ | 0.9 - 1.1 |
| PT | _ | 18 - 65+ | 9 - 11.5 |

Ranges are given for adults (age at least 18 years).

Age (Years) = "18 - 65+" indicates that there is no restriction on normal due to age in adults.

Listing 16.2.8.4
Clinical Laboratory Evaluations: Urinalysis

| Site/ Subject | Treatment | Visit | Day | Date | Laboratory Parameter (Units) | Value |
|---|---|---|---|---|---|---|
| xxx/xxxx | XXXXX | Pre-Study | | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | Baseline | | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | Cycle 1 | 8 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | Cycle 1 | 15 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | Cycle 2 | 1 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | Cycle 2 | 15 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | Cycle 3 | 1 | MM/DD/YYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |

Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Programming Notes: Continue for all cycles, Days 1 and 15. CFB is not computed for any urinalysis parameter.

Listing 16.2.8.5 Clinical Laboratory Evaluations: Thyroid Function

| | | | | T3 (U | nit) | T4 (U | nit) | TSH (I | Jnit) |
|---|---|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Visit | Date | Value (1) | CFB | Value (1) | CFB | Value (1) | CFB |
| xxx/xxxx | XXXXX | Pre-Study | MM/DD/YYYY | XXX | | XXX | | XXX | |
| | | Cycle 1 | MM/DD/YYYY | XXX | | XXX | | XXX | |
| | | Cycle 2 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Cycle 3 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| xxx/xxxx | xxxxx | Pre-Study | MM/DD/YYYY | XXX | | XXX | | xxx | |
| | | Cycle 1 | MM/DD/YYYY | XXX | | XXX | | XXX | |
| | | Cycle 2 | MM/DD/YYYY | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Cycle 3 | MM/DD/YYYY | XXX | xxx | XXX | XXX | XXX | XXX |

<sup>(1)</sup> H=Abnormal High, L =Abnormal Low

Normal ranges are given at the end of the listing. CFB=Change from Baseline

Baseline=Cycle 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

Programming Notes: Continue for all cycles. Include units. Column for "Day" deleted since Thyroid Function assessed only at Day 1.

Listing 16.2.8.5 Clinical Laboratory Evaluations: Thyroid Function Normal Ranges

| Parameter | Gender | Age (Years) | Low - High |
|-----------|--------|-------------|-------------|
| T3 | _ | 18 - 65+ | 3.5 - 6.5 |
| T4 | _ | 18 - 65+ | 10.3 - 23.2 |
| TSH | - | 20+ | 0.4 - 4.5 |

Ranges are given for adults (age at least 18 years).

Age (Years) = "18 - 65+" indicates that there is no restriction on normal due to age in adults.

**Listing 16.2.8.6**Pregnancy Test

| Site/ Subject | Treatment | Visit | Test Date | Result | Not Done? | Not Applicable? | Menopausal date/<br>Other Specify |
|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXXX | Pre-Study | DD/MM/YY | XXXX | | • • | |
| | | Cycle 1 | DD/MM/YY | XXXX | | | |
| | | Cycle 2 | DD/MM/YY | | XXXX | | |
| | | Cycle 3 | DD/MM/YY | XXXX | | | |
| xxx/xxxxx | XXXXX | Pre-Study | DD/MM/YY | | | XXXX | |
| | | Cycle 1 | DD/MM/YY | | | XXXX | |
| | | Cycle 2 | DD/MM/YY | | | XXXX | |
| | | Cycle 3 | DD/MM/YY | | | XXXX | |

Programming Note: Continue for all cycles. For "Not Applicable?", enter reason if not applicable.

Listing 16.2.9.1

Vital Signs

| | | | | Systol | | Diasto | | | <b>Femperat</b> | | Respirat | • | Pu | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | (mm | Hg) | (mm | ıHg) | | (degrees | C) | (/m | nin) | (beats | s/min) |
| Site/ Subject | Treatment | Visit | Time | Value | CFB | Value | CFB | Value | CFB | Method | Value | CFB | Value | CFB |
| xxx/xxxxx | XXXX | Pre-Study | | XXX | | XXX | | XXX | | Х | XXX | | XXX | |
| | | Cycle 1 | Day 1 | XXX | | XXX | | XXX | | X | XXX | | XXX | |
| | | | Day 1<br>Hour 1 | XXX | XXX | XXX | XXX | XXX | XXX | X | XXX | XXX | XXX | XXX |
| | | | Day 1<br>Hour 2 | xxx | XXX | XXX | XXX | XXX | XXX | Х | XXX | XXX | XXX | XXX |
| | | | Day 8 | XXX | xxx | xxx | xxx | xxx | xxx | х | xxx | xxx | xxx | XXX |
| | | | Day 15 | XXX | XXX | XXX | XXX | XXX | XXX | X | XXX | XXX | XXX | XXX |
| | | Cycle 2 | Day 1 | XXX | XXX | XXX | XXX | XXX | XXX | X | XXX | XXX | XXX | XXX |
| | | | Day 15 | XXX | XXX | XXX | XXX | XXX | XXX | X | XXX | XXX | XXX | XXX |
| | | Cycle 3 | Day 1 | XXX | XXX | XXX | XXX | XXX | XXX | x | XXX | XXX | XXX | XXX |
| | | | Day 15 | XXX | XXX | XXX | XXX | XXX | XXX | X | XXX | XXX | XXX | XXX |

CFB=Change from Baseline Baseline=Cycle 1 Day 1 (or Pre-Study if value at Cycle 1 Day 1 is missing) Method= 'O' for oral, 'A' for Axillary

Programming Note: Continue for all visits (Days 1 and 15 of each cycle, Day 8 of Cycle 1, and Hours 1, 2, 3, 4, 6 and 8 on Cycle 1 Day 1) with CFB.

Listing 16.2.9.2 Weight, Height, and BMI

| | | | | | Weigh | nt (kg) | BMI (k | g/m^2) |
|---|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Visit | Time | Height (cm) | Value | CFB | Value | ĆFB |
| xxx/xxxxx | XXXX | Pre-Study | | XXX | XXX | | XXX | |
| | | Cycle 1 | Day 1 | | XXX | | XXX | |
| | | | Day 8 | | XXX | XXX | XXX | XXX |
| | | | Day 15 | | XXX | XXX | XXX | XXX |
| | | Cycle 2 | Day 1 | | XXX | XXX | XXX | XXX |
| | | | Day 15 | | XXX | XXX | XXX | XXX |
| | | Cycle 3 | Day 1 | | XXX | XXX | XXX | XXX |
| | | | Day 15 | | XXX | XXX | XXX | XXX |
| xxx/xxxxx | XXXX | Pre-Study | | XXX | XXX | | XXX | |
| | | Cycle 1 | Day 1 | | XXX | | XXX | |
| | | | Day 8 | | XXX | XXX | XXX | XXX |
| | | | Day 15 | | XXX | XXX | XXX | XXX |
| | | Cycle 2 | Day 1 | | XXX | XXX | XXX | XXX |
| | | | Day 15 | | XXX | XXX | XXX | XXX |
| | | Cycle 3 | Day 1 | | XXX | XXX | XXX | XXX |
| | | | Day 15 | | XXX | XXX | XXX | XXX |

CFB=Change from Baseline
Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)
BMI=Body mass index.

BMI is computed using Height recorded at Pre-Study.

Programming Note: Continue for all cycles.

Listing 16.2.9.3 **ECOG Performance Status** 

| | | | Assessment | | CFB |
|---------------|-----------|-----------|------------|---------|---------|
| Site/ Subject | Treatment | Visit | Date | ECOG PS | ECOG PS |
| xxx/xxxxx | XXXX | Pre-Study | DD/MM/YY | XXX | |
| | | Cycle 1 | DD/MM/YY | XXX | |
| | | Cycle 2 | DD/MM/YY | XXX | XXX |
| | | Cycle 3 | DD/MM/YY | XXX | XXX |
| | | Cycle 4 | DD/MM/YY | XXX | XXX |
| xxx/xxxxx | XXXX | Pre-Study | DD/MM/YY | XXX | |
| | | Cycle 1 | DD/MM/YY | XXX | |
| | | Cycle 2 | DD/MM/YY | XXX | XXX |
| | | Cycle 3 | DD/MM/YY | XXX | XXX |
| | | Cycle 4 | DD/MM/YY | XXX | XXX |

CFB=Change from Baseline
Baseline=Cycle 1 Day 1 (or Pre-Study if <= 3 days prior to Cycle 1 Day 1 or if value at Cycle 1 Day 1 is missing)

PS = Performance Status

0=Normal activity, 1=Symptoms but ambulatory, 2= In bed <50% of time, 3=In bed >50% of time, 4=100% bedridden

Programming Notes: Continue for all cycles. Record CFB as Decrease, No Change, or Increase.

Listing 16.2.10.1

Electrocardiogram (ECG) – Continuous Variables

| | | | | | | | | | | | Interva | al (msec) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Heart<br>(bp | | Р | R | QF | RS | Q <sup>-</sup> | Γ | QTcF | <del>-</del> (1) |
| Site/ | | | | | | | | | | | | | | | |
| Subject | Treatment | Visit | Day | Hour | Time | Value | CFB | Value | CFB | Value | CFB | Value | CFB | Value | CFE |
| xxx/xxxxx | XXXXXXX | Pre-Study | | | XX:XX | XX | | XX | | XX | | XX | | XX | |
| | | Cycle 1 | 1 | 0 | XX:XX | XX | | XX | | XX | | XX | | XX | |
| | | | | 2 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | 4 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | 6 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | 8 | 0 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | 2 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | 4 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | | 6 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | 15 | 0 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Cycle 2 | 1 | 0 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | - | 15 | 0 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Cycle 3 | 1 | 0 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | | 15 | 0 | XX:XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Hour 0=Pre-Dose

CFB=Change from Baseline

Baseline=Cycle 1 Day 1 Hour 0 (or Pre-Study if the value at Cycle 1 Day 1 is missing)

(1) QTcF=QT Correction: Fridericia.

Programming Notes: Continue for QRS Complex (msec), PR Interval (msec), and QTcF (msec) in that order and all visits (Pre-Study, Predose on Days 1 and 15 of all cycles, Pre-dose on Day 8 of Cycle 1, and at 2, 4, and 6 hours post-dose on Days 1 and 8 of Cycle 1) with CFB. Compute QTcF=QT\*(HR/60)<sup>1/3</sup>.

Listing 16.2.10.2

Electrocardiogram (ECG) – Categorical Variables

| | | | | | | Overall | | Cardiac |
|---|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Visit | Day | Hour | Time | Impression (1) | ST Segment | Rhythm |
| xxx/xxxxx | XXXX | Pre-Study | | | | XX | XX | XX |
| | | Cycle 1 | 1 | 0 | XX:XX | XX | XX | XX |
| | | | | 2 | XX:XX | XX | XX | XX |
| | | | | 4 | XX:XX | XX | XX | XX |
| | | | | 6 | XX:XX | XX | XX | XX |
| | | | 8 | 0 | XX:XX | XX | XX | XX |
| | | | | 2 | XX:XX | XX | XX | XX |
| | | | | 4 | XX:XX | XX | XX | XX |
| | | | | 6 | XX:XX | XX | XX | XX |
| | | | 15 | 0 | XX:XX | XX | XX | XX |
| | | Cycle 2 | 1 | 0 | XX:XX | XX | XX | XX |
| | | | 15 | 0 | XX:XX | XX | XX | XX |
| | | Cycle 3 | 1 | 0 | XX:XX | XX | XX | XX |
| | | - | 15 | 0 | XX:XX | XX | XX | XX |

Programming Note: Continue for all visits (Pre-Study, Pre-dose on Days 1 and 15 of all cycles, Pre-dose on Day 8 of Cycle 1, and at 2, 4, and 6 hours post-dose on Days 1 and 8 of Cycle 1).

<sup>(1) 1=</sup>Normal, 2=Abnormal Not Clinically Significant, 3= Abnormal Clinically Significant Hour 0 = Pre-Dose

Listing 16.2.11.1
Physical Examination at Pre-Study Visit

| Site/ Subject | Treatment | Body System | Result | Description If 'Abnormal' |
|---|---|---|---|---|
| xxx/xxxxx | XXXXX | General Appearance | Normal | |
| | | Head and Neck | Normal | |
| | | Eyes, Ears, Nose, Throat | Abnormal | XXXXX |
| | | Skin | Normal | |
| | | Chest / Lungs / Breast | Normal | |
| | | Heart | Normal | |
| | | Abdomen | Abnormal | XXXXX |
| | | Genitourinary | Normal | |
| | | Extremities | Normal | |
| | | Musculoskeletal | Normal | |
| | | Lymph Nodes | Abnormal | XXXXX |
| | | Neurological | Normal | |
| | | Other | Normal | XXXXX |
| xxx/xxxxx | XXXXX | General Appearance | Normal | |
| | | Head and Neck | Normal | |
| | | Eyes, Ears, Nose, Throat | Normal | |
| | | Skin | Normal | |
| | | Chest / Lungs / Breast | Normal | |
| | | Heart | Not Done | |
| | | Abdomen | Normal | |
| | | Genitourinary | Normal | |
| | | Extremities | Normal | |
| | | Musculoskeletal | Normal | |
| | | Lymph Nodes | Abnormal | XXXXX |
| | | Neurological | Normal | |
| | | Other | Not Done | |

Programming Note: Record result as 'Normal', 'Abnormal', or 'Not Done'

**Listing 16.2.11.2**Physical Examination

| | | | Screening <= 3 days from | Clin, Sig, | | | Description If different From |
|---|---|---|---|---|---|---|---|
| Site/ Subject | Treatment | Visit | Baseline? | Changes (1) | Body System | Result | Previous Assessment |
| xxx/xxxxx | XXXXX | Cycle 1<br>Day 1 | No | No | | | |
| | | Cycle 1<br>Day 8 | | No | | | |
| | | Cycle 1<br>Day 15 | | No | | | |
| | | Cycle 2<br>Day 1 | | Yes | Eyes, Ears, Nose, Throat | Abnormal | XXXXX |
| | | • | | Yes | XXXXXXXXXXXXX | XXXXXX | xxxxxxxxxxxx |
| | | Cycle 2<br>Day 15 | | No | | | |
| | | Cycle 3<br>Day 1 | | Yes | Lymph Nodes | XXXXXX | XXXXX |
| | | Cycle 3<br>Day 15 | | No | | | |
| | | Cycle 4<br>Day 1 | | No | | | |
| xxx/xxxxx | xxxxx | Cycle 1<br>Day 1 | Yes | | | | |
| | | Cycle 1<br>Day 8 | | No | | | |
| | | Cycle 1<br>Day 15 | | No | | | |
| | | Cycle 2<br>Day 1 | | Yes | | | |

<sup>(1)</sup> Are there any clinically significant changes from the physical examination conducted at the previous assessment? Baseline=Cycle 1 Day 1

Programming Notes: Continue for other cycles. If there are 'No' clinically significant changes from the physical examination conducted at the previous assessment, then the assessments for individual body systems should not be completed.

If "Clin, Sig, Changes" = 'Yes', then results should be recorded for at least one body systems with a "Result" differing from the previous assessment list. If "Screening <= 3 days from Baseline?" is Yes, there should be no responses for Cycle 1 Day 1.

Listing 16.2.12 **Prior and Concomitant Medications** 

| Site/ Subject | Treatment | Medication | ATC Level 3 | Reason for Use | AE no.<br>(1) | Dose & Units | Regimen | Route (2) | Start Date<br>Stop Date<br>(3) |
|---|---|---|---|---|---|---|---|---|---|
| xxx/xxxxx | XXXXX | XXXX | XXXX | XXXXX | Х | XXXX | XXXX | XX | DD/MM/YY |
| xxx/xxxxx | xxxxx | XXXX | xxxx | xxxxx | x | xxxx | xxxx | xx | DD/MM/YY<br>DD/MM/YY<br>DD/MM/YY |
| xxx/xxxxx | xxxxx | xxxx | xxxx | XXXXX | х | xxxx | xxxx | xx | DD/MM/YY<br>O |

Includes medications taken within 30 days prior to Screening Visit.

Programming Note: Sort by start date for each subject.

<sup>(1)</sup> Blank if Not Applicable
(2) 1=PO; 2=IV; 3=SC; 5=IM; 11=T; 12=OU,OS,OD; 13=AU,AS,AD; 14=IN; 15=PV; 16=PR; 24=SL; 30=BUC; 37=IA; 71=NG; 136=INH; 358=TD; 135=Other; 139= Unknown

<sup>(3)</sup> O=Ongoing

Listing 16.2.13

# Investigator Comments

| Site/ Subject | Treatment | Date Event Occurred<br>or Study Visit | CRF Page(s) | Description of Event/Comment |
|---|---|---|---|---|
| xxx/xxxxx | XXXXX | DD/MM/YY | XX | XXXXXXXXXX |
| xxx/xxxxx | XXXXX | DD/MM/YY | XX | XXXXXXXXXXX |
| xxx/xxxxx | XXXXX | DD/MM/YY | XX | XXXXXXXXXXX |

Programming Notes: Sort by date/visit.
Include only subjects for whom the "None" box is not checked, i.e. only subjects with comments.